# **Statistical Analysis Plan**

Interventional, randomized, double-blind, parallel-group, placebo-controlled, multi-centre study to assess the efficacy, safety and tolerability of Lu AF82422 in patients with Multiple System Atrophy

### Lu AF82422

Trial No.: 18331A (AMULET – Delay Multiple System Atrophy)

Sponsor: H. Lundbeck A/S (Lundbeck)

2500 Valby (Copenhagen), Denmark

Biostatistician: PPD

SAP date: 20 December 2023

This document is the property of H. Lundbeck A/S and H. Lundbeck A/S is the holder of any and all related intellectual property rights, including, but not limited to, copyrights. This document is confidential. It is not to be copied or distributed to other parties without prior written authorization from H. Lundbeck A/S.

# **Table of Contents**

| List | t of Pa | nels and Tables | 6 |
|------|---------|--------------------------------------------------------|----|
| List | t of Ab | breviations and Definitions of Terms | 7 |
| 1 | Ohio | ectives | Q |
| 1 | 1.1 | Primary Objective | |
| | 1.2 | Secondary Objectives | |
| | 1.3 | Safety Objectives | |
| | 1.4 | Exploratory Objectives | |
| 2 | Stud | y Design | 9 |
| 3 | Defi | nitions | 10 |
| | 3.1 | Definition of Baseline | 10 |
| | | 3.1.1 Double Blind Period | |
| | | 3.1.2 Open-label Extension Period | |
| | 3.2 | Definition of Periods. | |
| | 3.3 | Definition of Withdrawal | 11 |
| 4 | Endi | points | 11 |
| | 4.1 | Primary Endpoint, Double-Blind Period | |
| | 4.2 | Key Secondary Endpoint, Double-Blind Period | |
| | 4.3 | Secondary Endpoints, Double-Blind Period | |
| | 4.4 | Safety Endpoints | |
| | | 4.4.1 Double-Blind Period | |
| | | 4.4.2 Open-label Extension Period | 13 |
| | 4.5 | Exploratory Endpoints | |
| | | 4.5.1 Double-Blind Period | |
| | | 4.5.2 Open-label Extension Period | 14 |
| 5 | Anal | ysis Sets | 15 |
| 6 | Desc | riptive Statistics | 16 |
| 7 | Patie | ent Disposition | 16 |
| | 7.1 | Summary of Patient Disposition | |
| | 7.2 | Withdrawals | |
| 8 | Dem | ographics and Baseline Characteristics | 16 |
| 9 | Rece | ent and Concomitant Medication | 17 |
| 10 | Expo | osure | 17 |
| 11 | Fall | Diary Compliance | 18 |
| 12 | Wea | rable Compliance | 18 |
| 13 | Prim | nary Estimand | 19 |
| 14 | Effic | acy | 20 |
| - | 14.1 | Overview of Planned Efficacy Analyses in the DB-Period | |
| | 14.2 | General Efficacy Analysis Methodology | |
| | 14.3 | • • | |

| | | 14.3.1 Primary Analysis of the Primary Endpoint | |
|---|---|---|---|
| | | 14.3.2 Posterior Summaries | |
| | | <ul> <li>14.3.3 Rationale for Selected Analysis Method for the Primary Endpoint</li> <li>14.3.4 Evaluation of Model Assumptions for the Primary Analysis of the Primary</li></ul> | |
| | | Endpoint | • |
| | | 14.3.5 Sensitivity Analyses of the Primary Endpoint | |
| | | 14.3.6 Subgroup Analyses of the Primary Endpoint | |
| | | 14.3.7 Covariate Analyses of the Primary Endpoint | |
| | 14.4 | Analysis of the Secondary Endpoints | |
| | | 14.4.1 Analysis Methodology for the Key Secondary Endpoint | |
| | | 14.4.2 Analysis Methodology for the Secondary Endpoint | |
| | 14.5 | Additional Analyses of Primary and Secondary Endpoints | |
| | 14.6 | Analysis of Exploratory Endpoints | 30 |
| 15 | Testir | ng Strategy | 31 |
| 10 | 15.1 | Calibrating primary analysis | 31 |
| | 15.2 | Testing Strategy including Secondary Endpoint(s) | |
| 16 | | | |
| 16 | <b>Sarety</b> 16.1 | Adverse Events | |
| | 10.1 | 16.1.1 General Methodology for Adverse Events | |
| | | 16.1.2 Coding of Adverse Events | |
| | | 16.1.3 Classification of Adverse Events | |
| | | 16.1.4 Allocation of TEAEs to Study Periods | |
| | | 16.1.5 Presentation of Adverse Events | |
| | | 16.1.6 Presentation of Treatment-emergent Adverse Events | |
| | | 16.1.7 Presentation of Deaths | |
| | | 16.1.8 Presentation of Serious Adverse Events | 34 |
| | | 16.1.9 Presentation of Adverse Events Leading to Withdrawal | 34 |
| | | 16.1.10 Presentation of Adverse Events Leading to Study Drug Infusion | |
| | | Interruption or Infusion Rate Reduction | |
| | | 16.1.11 Presentation of Adverse Events requiring additional data collection | |
| | 16.2 | General Methodology for Other safety Data | |
| | 16.3 | Clinical Safety Laboratory Test Data | |
| | 164 | 16.3.1 Data Presentation | |
| | 16.4 | Vital Signs and Weight | |
| | 16.5 | ECG Columbia-Suicide Severity Rating Scale (C-SSRS) Scores | |
| | 16.6<br>16.7 | MRI Safety Findings | |
| | 16.7 | Pregnancy Test | |
| | 16.9 | Events of Death | |
| 17 | Phari | nacokinetic/Pharmacodynamic Analysis | 38 |
| 18 | | unogenicity Analysis (ADA) | |
| 19 | | ed Data Reviews | |
| 20 | | m Analyses | |
| | | • | |
| 21 | • | le Size Considerations | |
| 22 | | tical Software | |
| 23 | ('han | ges to Analyses Specified in the Protocol | 41 |

| 24 | Detai | ls on Data | a Handling | 41 |
|---|---|---|---|---|
| | 24.1 | | Variables | |
| | | 24.1.1 | Missing Item Scores | 41 |
| | | 24.1.2 | UMSARS scale | |
| | | 24.1.3 | Composite Autonomic Symptom Score Select (COMPASS Select) | 45 |
| | | 24.1.4 | Schwab & England Activity Daily Living Scale (SE-ADL) | |
| | | 24.1.5 | Clinical Global Impression Severity Scale (CGI-S) | |
| | | 24.1.6 | Patient global Impression Scale (PGI-S) | |
| | | 24.1.7 | Observer-reported Global Impression – Severity of Illness (OGI-S) | 47 |
| | | 24.1.8 | EuroQoL five-dimensional five-levels Scale (EQ-5D-5L) | 47 |
| | | 24.1.9 | FeetMe® gait parameters | 48 |
| | | 24.1.10 | BioSensics <sup>TM</sup> PAMSys sensor | 49 |
| | | 24.1.11 | Fall Diary | 50 |
| | | 24.1.12 | Magnetic Resonance Imaging (MRI) | 51 |
| | 24.2 | Assignir | ng Data to Visits | 52 |
| | | 24.2.1 | UMSARS and additional efficacy COAs | 52 |
| | | 24.2.2 | MRI parameters | 54 |
| | | 24.2.3 | Blood sampling parameters | 55 |
| | | 24.2.4 | Vital signs and C-SSRS | 56 |
| | | 24.2.5 | Weight | 56 |
| | | 24.2.6 | ECG | 57 |
| | | 24.2.7 | Fall Diary | 57 |
| | 24.3 | Assignir | ng Adverse Events to Analysis Phases | 58 |
| | 24.4 | Handlin | g Missing or Incomplete Dates/Times | 58 |
| | | 24.4.1 | IMP Start and Stop Dates | 58 |
| | | 24.4.2 | Withdrawal Date | 59 |
| | | 24.4.3 | Medication Start and Stop Dates | 59 |
| | | 24.4.4 | Adverse Event Start and Stop Dates | 59 |
| | | 24.4.5 | Diagnosis and Symptom onset Start Dates | 59 |
| | 24.5 | Data wit | th Multiple Records | 60 |
| | | 24.5.1 | Dose Changes in Medication | 60 |
| | | 24.5.2 | Changes in Intensity or Seriousness of Adverse Events | 60 |
| | 24.6 | Handlin | g Exposure Data | 61 |
| | 24.7 | Handlin | g digital-device data | 61 |
| Ref | erence. | | | 62 |

# Appendices

| Appendix I | Statistical Analysis Plan Authentication and Authorization | 63 |
|---|---|---|
| Appendix II | SAS® Code | 65 |
| Appendix III | 'R' code | 68 |
| Appendix IV | Study Flow Chart | 71 |
| Appendix V | PCS Criteria | 78 |
| Appendix VI | Definition of Hypersensitivity related reactions | 82 |
| Appendix VII | Definition of Concomitant Medication Category | 93 |

# **List of Panels and Tables**

| Panel 1 | Study Design | 10 |
|---|---|---|
| Panel 2 | Overview of Planned Efficacy Analyses (DB-Period) | 20 |
| Panel 3 | C-SSRS Scores | 37 |
| Panel 4 | ADA definitions. | 38 |
| Panel 5 | Published UMSARS Progression | 40 |
| Panel 6 | Maximum Number of Missing Items on Rating Scales | 42 |
| Panel 7 | Imputation of worst rank following events of death | 42 |
| Panel 8 | UMSARS Scale Overview | 43 |
| Panel 9 | Derivation of UMSARS total score and domain scores | 45 |
| Panel 10 | COMPASS Select Change domain scores | 46 |
| Panel 11 | SE-ADL Scoring | 46 |
| Panel 12 | Derivation of gait parameters, by-step | 49 |
| Panel 13 | Derivation of PAMSys parameters | 50 |
| Panel 14 | Derivation of Fall Diary parameters | 51 |
| Panel 15 | Derivation of MRI parameters | 52 |
| Panel 16 | Visit Windows for UMSARS | 53 |
| Panel 17 | Visit Windows for MRI | 54 |
| Panel 18 | Visit Windows for Blood Sampling Parameters | 55 |
| Panel 19 | Visit Windows for Weight | 57 |
| Panel 20 | Visit Windows for ECG | 57 |
| Panel 21 | Windows for Fall Diary (Periods) | 58 |
| Table 1 | Study Procedures and Assessments - Double-blind Treatment Period | 72 |
| Table 2 | Optional Open-label Long-term Extension Treatment Period | 76 |
| Table 3 | PCS Criteria for Clinical Safety Laboratory Tests | 79 |
| Table 4 | PCS Criteria for Vital Signs, Weight/BMI, and Waist Circumference | 81 |
| Table 5 | PCS Criteria for ECG Parameters | 81 |

# List of Abbreviations and Definitions of Terms

ANCOVA Analysis of Covariance APTS all-patients-treated set

aUMSARS abbreviated Unified Multiple System Atrophy Rating Scale

CI confidence interval

DMC Data Monitoring Committee
DTI Diffusion-tensor imaging
eCRF electronic case report form

EoTDBP End of treatment double-blind period

EoTOLEP End of treatment open-label extension period

FAS full-analysis set

IMP investigational medicinal product

MedDRA Medical Dictionary for Regulatory Activities

ML maximum likelihood

MMRM mixed model for repeated measurements

MSA multiple system atrophy

mUMSARS modified Unified Multiple System Atrophy Rating Scale

NfL neurofilament light chain

OC observed case(s)

PYE patient years of exposure

R Open source statistical software package

SAE serious adverse event

SAS<sup>®</sup> statistical software package from the SAS<sup>®</sup> Institute

SD standard deviation SOC system organ class

TEAE treatment-emergent adverse event

UMSARS Unified Multiple System Atrophy Rating Scale

vMRI volumetric magnetic resonance imaging

# 1 Objectives

### 1.1 Primary Objective

• To evaluate the efficacy of Lu AF82422 on disease progression in patients with Multiple System Atrophy (MSA) during the Double-blind Period (DBP)

### 1.2 Secondary Objectives

- To evaluate the efficacy of Lu AF82422 on:
  - Function
  - Global impression, severity of illness
  - Autonomic symptoms
  - Global disability
  - Disease milestones
  - Health-related quality of life
- To evaluate the efficacy of Lu AF82422 on disease progression measured by brain Magnetic Resonance Imaging (MRI)
- To evaluate the efficacy of Lu AF82422 on biofluid biomarkers of disease progression
- To evaluate the pharmacokinetics of Lu AF82422

All during the Double-blind Period (DBP).

### 1.3 Safety Objectives

• To evaluate the safety and tolerability of Lu AF82422 in patients with MSA during the Double-blind Period (DBP) and the open-label extension (OLE)

### 1.4 Exploratory Objectives

- To explore the target engagement of Lu AF82422 to α-synuclein
- To explore the target engagement of Lu AF82422 on pathological species of α-synuclein
- To explore the relationship between UMSARS, MRI parameters and NfL
- To explore the efficacy of Lu AF82422 for up to 72 weeks of treatment on clinical scales and biomarkers
- To collect patient experience with impaired functions due to MSA to support the interpretation of change on the UMSARS (Exit Interview subset)
- To collect patient experience with study participation (Study Experience Interview subset)

All during the Double-blind Period (DBP).

• To explore the effect of long-term treatment with Lu AF82422 during the open-label extension (OLE)

# 2 Study Design

- This is a phase II, interventional, randomized, double-blind, parallel-group, placebo-controlled, multi-centre study of the efficacy (slowing disease progression), safety, and tolerability of Lu AF82422 in patients with MSA. The efficacy of Lu AF82422 is assessed using the UMSARS TS; supportive assessments include evaluation of function, global impression of severity of illness, autonomic symptoms, disability, health-related quality of life, biofluid biomarkers, and imaging.
- The target population for this study is patients with possible or probable MSA, as defined by the 2008 Gilman diagnostic criteria. The study will recruit patients with evidence of parkinsonism (MSA-P) and/or cerebellar syndrome (MSA-C). Patients will be allowed stable treatment for managing their symptoms of MSA during the study.
- The patients [N=60] will be randomized to Lu AF82422 CCl or placebo (2:1) via a centralized randomization system (Interactive Response Technology [IRT]). Two strata variables will be applied to ensure a balanced treatment allocation of Lu AF82422 and placebo: CCl and Region (US/Japan, with a maximum of 25% of patients from Japan).
- The study duration from the Screening Visit to the Safety follow-up Visit is between 70 to 94 weeks for patients not entering the optional OLE period and between 118 to 142 weeks for patients continuing in the OLE. The study includes the following periods:
  - Screening period (4 weeks)
  - o Randomization period (2 weeks)
  - o Double-blind treatment period (48 weeks up to 72 weeks)
  - o Optional OLE treatment period (48 weeks)
  - o Safety Follow-up Period (20 weeks; will take place after last investigational medicinal product [IMP] administration)
- The individual double-blind period will vary from 48 weeks up to 72 weeks. Once the last patient will reach Week 48, this visit will be the EoTDBP Visit for that patient. Patients who have not completed the visit at Week 72 at the time of Last Patient reaches EoT will have their next visit converted to an DBP EoT Visit with assessments as listed for Visit 24, according to study procedures and assessments (Appendix IV). During the double-blind treatment period, patients will attend IMP Visits to follow a dosing schedule with either Lu AF82422 or placebo every four weeks (Q4W).
- Patients who enter the OLE will receive the first open-label dose (Visit 1E) at the same day as the EoTDBP or as soon as possible thereafter, but not later than 5 months after EoT Visit of the DBP and will be enrolled to OLE no later than end of Q1 2024.
- After the DBP EoT/ End of Open-Label Treatment/Withdrawal Visit, patients will be scheduled for a Safety Follow-up Visit 20 weeks after last IMP dose.
- An independent Data Monitoring Committee (iDMC) will regularly monitor the patients' safety and tolerability data according to the Data Monitoring Committee (DMC) Charter.

An overview of the study is presented in Panel 1.

### Panel 1 Study Design



- Variable treatment period of minimum 48 weeks up to 72 weeks of treatment. Patients who have not completed Week 72 Visit at
  the time Last Patient reaches Week 48, will be scheduled for the EoT DBP Visit 4 weeks after latest dose of IMP
- 2. Patients who do not continue in the optional Open-Label Extension will enter the Safety Follow-up Period after the EoT DBP Visit

DBP = Double-Blind Period; EoT = End of Treatment; SoC = Standard of Care; Q4W = every 4 weeks

## 3 Definitions

#### 3.1 Definition of Baseline

### 3.1.1 Double Blind Period

The baseline value for the DBP is the value captured at the Baseline Visit (week 0). In case an assessment has not been performed at the Week 0 Baseline visit or the Week 0 value is missing or invalid, the value from the last completed pre-IMP assessment will be used as baseline.

The screening visit takes place approx. 6 weeks prior and the randomisation visit approx. 2 weeks prior the baseline visit.

### 3.1.2 Open-label Extension Period

The baseline value for patients who enter the OLE and who have the first visit of the OLE at the same day of the EoTDBP Visit or up to 7 days after the EoTDBP, clinical assessments performed at the EoTBDP Visit will serve as the baseline value for the OLE. For patients entering OLE >7 days after EoTDBP, the OLE baseline value is the value captured at the dedicated Visit 1E.

### 3.2 Definition of Periods

The study consists of the following periods:

- Screening Period (4 weeks): Screening Visit (V1) to Randomization Visit (V2)
- Randomization Period (2 weeks): Randomization Visit (V2) to Baseline DB Visit (V3)
- Double-blind Treatment Period (varying: 48 to 72 weeks): Baseline DB Visit (V3) to
   EoTDB Visit (V24) Time point to be defined by IMP initiation on V3
- Optional Open-Label Treatment Period (48 weeks): from Baseline OLE Visit (V1E) to EoTOLE (V13E) - Time point to be defined by IMP initiation on V1E

Patients will subsequently after end IMP administration enter:

- Safety Follow-up Period 1 following DB (20 weeks): following the EoTDBP Visit (V24) to Safety Follow-up Visit (V25)
- Safety Follow-up Period 2 following OLE (20 weeks): following the EoTOLE Visit (V13E) to Safety Follow-up Visit (SFU-E)

Due to the late approval of the OLE protocol amendment some participants entering the OLE might have entered the first safety follow-up period prior to entering the OLE, and hence would have two safety follow-up periods.

### 3.3 Definition of Withdrawal

The group of patients who withdrew from treatment at the scheduled visits in the Double-blind Treatment Period will be described as *withdrawn from study*. This group will also contain randomized patients who withdrew from treatment prior to receiving any IMP and patients who died. The complementary group will be described as *completed study*. Patients who withdraw, except for those who withdraw their consent or died, will be asked to attend a Safety Withdrawal Visit 20 weeks after the last dose of IMP and undergo Safety Follow-Up evaluations.

Participants that drop out of the OLE will also undergo Safety Follow-Up evaluations according to trial procedures.

# 4 Endpoints

### 4.1 Primary Endpoint, Double-Blind Period

### **Disease progression**

• as assessed by longitudinal changes from baseline in the Unified Multiple System Atrophy Rating Scale (UMSARS) Part I and Part II Total Score (UMSARS TS) up to EoTDB

### 4.2 Key Secondary Endpoint, Double-Blind Period

### Disease progression

 as assessed by longitudinal changes from baseline in the modified UMSARS Part I (mUMSARS) score up to EoTDB

## 4.3 Secondary Endpoints, Double-Blind Period

### **Disease progression**

 as assessed by longitudinal changes from baseline in the UMSARS Part I, and UMSARS Part II scores up to EoTDB

#### **Function**

- Change from baseline to Week 48 in UMSARS TS
- Change from baseline to Week 48 in UMSARS Part I score
- Change from baseline to Week 48 in mUMSARS score
- Change from baseline to Week 48 in UMSARS Part II score
- Change from baseline to Week 48 in Schwab and England Activities of Daily Living scale (SE-ADL)

### **Global impression**

- Change from baseline to Week 48 in Clinical Global Impression Severity (CGI-S) score
- Change from baseline to Week 48 in Patient Global Impression Severity (PGI-S) score
- Change from baseline to Week 48 in Observer-reported Global Impression Severity of Illness (OGI-S)

### **Autonomic symptoms**

• Change from baseline to Week 48 in Composite Autonomic Symptom Score Select Change (COMPASS Select Change) score

# Global disability

Change from baseline to Week 48 in UMSARS Part IV score

### **Disease milestones**

- Change from baseline to Week 48 in speech, swallowing, falls, and walking, as assessed by the UMSARS Part I sub-items
- Change from baseline to Week 48 in frequency, cause and consequence of falls, as assessed by the fall diary in dedicated periods

### Health-related quality of life

• Change from baseline to Week 48 in EQ-5D-5L score (individual items and VAS score)

#### MRI biomarkers

• Percentage change from baseline to Week 48 in brain volume in brain regions-of-interest (ROIs); primary ROIs: pons and cerebellum; secondary ROIs: caudate nucleus, putamen, brain stem and total grey matter, as measured by volumetric MRI (vMRI)

#### **Biofluid biomarkers**

• Blood: Change from baseline up to Week 48 in neurofilament light chain (NfL) concentrations

### **Pharmacokinetics**

- Lu AF82422 plasma concentration during treatment and safety follow-up
- Lu AF82422 cerebrospinal fluid (CSF) concentrations and the CSF/plasma concentration ratios

### 4.4 Safety Endpoints

#### 4.4.1 Double-Blind Period

- Treatment emergent adverse events
- Absolute values and changes from baseline in clinical safety laboratory test values, vital signs, weight, and ECG parameter values
- Development of specific anti-drug antibodies (ADA)
- Findings on MRI, as specified in the *Imaging Charter*
- Columbia-Suicide Severity Rating Scale (C-SSRS) score

### 4.4.2 Open-label Extension Period

- Treatment-emergent adverse events
- Absolute values and changes from baseline in clinical safety laboratory test values, vital signs, and weight parameter values
- Development of specific anti-drug antibodies (ADAs)
- Columbia-Suicide Severity Rating Scale (C-SSRS) score

### 4.5 Exploratory Endpoints

### 4.5.1 Double-Blind Period

### **Disease progression**

 as assessed by longitudinal changes from baseline in the abbreviated UMSARS (aUMSARS) score up to EoTDB

### Function

Changes from baseline to Week 48 in aUMSARS

### **Autonomic symptoms**

• Change from baseline to Week 48 in heart rate, blood pressure, and orthostatic symptoms, as assessed in UMSARS Part III

#### **Disease milestones**

- Time to wheelchair use, as assessed by the recording of wheelchair use in the physical examination CRF Form
- Change from baseline to Week 48 in frequency of falls, as assessed by PamSys device
- Change from baseline to Week 48 in gait parameters, as assessed by FeetMe device

### MRI biomarkers

- Percentage change from baseline to Week 48 in cerebral blood flow in ROIs; putamen and cerebellum, as measured by arterial spin labelling (ASL) MRI
- Percentage change from baseline to Week 48 in tissue integrity in ROIs; primary ROIs: putamen, cerebellar cortex and white matter; secondary ROIs: caudate nucleus, globus pallidus and middle cerebellar peduncle, as measured by diffusion-tensor imaging (DTI) MRI

#### **Blood/CSF** biomarkers

- CSF: Change from baseline up to Week 48 in t-tau and NfL concentrations
- CSF: Concentrations of 'free' and 'total' α-synuclein at baseline and Week 48
- CSF: Changes from baseline up to Week 48 in pathological species of α-synuclein
- Blood: Plasma concentrations of 'free' and 'total' α-synuclein during treatment and safety follow-up

### 4.5.2 Open-label Extension Period

Effect on long-term treatment:

- Change from baseline of the DBP and baseline of the OLE to End-of-Treatment of the OLE (EoTOLE) in UMSARS TS and mUMSARS score
- Change from baseline of the DBP and baseline of the OLE to EoTOLE in CGI-S score
- Change from baseline of the DBP and baseline of the OLE to EoTOLE in PGI-S score
- Change from baseline of the DBP and baseline of the OLE to EoTOLE in SE-ADL score
- Change from baseline of the DBP and baseline of the OLE to EoTOLE in health-related quality of life, as assessed using EQ-5D-5L score
- Percentage change from baseline of the DBP and baseline of the EoTOLE in brain atrophy in ROIs, as measured using vMRI
- Change from baseline of the DBP and baseline of the OLE to EoTOLE in blood NfL concentrations

# 5 Analysis Sets

The patients will be assigned to analysis sets based on IMP intake and post-baseline assessments of the primary efficacy variable in the Treatment Period.

The following analysis sets will be used for the analyses:

- all-patients-randomized set (APRS) all randomized patients
- *all-patients-treated set* (APTS) all patients in the APRS who took at least one dose of double-blind IMP
- *full-analysis set* (FAS) all patients in the APTS who had a valid baseline assessment and at least one valid post-baseline assessment of the UMSARS TS, prior to, or at withdrawal from treatment
- *PK sub-set* (PKS) all patients in the APTS with quantifiable plasma or CSF concentration of Lu AF82422
- Sensor-based subset (SBS) all patients in the APTS who consented to wear at least one of the included sensor-based devices and who had a valid baseline assessment and at least one valid post-baseline assessment, where 'valid assessment' covers that gait parameters can be derived within the observation period
- Exit Interview subset all patients in the FAS having a complete Exit interview with the patient and/or the caregiver
- *Study Experience subset* all patients in the FAS having a complete Study Experience interview with the patient and/or the caregiver
- Open-label treatment extension set (OLES) all patients in the FAS who consented to participate in the OLE and who had at least one dose of Open-Label IMP for the OLE

All data from the Placebo-controlled Period will be cleaned and the database for the DB-Period will be locked when there are no more patients in the DB-Period. The patients and data will be classified into the analysis sets according to these definitions at a Classification Meeting held after the database containing all efficacy measures from the DB-Period has been released but before unblinding of the study.

Demographics, baseline characteristics and baseline efficacy variables will be summarized based on the APTS and on the OLES, respectively.

The efficacy analyses for the DB-Period will be based on the FAS. Analyses for the Extension Period will be based on the OLES.

Safety outputs (including exposure and concomitant medications) will be based on APTS in the DB-Period and OLES for the Extension Period, respectively. Relevant safety outputs for data collected during the Safety Follow-up Period for participants not entering the OLE will be based on the APTS.

Listings will be based on the APTS.

# **6** Descriptive Statistics

Unless otherwise specified, summary statistics (n, arithmetic mean, standard deviation [SD], median, lower and upper quartiles, minimum and maximum values) will be presented for continuous variables, and counts and, if relevant, percentages will be presented for categorical variables. Shift-tables will be presented for categorical variables where specified.

Unless otherwise specified, data listings will include site, treatment group, patient number, sex, age, region and race.

# 7 Patient Disposition

### 7.1 Summary of Patient Disposition

Patient disposition will be summarized overall and by region. Summaries will include the number of patients in each analysis set defined in chapter 5, and the number of patients in the APTS who completed or withdrew from study.

The number of patients with a completed OLE and Safety Follow-up visit will be presented.

### 7.2 Withdrawals

The number of patients who withdrew from the study will be summarized by primary reason for withdrawal and all reasons for withdrawal by period.

If relevant, Kaplan-Meier failure plots of time to withdrawal will be presented by treatment group for the DB-Period. The time will be calculated from the date of first dose of IMP to the date of withdrawal in the DB-Period. Patients who completed the DB-Period according to their individual treatment duration (48-72 weeks) will be regarded as censored at the End of treatment visit.

Patients who withdrew from the study will be listed and the listing will include the number of days in the study until withdrawal, the number of days on IMP, the primary reason for withdrawal, and all reasons for withdrawal.

All tables, graphs, and listings will be based on the FAS.

# 8 Demographics and Baseline Characteristics

Demographics (sex, age, race, region), Screening MRI findings supporting MSA diagnosis and CCl ; baseline disease characteristics (incl. MSA sub-type, CSF/blood NfL level, result from the qualitative alpha-synuclein seeding assay (SAA), time since symptom onset and diagnosis); baseline physical examinations and baseline efficacy variables will be summarized by treatment group and overall.

Study 18331A - Statistical Analysis Plan

Page 16 of 96

Concurrent as well as relevant past medical and psychiatric disorders will be coded using the *Medical Dictionary for Regulatory Activities* (MedDRA) and summarized.

A concurrent medical or psychiatric disorder is a disorder that is ongoing at the baseline Visit. A past medical or psychiatric disorder is a disorder that ended prior to the baseline Visit.

Demographics and baseline characteristics will be summarized based on the APTS, PKS and SBS, and baseline efficacy variables will be summarized based on the FAS.

## 9 Recent and Concomitant Medication

Recent and concomitant medication will be coded using the *WHO Drug Dictionary* (WHO-DDE).

Medications will be classified according to the start and stop time and summarized by anatomical therapeutic chemical (ATC) code, and generic drug name:

- medication discontinued prior to first dose of IMP
- concomitant medication continued after first dose of IMP
- concomitant medication started at or after first dose of IMP

In addition, concomitant medications continued or started after first dose of IMP will classified into two overall groups depending on purpose, i.e., treatment of motor symptoms ('anti-Parkinson medication') and treatment of autonomic dysfunction ('Autonomic dysfunction medication'). The classification will be done prior to unblinding according to Protocol Appendix VII.

The tables will be based on the APTS.

# 10 Exposure

For each infusion visit, information related to infusion completed as planned (yes/no), infusion temporarily interrupted (yes/no), and infusion lasted longer than 30 (+10) minutes (yes/no), as well as descriptive statistics for the duration of infusions (this duration includes duration of any infusion interruptions) and duration of temporary interruptions will be summarized by treatment group for the DB-Period and the OLE-Period, respectively.

Patients, who at any point during the study received a different dose than what was planned, will be listed for each period. The listing will include date of infusion visit, planned dose for the patient and actual dose received for the patient.

Exposure (days) to IMP will be calculated as: (Date of last dose + 28 days) – Date of first dose + 1

Exposure to IMP will be summarized in weeks using descriptive statistics.

Patient years of exposure (PYE) will be calculated as the sum of the number of days of exposure to IMP for each patient, divided by 365.25 days.

The number and percentage of patients with different durations of exposure ( $\leq$ 4 weeks, >4 to  $\leq$ 8 weeks, >8 to  $\leq$ 12 weeks, ..., >68 to  $\leq$ 72 weeks) will be presented.

Exposure will be summarized based on the APTS. In addition, all infusion data will be listed.

# 11 Fall Diary Compliance

The Fall Diary is planned to be dispensed and filled out in 5 periods during the study, i.e., at a two-week Baseline period and at four post-baseline four-week periods, respectively. For each period, days where the fall diary has been missed will be summarized and presented by period and treatment group. Furthermore, the number of patients missing 7 days or more (at Baseline and at subsequent periods) and 14 days or more (at subsequent periods) in each period will be presented by period and treatment group.

A day where the fall diary has been missed is defined as a day where the subject did not fill out anything in the diary.

The summaries will be based on the FAS.

# 12 Wearable Compliance

For both Baseline and the DB-Period, compliance is evaluated as number of days used for each of the two wearables, i.e., FeetMe and PanSys, which will be summarized within each interval where applied and treatment group. Furthermore, the number of patients missing 7 days or more and 14 days or more in a 28-day period will be presented by interval and treatment group. The following intervals will be evaluated:

- BL interval: V2 to V3 (2 weeks)
- Interval 1: V7 to V9 (4 weeks)
- Interval 2: V10 to V11 (4 weeks)
- Interval 3: V13 to V14 (4 weeks)
- Interval 4: V17 to V18 (4 weeks)

Records outside the above predefined intervals will be included as long as they can be mapped to one of the above intervals according to the defined visit windows (See section 24.2). Individual wearable data will be mapped to the end visit defining each interval, corresponding to the visit where the wearable is handed back.

The summaries will be based on the SBS.

# 13 Primary Estimand

The following primary estimand is defined as:



# Proposed handling of IE's



For evaluating the appropriateness of this overall strategy, a number of sensitivity analyses will be performed using different imputation strategies for missing data. For additional information see section 14.3.5: Sensitivity Analyses of the Primary Endpoint, also covering sensitivity analyses for the key Secondary Endpoint.

## **Key Secondary Estimand**

A key secondary study estimand will be defined in a similar manner with the endpoint of interest being the CCI

# 14 Efficacy

# 14.1 Overview of Planned Efficacy Analyses in the DB-Period

An overview of all planned efficacy analyses is provided in Panel 2. Where relevant, the analyses will be presented by visit. Endpoints related to as 'disease progression' (primary and selected secondary endpoints) will be analysed using a 'Bayesian' progression model; remaining continuous variables will be analysed applying a MMRM in a Frequentist framework, where stated.

Panel 2 Overview of Planned Efficacy Analyses (DB-Period)

| Variables | Type | Priority | Description |
|---|---|---|---|
| UMSARS TS | 1 | 1 | Sum of UMSARS Part I+II items (Primary) |
| mUMSARS score | 1 | 2 | Sum of Part I items with respond option 0 and 1 collapsed |
| UMSARS Part I score | 1 | 3 | Sum of UMSARS Part I items |
| UMSARS part II score | 1 | 3 | Sum of UMSARS Part II items |
| aUMSARS score | 1 | 4 | Sum of UMSARS Part I+II selected items - PI: 1,3,4,7,8 & PII: 2,6,8,11,14 |
| SE-ADL score | 2 | 3 | Schwab and England Activities of Daily Living scale: sum of items |
| CGI-S score | 2 | 3 | Global impression severity, Clinical: sum of items |
| PGI-S score | 2 | 3 | Global impression severity, Patient: sum of items |
| OGI-S score | 2 | 3 | Global impression severity, Observer-reported: sum of items |
| COMPASS select change | 2 | 3 | Composite autonomic symptom: a score for each domain |
| UMSARS part III items | 2 | 4 | Heart rate, sys/dia blood pressure; individual items |
| UMSARS part III items | 3 | 4 | orthostatic symptoms; individual item |
| UMSARS part IV item | 3 | 3 | Global disability: UMSARS single item |
| UMSARS part I items | 3 | 3 | Disease milestones: Speech, swallowing, walking and falls; UMSARS Part I single items |
| Patient fall diary | 3 | 3 | Disease milestones: Frequency, cause and consequence of falls; patient dairy derived |
| Use of wheelchair | 4 | 4 | Disease milestones: Wheelchair – time to full time user; according to physical examination |
| PamSys digital device | 3 | 4 | Disease milestones: Frequency of Falls; PamSys derived |
| FeetMe digital device | 2 | 4 | Disease milestones: gait parameters; FeetMe derived |
| EQ-5D-5L items | 3 | 3 | Health-related quality of life: domain scores |
| EQ-5D-5L VAS score | 2 | 3 | Health-related quality of life: VAS score |
| MRI, volumetric (vMRI) | 2 | 3 | volume in ROIs (e.g., caudate nucleus, putamen, striatum, pons, brain stem, grey matter and cerebellum) |

| Variables | Type | Priority | Description |
|---|---|---|---|
| MRI, diffusivity (DTI MRI) | 2 | 4 | Mean diffusivity in ROIs (e.g., caudate nucleus, putamen, globus pallidus, pons, cerebellar cortex and white matter and middle cerebellar peduncle, both FA and MD) |
| Blood biomarkers | 2 | 3, 4 | neurofilament light (NfL) concentrations [2], 'free' and 'total' $\alpha$ -synuclein [3] |
| CSF biomarkers | 2 | 4 | concentrations of t-tau, NfL, 'free' and 'total' $\alpha$ -synuclein, pathological species of $\alpha$ -synuclein |
| MRI, arterial spin (ASL) | 2 | 4 | Mean Cerebral blood flow in ROIs (e.g., putamen and cerebellum) |

Type: 1 = continuous\_Bayes; 2 = continuous\_Other; 3 = categorical; 4 = time to event; Priority: 1 = Primary; 2 = Key Secondary; 3 = Secondary; 4 = Exploratory

### 14.2 General Efficacy Analysis Methodology

Unless otherwise specified, all efficacy analyses will be based on the FAS for the observed case (OC) data.

For endpoints analysed in the Bayesian framework, the success threshold for the Bayesian posterior probability of superiority relative to placebo [Prob( $\theta$ <1)] has been calibrated using simulations to correspond to a significance level of 5% applied one-sided. By doing so a success threshold of 0.975 has been identified which will be used to evaluate the primary endpoint and remaining endpoints evaluated by the Bayesian progression model. A burn-in of 1000 samples will be used for the Bayesian analysis.

All statistical tests of the secondary efficacy endpoints will be presented two-sided on a 5% significance level.

A testing strategy will be applied including the primary analysis on UMSARS TS and the key secondary analysis on mUMSARS to protect the type I error on an overall one-sided 5% significance level for these analyses. Further details to be found in chapter 15.

For analysis of exploratory efficacy data collected in the open-label extension, the original placebo patients will be presented as a separate group and hence there will be no pooling of treatment groups.

### 14.3 Analysis Methodology for the Primary Endpoint

### 14.3.1 Primary Analysis of the Primary Endpoint

The primary efficacy analysis following up to 72 weeks of treatment will be based on a Bayesian repeated measures model, also referred to as a Bayesian functional-impairment

progression model (BFPM), of the changes from baseline in the UMSARS TS. The BFPM incorporates the following aspects:

- Repeated measures for the change from baseline in the UMSARS TS score over the recurring 72-week's visit schedule
- Piece-wise linear rate of progression per 12-week time interval. However, does not require equally spaced intervals between observations. Time modelled continuously
- Patient-level random effect in rate of progression
- Proportional treatment effect,  $\theta$ , for slowing of disease progression rate when treated relative to placebo. In particular, if  $\theta$ <1, the active treatment slows the rate of progression relative to placebo. If  $\theta$ >1, the active treatment increases the rate of progression relative to placebo. If  $\theta$ =1, the rate of progression of UMSARS TS is the same for both active treatment and placebo
- Fixed multiplicative covariate effects in the increase or decrease in the overall rate of progression of UMSARS TS for categorized CCI and region (US and Japan) common across all visits
- Prior distributions for model parameters selected in a conservative and non-informative manner using relatively large outcome spaces
- The primary analysis considers only actual observations and does not impute missing data

Let change from baseline in the UMSARS TS at visit j for subject i be labelled  $Y_{i,j}$ , i = 1, ..., N,  $j = 1, ..., J_i$  where there are  $J_i$  total post-baseline visits for subject i. Change from baseline will be modelled as piece-wise linear with time intervals, k = 1, ..., K, defined every 12 weeks. Let  $X_{i,j,k}$  be the exposure (time since baseline in weeks) for subject i at visit j during the time interval k. The MSA progression model is:

$$\begin{split} Y_{i,j} \sim & N \left( \mu_{i,j}, \sigma_{t(i)}^{2} \right); i = 1, \dots, N; j = 1, \dots, J_{i} \\ \\ \mu_{i,j} = 0 + \sum_{k=1:K} \left( \beta_{k} + \beta_{k,i} \right) * \left( X_{i,j,k} / 12 \right) * \theta_{t(i)} * \exp \left( \delta_{g(i)} + \eta_{r(i)} \right) \end{split}$$

where each parameter is defined below and the prior distribution for the parameter is given:

 $\beta_k$ : Mean expected change from baseline over each 12-week interval

$$\beta_k \sim Norm(0.10^2); k = 1, ..., K$$

 $\beta_{k,i}$ : Subject-level additive random effect in change from baseline over each 12-week interval for subject i

$$\beta_{k,i} = \beta_i; \ \beta_i \sim Norm(0, \sigma_{\beta}^2); \ \sigma_{\beta} \sim Unif(0,20)$$

 $\theta_t$ : Multiplicative proportional slowing in rate of progression for treated (t=2) relative to placebo (t=1).

$$\theta_1 = 1$$
;  $\theta_2 \sim Unif(0,2)$ 

 $\delta_g$ : Multiplicative fixed covariate effects for the increase or decrease in rate of progression for plasma NfL level, i.e., missing (g=3) and high (g=2) relative to low (g=1) common across all visits

$$\delta_1 = 0$$
;  $\delta_2 \sim Normal(0,10^2)$ ;  $\delta_3 \sim Normal(0,10^2)$ 

 $\eta_r$ : Multiplicative fixed covariate effects for the increase or decrease in rate of progression for regions, i.e., Japan (r=2) relative to US (r=1) common across all visits

$$\eta_1 = 0$$
;  $\eta_2 \sim Normal(0.10^2)$ 

 $\sigma_t$ : Measurement error per treatment arm

$$\sigma_t \sim Unif(0,10); t = 1,2$$

The  $\theta_t$  parameters represent the multiplicative proportional slowing in rate of progression for treated relative to placebo (t=l); also referred to as the functional-impairment progression rate ratio (FPRR). For placebo, the FPRR is assumed to be 1 ( $\theta_1$  = 1). Thus, the FPRR parameter for treatment (Lu AF82422) represents the multiplicative change to the mean progression of a placebo patient. If the FPRR is less than 1 then the progression for treatment t is slower than for placebo. A value of FPRR = 0.75 corresponds to a 25% slowing in progression and a value of 0.25 represents a 75% slowing in progression. The errors for the individual observations are modelled as independent normal distributions with a standard deviation of  $\sigma$ .

### 14.3.2 Posterior Summaries

The Bayesian posterior distributions of all model parameters are calculated using Markov chain Monte Carlo (MCMC). The algorithm allows the generation of at least M=100,000 draws from the joint posterior distribution for all model parameters. In particular, summaries of the Bayesian posterior distribution for the effect of Lu AF82422 compared to placebo,  $\theta_2$ , will be provided including the mean, median and 95% credible intervals together with the probability that the active dose is superior to placebo,  $Pr(\theta_2 < 1)$ . In addition, the probability of at least a 20% slowing effect will be presented,  $Pr(\theta_2 < 0.8)$ , and the probability of at least a 30% slowing effect will be presented,  $Pr(\theta_2 < 0.7)$ .

Finally, summaries of the Bayesian posterior distribution for the remaining model parameters will be provided including the mean, median and 95% credible intervals.

### 14.3.3 Rationale for Selected Analysis Method for the Primary Endpoint

It is believed, that applying the Bayesian progression model is an appropriate and powerful way of analysing MSA disease progression data in this context, since:

- The Bayesian methodology provides relatively simple computational and interpretable posterior probabilities for decision-making. In addition, it offers a robust performance in relation to convergence, as well as consistency across the performed analyses.
- There is a strong indication based on available 12-24 months MSA progression data<sup>1</sup> (i.e., UMSARS total and part I scores) of a steep and nearly linear disease progression trajectory; especially for the earlier patient segment, making it meaningful to talk about a change in the slope or a slowing down of progression.
- Due to the parametrization of effect expressed common across all visits, the model offers an easy interpretable target of estimation being the percentage-wise slowing in progression through up to 72 weeks treatment for Lu active dose compared to placebo.
- Based on the Lu AF82422 hypothesized mechanism of action, an early trend in UMSARS in favor of Lu AF82422 is reasonable due to the expected immediately steep MSA progression curve. Furthermore, the UMSARS is assessed for the first time at Week 12 following multiple dosing allowing time for initial treatment manifestation. Assuming that such an early trend will be further substantiated over time in a proportional-like manner due to the hypothesized moderation of the MSA pathology by Lu AF82422 (i.e., inhibition of seeding of pathological form(s) of alpha-synuclein, inhibition of the C-terminal proteolytic cleavage of alpha-synuclein, and potential immune-mediated clearance of alpha-synuclein/mAb complexes by the active Fc region), it seems less likely that the effect will significantly wear-off within the up to 72 weeks treatment period.
- The progression model is better suited for handling individual differences in treatment duration (i.e., when having differences in treatment duration due to the study design or a notable number of drop-outs/deaths); despite incomplete data (<72 weeks), a slope can still be estimated making full use of all patients. In particular, the long duration of the study (48-72 weeks) makes it more relevant to consider the effect integrated over time instead of the change from baseline for a single chosen timepoint.
- The progression model is well suited for handling also differences between visits due to the study design, where all ongoing patients will be called in for their respective end-of-treatment visit when the last patients randomized has completed 48 weeks of treatment.
- For treatment effect, the prior has been selected uniformly within [0, 2] for the active arms compared to placebo. In this way the prior is centred around no effect, i.e.,  $\theta_t = 1$ , with  $\theta_2 < 1$  referring to a slowing in progression, and  $\theta_2 > 1$  referring to an increase.
- Remaining priors have been selected in a conservative and basically 'non-informative' manner by using relatively large outcome spaces. For the fixed effects of visit,  $\beta_j$ , a normal distributed prior centred around zero with a variance of 100 has been selected, since between-visit changes in the UMSARS scale can be both positive and negative with a relatively high variability. However, due to the rather aggressive disease progression observed within MSA, it is expected that the cumulated sums of  $\beta_j$ 's are positive leading to an interpretation of  $\theta_2 < 1$  being an improvement.

- For the subject-level effect a fairly simple parametrization has been selected by assuming these to be random with a uniformly shaped hyper-prior on the standard deviation within [0, 20]. In this way the covariance structure is assumed to be relatively simple.
- Since used for stratification, CC and study region, respectively, will be accounted for by including as multiplicative fixed covariate effects parametrized on the logarithmic scale. For both parameters, a reference level will be set to zero and for the remaining level(s) a normally distributed prior will be selected centred around zero (for no difference) with a variance of 100. In this way the effect can go in either direction with little restriction on the size.
- The model has shown little bias in the treatment estimate for the selected scenarios.
   Additionally, under various formulations of the null hypothesis the model has with the chosen thresholds shown to adequately control the type 1 error on an overall 5% significance level evaluated 1-sided and has attractive type II error control under the alternative.
- It is already an established approach within other neurodegenerative diseases (e.g., AD<sup>2</sup>,<sup>3</sup>) and within diseases that cause progressive weakness and loss of muscle mass (e.g., Duchenne muscular dystrophy<sup>4</sup> or GNE myopathy<sup>5</sup>) to model disease progression and show changes to expected disease deterioration as a change in the slope of progression.

To evaluate the appropriateness of the proposed progression model and the underlying assumptions, a number of sensitivity analyses will be conducted, incl. a MMRM to evaluate consistency across models especially in relation to how effect matures over time. Such approach will also be used to evaluate potential bias in effect estimates. See 14.3.5 Sensitivity Analyses of the Primary Endpoint for further details.

# 14.3.4 Evaluation of Model Assumptions for the Primary Analysis of the Primary Endpoint

The following goodness-of-fit diagnostics will be performed to assess the goodness-of-fit of the Bayesian primary repeated measures analysis:

- Residual plots for UMSARS TS: residuals vs. fitted values of UMSARS TS at each visit and for each treatment group.
- Mean and SD in change from baseline of UMSARS TS at each 12-week visit for each treatment group compared to model fitted expected values from primary analysis model.

### 14.3.5 Sensitivity Analyses of the Primary Endpoint

### **Handling of Missing Data**

The following sensitivity analyses will be performed in case of drop-out/withdrawal/death, where the below rules will be applied for the visit following the event for subjects not having

complete data from the Withdrawal Visit, assuming that intermediate missingness will be 'missing at random':

- For withdrawal due to death, impute individual missing UMSARS items as worst possible score in case of death.
- For withdrawal due to other reasons, impute individual missing UMSARS items as worst observed within-subject value for the specific item at any post-IMP time point.
- For withdrawal due to other reasons, impute individual missing UMSARS items as the
  worst value observed within the combined treatment and control arms at any post-IMP
  time point.

Two analyses will be performed in both cases using the above strategy to handle withdrawal due death. Following each of the above strategies for handling withdrawals due to other reasons will then be applied.

To explore further the impact of death, a non-parametric joint-rank analysis will be performed to account for informatively missing data by ranking patients based jointly on their Week 48 UMSARS score (UMSARS TS and mUMSARS) and 48-week survival, i.e., time-to-death. Such analysis corresponds to a composite strategy. In case of missing Week 48 data for survivors, Multiple Imputation (MI) will be performed in which the remaining missing data will be imputed corresponding to a missing-at-random assumption.

Missing data for UMSARS Week 12 up to Week 48 will be addressed by using Multiple Imputation. Missing data will be imputed using a sequential regression-based multiple imputation method, based on the imputation models established from the corresponding randomized treatment group. Example SAS code for this imputation can be found in Appendix II.

200 imputed datasets will be created, which will each be analysed and combined as follow.

Define score,  $u_{ij}$ , which is chosen to reflect whether patient i has had the more favourable UMSARS score than patient j. In the case where both patient i and j died prior to the Week 48 assessment:

- $u_{ij} = 1$  in the case where patient i died after patient j
- $u_{ij} = -1$  in the case where patient i died before patient j
- $u_{ij} = 0$  in the case where it cannot be determined who died first

In the case where patient i died prior to the Week 48 assessment, and patient j has not died prior to the Week 48 assessment:

• 
$$u_{ij} = -1$$

In the case where patient i did not die prior to the Week 48 assessment, and patient j died prior to the Week 48 assessment:

• 
$$u_{i,i} = 1$$

In the case where both patient i and patient j are alive at Week 48 assessment:

- $u_{ij} = -1$  when UMSARS score for patient i at Week 48 > UMSARS score for patient j at Week 48
- $u_{ij} = 1$  when UMSARS score for patient i at Week 48 < UMSARS score for patient j at Week 48
- $u_{ij} = 0$  when UMSARS score for patient i at Week 48 = UMSARS score for patient j at Week 48

Using the  $u_{ij}$  for every pair of patients defined above, a score is assigned to each subject,  $U_i = \sum_{i \neq i} u_{ij}$ .

A t-test is applied to the  $U_i$  scores to compare the treatment groups. The estimated mean difference and associated SE from each of these analyses will be combined using Rubin's Rule. The p-value from this combined analysis will be presented.

### **Assumptions of Primary Efficacy Model**

The following analyses will be conducted to test the sensitivity of the results to the primary efficacy model assumptions:

- The Bayesian repeated measures primary analysis model will be explored for sensitivity to priors by using a sceptical alternative for  $\theta_2$ , i.e., using a PERT distribution with mode 1.1 and a shape of 7.44 corresponding to a prior that Lu AF82422 is doing 60% worse than placebo.
- The UMSARS TS will be analysed using a restricted maximum likelihood (REML)-based mixed model for repeated measures (MMRM). The model will include the following: region, CCl and treatment (Lu AF82422 and placebo) as fixed factors, baseline UMSARS TS as continuous covariate, treatment-by-week interaction and baseline UMSARS TS-by-week interaction. An unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom. The analysis will be performed using all available observations (observed cases [OC] data) in the DBP. The estimated treatment differences between Lu AF82422 and placebo obtained at Week 48 will be estimated based on the least squares means for the treatment-by-week interaction in the MMRM model. Estimated treatment differences at Week 60 and 72 will be exploratory. In case of issues converging, a Toeplitz structure will be fitted instead.
- A constrained longitudinal data analysis with natural cubic splines that treats time as continuous, which allows separate splines for each treatment (Donohue et al, 2023)<sup>6</sup>. The natural cubic spline model assumes:

$$Y_{i,j} = \beta_0 + \sum_{k=1:m} (\beta_k \cdot b_k(t_j)) + Active_i \cdot \sum_{k=1:m} (\gamma_k \cdot b_k(t_j)) + \varepsilon_{ij},$$

where  $b_k(t)$  are the known spline basis functions for a given set of knots and extreme values of t, with Interior knots spaced according to quantiles of t. The resulting curve for the placebo group is defined by the natural cubic spline  $f(t) = \beta_0 + \sum_{k=1:m} (\beta_k \cdot b_k(t_j))$ ; while the natural cubic spline  $g(t) = \sum_{k=1:m} (\gamma_k \cdot b_k(t_j))$  represents the treatment group difference over time and is constrained to be zero at time zero. Estimation of the unknown parameters ( $\beta$ s and  $\gamma$ s) is accomplished with maximum likelihood estimation. It is to be noted, that a special case of the spline parameterization with visit times set to the planned times and knot locations chosen to match the planned visit times is equivalent with a categorical-time mean structure as found in the MMRM.

In fitting the model, the basis for the natural cubic splines is generated using the SAS® code given in the Appendix II.

### 14.3.6 Subgroup Analyses of the Primary Endpoint

Subgroup analyses of the primary endpoint will be performed using the Bayesian repeated measures primary analysis model for the following subgroups:

- Use of concomitant medication (categorised into PD and autonomic dysfunction medication according to chapter 9). Two analyse will be performed: 1) where concomitant medication was already started up prior to baseline and continued after baseline, and 2) where concomitant medication was initiated or change in dose of existing medication after baseline
- Presence of MRI abnormalities at Screening supporting the diagnosis of MSA (i.e., 'yes' to at least one of the MRI abnormalities according to Screening MRI procedure)
- MSA sub-group (MSA-P and MSA-C)
- Pre-dose MSA positive result in the qualitative alpha-synuclein seeding aggregation assay (SAA), i.e., positive for alphaSyn seed amplification pattern predominantly found in subjects with MSA

### 14.3.7 Covariate Analyses of the Primary Endpoint

- age (categorized as <50yrs; 50-60; >60yrs)
- gender (female/male)
- race
- time-since-symptom onset (as yearly intervals)

- baseline plasma/CSF alpha-synuclein and CSF NfL (defined as baseline lower/middle/upper tertile)
- baseline disease severity according to category of CGI-S and UMSARS part IV (global disability score 1-5), and SE-ADL (defined as baseline lower/middle/upper tertile)

### 14.4 Analysis of the Secondary Endpoints

### 14.4.1 Analysis Methodology for the Key Secondary Endpoint

• For the key secondary endpoint, i.e., the changes in mUMSARS from baseline up to EoTDB, a Bayesian repeated measures model will be applied similar to the primary analysis.

Sensitivity analyses to the key secondary analysis will be set up similar to the sensitivity analyses described for the primary endpoints under section 14.3.5 Sensitivity Analyses of the Primary Endpoint(s).

### 14.4.2 Analysis Methodology for the Secondary Endpoint

- For the UMSARS Part I, UMSARS Part II and the aUMSARS, a similar Bayesian progression model and estimand strategy to the primary analysis will be applied.
- For remaining continuous secondary endpoints (e.g., clinical scales/assessments and MRI parameters), the change from baseline to EoTDB will be analysed using a restricted maximum likelihood (REML)-based mixed model for repeated measures (MMRM). The model will include the following: region, CCl and treatment (Lu AF82422 and placebo) as fixed factors, baseline as continuous covariate, treatment-byweek interaction and baseline-by-week interaction. An unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom. The analysis will be performed using all available observations (observed cases [OC] data) in the DBP. The estimated treatment differences between Lu AF82422 and placebo obtained at Week 48 will be estimated based on the least squares means for the treatment-by-week interaction in the MMRM model. Estimated treatment differences at Week 60 and 72 will be exploratory. In case of issues converging, a Toeplitz structure will be fitted instead.
- Categorical secondary endpoints will be evaluated using shift-tables evaluated at Week 48.
- Adjusted number of falls per individual per fall diary period in the DBP, according to the patient fall diary, will be analysed applying a MMRM as described above, if appropriate. Cause and consequence of falls will be evaluated descriptively.
- Time-to-wheelchair endpoint as assessed in the physical examination (first time point as 'full time user') following up to 72 weeks of treatment will be presented by a Kaplan-Meier plot and analysed applying a Cox proportional-hazards model. The model will be adjusted for stratification factors.
- Lu AF82422 plasma concentrations, CSF concentrations, and the CSF/plasma concentration ratios during treatment for all patients will be presented descriptively. A

- population pharmacokinetics analysis (popPK) will also be performed and included in a separate reported.
- Absolute values and changes from baseline to EoTDB in blood and CSF biomarkers will be analysed descriptively (i.e., NfL, t-tau, truncated alpha synuclein). A MMRM will be applied for the changes from baseline to EoTDB. If required, a log transformation will be applied for normalization.
- TE of Lu AF82422 to α-synuclein in plasma and CSF will be presented descriptively as 'free' α-synuclein, 'total' α-synuclein and ratio of 'free' to 'total' α-synuclein. In addition, TE will be plotted vs. concentration of Lu AF82422 to characterize the relationship.
- Results from the semi-quantitative alpha synuclein seeding assay (SAA), i.e., the SD50 representing the time to reach 50% max, will be presented descriptively over time.
- Gait and balance parameters derived from the sensor based FeetMe® device will primarily be analysed descriptively for the SBS. a MMRM model, like the one described above for continuous secondary and exploratory endpoints, will be applied to the change from baseline. Correlation to the key progression markers, that is the UMSARS scores and MRI parameters, will be explored graphically using scatterplots.

### 14.5 Additional Analyses of Primary and Secondary Endpoints

A number of additional analyses is planned to evaluate the relationship between the primary and selected secondary/exploratory endpoints:

- Relationships between selected continuous endpoints, i.e. UMSARS total score and subdomains, MRI, blood/CSF NfL, α-synuclein, COMPASS-S/SC, CGI-S, PGI-S, SE-ADL, gait parameters and EQ-5D-5L VAS will be explored using scatterplots for both absolute values and change from baseline.
- The minimal clinically important difference within-patient (MCID) on each scale will be investigated. Further details on the work identifying the MCID will be described in a specific separate *Psychometric SAP*. The outcome of the MCID analysis will be reported in a separate report.

### 14.6 Analysis of Exploratory Endpoints

For exploratory endpoints the following methodology will be applied:

- For continuous exploratory endpoints, a MMRM will be applied for observed data (OC), using observed data from the Withdrawal Visit for patients dropping out (for other reasons than death), if available. The model will contain the following effects: baseline score, treatment, visit, CCl Region, treatment\*visit and baseline score\*visit as fixed effects and subject as random effect. The main comparison will be at Week 48. Initially, an unstructured covariance matrix will be fitted. In case of issues converging, a Toeplitz structure will be used.
- Time-to-event exploratory endpoints up to EoTDB will be analysed applying a Cox proportional-hazards model.

- Number of falls per individual according to the sensor-based PAMSys device will be analysed descriptively including data from the pre-defined periods only.
- Target engagement and biofluid markers in general will primarily be explored graphically. If applicable, relevant efficacy endpoints will be evaluated especially for patients obtaining target engagement.
- The analysis of Screening and Exit semi-structured, qualitative interviews will be prespecified in a specific Qualitative Analysis Plan (QAP). Whenever a combined quantitative and qualitative approach is considered, a dedicated Mixed Method QAP will be developed.

### **Open-label extension (OLE)**

• All continuous endpoints following treatment extension will primarily be analysed descriptively. In addition, a MMRM will be applied similar to the one described above to the change from the original baseline (DB baseline), where patients originally treated with pbo will be kept as a separate group. No formal testing will be applied.

# 15 Testing Strategy

### 15.1 Calibrating primary analysis

The final analysis will use all available data on all enrolled participants at baseline through 48-72 weeks. A success threshold is defined for the final analysis to maintain an overall alpha of 5% evaluated one-sided. The effect of Lu AF82422 will be evaluated using a Bayesian posterior probability of superiority relative to placebo with a threshold of 97.5% identified through simulations.

Lu AF82422, CCI dose: 
$$Pr(\theta_2 < 1) > .975$$
;

### 15.2 Testing Strategy including Secondary Endpoint(s)

To protect the type I error for the primary analysis, i.e., analysis of UMSARS TS and the key secondary analysis, i.e., analysis of mUMSARS, both using the Bayesian progression model, a testing strategy will be applied. Firstly, both endpoints will be evaluated individually by applying the pre-defined threshold to the posterior probability for Lu AF82422 being superior to placebo, where the thresholds have been calibrated to be equivalent to the targeted 5% significance level evaluated one-sided. Following, the Fixed-Sequence Method will be applied evaluating the two prioritized analyses in a hierarchical manner:

- Step 1: UMSARS TS evaluated using the derived posterior probability (test equivalent to a one-sided 5% level). If significant,
- Step 2: mUMSARS evaluated using the derived posterior probability (test equivalent to a one-sided 5% level).

# 16 Safety

### 16.1 Adverse Events

### 16.1.1 General Methodology for Adverse Events

Unless otherwise specified, tables, graphs, and listings will be based on the APTS.

Tables by preferred term and tables by system organ class (SOC) and preferred term (PT) will be sorted in descending order based on the percentages of patients with these adverse events.

Unless otherwise specified, the summaries of adverse events will include the number and percentage of patients with an adverse event, and the total number of events.

In summaries of TEAEs by preferred term and intensity, and in summaries of causally related TEAEs by preferred term and intensity, the maximum intensity for the preferred term within an analysis phase will be used.

Listings of adverse events will be sorted by site, patient number, and adverse event start date, and will include preferred term, investigator term, adverse event start date, end date,, duration of the adverse event, date of death, action taken, causality, intensity, seriousness, and outcome. For adverse events that change in intensity, each intensity will be included.

### **16.1.2** Coding of Adverse Events

Adverse events will be coded using MedDRA, Version 26.0 or later.

### 16.1.3 Classification of Adverse Events

Adverse events will be classified according to the date of onset (or worsening of intensity/seriousness) of the adverse event and end date as follows:

- pre-treatment adverse event an adverse event that starts (or worsens) on or after the date the patient signed the *Informed Consent Form* and prior to the date and time of first dose of IMP
- treatment-emergent adverse event (TEAE) an adverse event that starts (or worsens) on or after the date of first dose of IMP

An adverse event is considered causally related to the use of the IMP when the causality assessment by the investigator is probable or possible.

Data handling of change in intensity or seriousness of adverse events is described in section 24.5.2.

### 16.1.4 Allocation of TEAEs to Study Periods

TEAEs will be assigned to periods according the following:

- Adverse events in the double-blind period (DBP) all TEAEs with date of onset or worsening of intensity/seriousness after first dose of IMP in the DBP and until first dose of IMP in the OLE period (planned for Visit 1E for patients entering the OLE) or the Safety Follow up visit for the DBP (SFU Visit 25 for patients NOT entering the OLE) (assigned APHASE = DOUBLE BLIND).
- Adverse events in the Open-Label Extension period TEAEs with date of onset or worsening of intensity/seriousness after first dose of IMP in the OLE period (Visit 1E) and until the final Safety Follow up visit for the OLE (Visit 64E) (assigned APHASE = OLE).

The above imply that an adverse event, with multiple levels of intensity/seriousness, may be reported for more than one phase but only if it worsens. For instance, an adverse event ongoing at the end of the End-of-Treatment (EoT) visit which worsens after the first dosing in the OLEP, will be reported both for the double-blind period (DBP) and for the open-label period, but an adverse event ongoing at the EoT visit, which reduces in intensity/severity will only be reported in the DBP.

#### 16.1.5 Presentation of Adverse Events

All adverse events will be listed for the APRS.

An overview of the PYE and number and percentage of patients with TEAEs, serious adverse events (SAEs), or adverse events leading to withdrawal, and of patients who died will be provided based on the APTS for the open-label and safety follow-up period.

For TEAEs, SAEs, and adverse events leading to withdrawal/death, the total number of events will be included.

### 16.1.6 Presentation of Treatment-emergent Adverse Events

For TEAE's, the following summaries will be provided by study period (DBP, OLEP and the safety follow-up periods, if appropriate) for the APTS:

- TEAEs by SOC and preferred term
- TEAEs by preferred term
- TEAEs with an incidence  $\geq$  5% by preferred term
- TEAEs by causality (possible, probable, not related), SOC and preferred term
- TEAEs by intensity (mild/moderate/severe), SOC, and preferred term

The summaries will be provided for the APTS for the study periods.

For TEAEs occurring on the day of dosing after infusion start, TEAEs with missing start times will also be included.

#### 16.1.7 Presentation of Deaths

All the adverse events in patients who died will be listed for the APRS.

#### 16.1.8 Presentation of Serious Adverse Events

All the SAEs will be listed for APRS by study period.

Treatment-emergent SAEs for the APTS will be summarized by:

- SOC and preferred term
- preferred term

# 16.1.9 Presentation of Adverse Events Leading to Withdrawal

All the adverse events leading to withdrawal will be listed for the APRS.

TEAEs leading to withdrawal will be summarized by:

- SOC and preferred term
- preferred term

# 16.1.10 Presentation of Adverse Events Leading to Study Drug Infusion Interruption or Infusion Rate Reduction

All AEs leading to study drug infusion interruption or infusion rate reduction will be listed for the APRS.

TEAEs leading to study drug infusion interruption or infusion rate reduction will be summarized based on APTS by:

- SOC and preferred term
- preferred term

### 16.1.11 Presentation of Adverse Events requiring additional data collection

Treatment-emergent adverse events related to Type I, II and III Hypersensitivity reactions have been defined as study-specific AE's requiring additional data collection. Events considered Hypersensitivity reactions by the Investigator will be collected during the study using a dedicated Hypersensitivity Form.

Summaries will be provided for each period for the APTS for Hypersensitivity Reactions (as reported by the investigator) and for each of the following sponsor defined categories (see Appendix VI).

- TEAEs with a PT within the SMQ of Hypersensitivity (narrow scope)
- TEAEs with a PT 'Cytokine release syndrome'
- TEAEs with a PT within the SMQ Vasculitis (narrow scope) or any of the 15 defined single PTs

Hypersensitivity reactions will be listed by category by the APRS.

### 16.2 General Methodology for Other safety Data

Unless otherwise specified, tables, graphs, and listings will be based on the APTS.

All tables and graphs will be presented by treatment group.

The denominators for the summaries of a given variable will be based on the number of patients with non-missing values at a given visit or during the assessment period.

Descriptive statistics for the safety variables, both absolute values and changes from baseline, will be presented by visit, separately for each period.

The number and percentage of patients with at least one PCS value at any post-baseline assessment time point will be summarized by variable, separately for each period. All available assessments in each period will be included in the evaluation of PCS values.

For patients with post-baseline PCS values, listings will be provided including all the values for those patients for the variable, with flagging of PCS values and out-of-reference-range values.

For vital signs being measures multiple time during a visit values will be presented graphically within visit over time, where the position will be indicated.

All the adverse events in patients with post-baseline PCS values will be listed by treatment group and patient screening number; the listing will include the PCS value, the assessment date, the change from baseline in PCS value, the preferred term for the adverse event, and start date and stop date of the adverse event. The PCS values and adverse events will be listed in chronological order according to assessment date and the start date of the adverse event

### 16.3 Clinical Safety Laboratory Test Data

### 16.3.1 Data Presentation

The PCS criteria used for the clinical safety laboratory tests can be found in Appendix V.

The clinical safety laboratory test values will be presented both in conventional and Système International (SI) units.

### 16.4 Vital Signs and Weight

The PCS criteria used for vital signs and weight are the Lundbeck standard PCS criteria described in SOP\_09978: *GPV – PCS and standard reference values for laboratory investigations, vital signs and ECGs in clinical studies*, version 6, and are also included in Table 4.

#### 16.5 ECG

The PCS criteria used for the ECG parameters are the Lundbeck standard PCS criteria described in SOP\_09978: *GPV – PCS and standard reference values for laboratory investigations, vital signs and ECGs in clinical studies*, version 6, and are also included in Table 5.

In addition to the tables and listings specified in section 16.2, absolute values and changes from Baseline in QTcF will also be summarized categorically by visit and treatment. The categories that will be used are as follows for the absolute QTcF values:

- QTcF interval < 450 msec
- QTcF interval 450 480 msec
- OTcF interval > 480 500 msec
- QTcF interval > 500 msec

The categories that will be used for the change from baseline QTcF values are:

- QTcF interval increase from baseline > 30 msec
- QTcF interval increase from baseline > 60 msec

Furthermore, the number and percentage of patients being classified as having either a normal, abnormal but not clinically significant, abnormal and clinically significant, or not interpretable ECG result based on the overall interpretation of the ECG from the investigator will be summarized by visit and treatment group.

### 16.6 Columbia-Suicide Severity Rating Scale (C-SSRS) Scores

The C-SSRS was administered:

- for Screening at Visit 1: The C-SSRS assessment that collects a lifetime and 6 months recall (using the *Baseline/Screening Version*)
- for Baseline at Visit 3: The C-SSRS assessment that collects a lifetime and 6 months recall (using the *Baseline/Screening Version*)
- For subsequent visits: The C-SSRS assessment that collects information since the previous visit (using the *Since Last Visit Version*)

The numbers and percentages of patients with lifetime, 6 months pre-baseline or post-baseline suicide-related events based on the C-SSRS will be summarized by treatment group. For each summary, the most severe item with an answer "Yes" for each patient according to the ordering given in Panel 3 is displayed. For the post-baseline assessments, the summaries will be by treatment group and the most severe item with an answer "Yes" for the whole period for each patient related to suicidal ideation and/or behaviour will be summarized.

The number and percentage of patients with *no suicidal ideation or behaviour* will be included in the summaries.
#### Panel 3 C-SSRS Scores

| C-SSRS Score | | Related to: |
|---|---|---|
| 1 | Wish to be dead | Suicidal ideation |
| 2 | Non-specific active suicidal thoughts | |
| 3 | Active suicidal ideation with any methods (not plan) without intent to act | |
| 4 | Active suicidal ideation with some intent to act, without specific plan | |
| 5 | Active suicidal ideation with specific plan and intent | |
| 6 | Preparatory acts or behaviour | Suicidal behaviour |
| 7 | Aborted attempt | |
| 8 | Interrupted attempt | |
| 9 | Non-fatal suicide attempt | |
| 10 | Completed suicide (only applicable for the post-baseline assessments) | |

The C-SSRS scores will be summarized based on the APTS.

Missing C-SSRS scores will not be imputed.

Positive responses to *non-suicidal self-injurious behaviour* will be summarized separately.

For patients with any post-baseline suicidal ideation or behaviour (C-SSRS scores of 1 to 10), listings will be provided based on APRS including all C-SSRS scores for those patients

#### 16.7 MRI Safety Findings

MRI safety findings will be listed.

#### 16.8 Pregnancy Test

Pregnancy test results will be listed for patients with any positive results.

#### 16.9 Events of Death

Events of deaths will be summarized by treatment group, reason of death and study period . In addition, events of death will be listed.

Time-to-death will be investigated graphically using a Kaplan Meier plot and modelled, if applicable, by applying a Cox proportional-hazards model incl. treatment group, and region as covariates. For patients with no unique date-of-death the date of the last completed visit will be used. Patients still alive at the time of the safety follow-up visit will be censored using the date of the last safety follow-up visit as last observed time point.

## 17 Pharmacokinetic/Pharmacodynamic Analysis

The population pharmacokinetics of Lu AF82422 will be determined by means of non-linear mixed effect analysis. Estimated parameters of plasma exposure per patient (e.g. AUC and Cav) will be related to the efficacy and safety/tolerability in an exploratory PK/PD analysis. Details of the popPK and PK/PD analyses will be given in a separate popPK/PD analysis plan. The results of the popPK and PK/PD analyses will be reported in a popPK/PD report and relevant parts of it might be given in the clinical study report.

## 18 Immunogenicity Analysis (ADA)

The analysis of anti-Lu AF82422 antibodies will be performed for all subjects in the APTS receiving at least one dose of Lu AF82422. Subjects receiving placebo will not be analyzed for anti-Lu AF82422 antibodies.

#### Panel 4 ADA definitions

| Pre-existing ADA | Refers to antibodies reactive with the biologic drug that are present in subjects before drug administration |
|---|---|
| Treatment-induced ADA | ADA developed de novo following drug administration |
| Treatment-boosted ADA | Pre-existing ADA that were boosted to a higher-level following drug administration, i.e., titer is greater than the baseline titer by a fourfold increase |
| Neutralizing ADA (NAb) | ADA that inhibits or reduces the pharmacological activity of the drug |
| ADA-positive subject | A subject with at least one treatment-induced or treatment-boosted ADA-positive sample at any time during the treatment or follow-up observation period |
| ADA-negative subject | A subject without a treatment-induced or treatment-boosted ADA-positive sample during the treatment or follow-up observation period |
| ADA-inconclusive subject | A subject who cannot irrefutably be classified as ADA-negative since drug is present in the same sample at a level exceeding the validated drug tolerance level, i.e., drug tolerance |
| Transient ADA | ADA detected only at one sampling time point during the treatment or follow-up observation period, or ADA detected at two or more sampling time points during the treatment separated by a period less than 16 weeks, and the subject's last sampling time point is ADA-negative |
| Persistent ADA | Treatment-induced ADA detected at two or more sampling time points during the treatment (including safety follow-up period) where the first and last ADA-positive samples are separated by a period of 16 weeks or longer, or ADA incidence only in the last sampling time point of the treatment study period or at a sampling time point with less than 16 weeks before an ADA-negative last sample |
| Onset of ADA | Onset defined as the time period between the initial administration of IMP and the first instance of treatment-induced ADA |
| Duration of ADA | Referring to the longevity of treatment-induced ADA |
| ADA prevalence | The proportion of subjects having anti-drug antibodies (including pre-existing antibodies) at any point in time |
| ADA incidence | The proportion of subjects found to have seroconverted or boosted their pre-<br>existing ADA during the study period |

The following analysis will be carried out to the extent meaningful based on the total number of subjects identified with pre-existing or treatment-induced ADA.

If appropriate, data will be provided for:

- Pre-existing antibodies: ADA-positive subjects as a percentage of the total number of subjects, titer range (median and interquartile range (IQR)), percentage of treatment-boosted ADA-positive subjects, and duration of only pre-ADA, i.e., pre-ADA remained of same titer during the duration of study.
- Overall ADA prevalence: the number of ever-ADA-positive subject as portion of all study participants.
- Overall ADA incidence: combined results of treatment-boosted ADA-positive subjects and treatment-induced ADA-positive subjects (i.e., ADA-negative at baseline). For treatmentinduced ADA incidence, peak positive titer and range (median, IQR). For treatmentboosted ADA, incl. the computed fold increase in titer (ratio of peak post-administration titer to baseline titer) and range of titer increases (median, IQR).
- Onset and duration of treatment-induced ADA. Regarding duration, a differentiation will be made between transient and persistent treatment-induced and boosted ADA.

Furthermore, the potential impact of ADA on PK, PD (as assessed by target engagement (TE)), clinical safety and efficacy will be explored descriptively for subjects with pre-existing or treatment-induced ADA.

- PK and PD: will be evaluated stepwise firstly looking into mean exposure for ADA-positive vs. ADA-negative. In case any notable difference is found, PK will be considered by categorizing subjects into patients with impact of ADA vs. patients with no impact of ADA based on individual exposure over time to identify potential neutralizing/clearing ADA. To explore the ADA impact on PD, Safety and Efficacy the following analyses will be performed for ADA-positive vs. ADA-negative. Whether ADA is evaluated to have impact or not for an individual patients will be documented in patient listing.
- PD: TE as assessed by the plasma ratio of 'free' alpha-synuclein over 'total' alpha synuclein, plasma NfL, and MRI volumetric (as assessed by changes in primary regions)
- Safety: The number of hypersensitivity relevant TEAE's presented by SOC and PT, with focus on nature and timing of TEAE's (see below)
- Efficacy: Changes-from-baseline in UMSARS TS.

#### **Nature of TEAEs**

Consequences of immunogenicity on safety include the following TEAEs:

- Hypersensitivity reactions (as reported by Investigator)
- Hypersensitivity related TEAEs as Type I, II and III jointly, i.e., with a PT within 1) the SMQ of Hypersensitivity (narrow scope), 2) 'Cytokine release syndrome', and 3) the SMQ Vasculitis (narrow scope) or any of the 15 defined single PTs (see Appendix VI)

#### Timing of the TEAE

TEAE is only potentially related to immunogenicity if there is a temporal relationship to the ADA response, i.e., if there is a temporal relation between the onset of the TEAE and participants being or turning ADA positive, i.e., the participant is 'TEAE coincident ADA positive'.

All immunogenicity data will be listed by subject and period.

#### 19 Blinded Data Reviews

A blinded data review will take place throughout the study to ongoing handle data issues. The reviews may include, but are not limited to, data quality, protocol adherence, and the appropriateness of design assumptions.

An independent Safety Data Monitoring Committee (DMC) will regularly monitor the patients' safety data according to the DMC Charter. The DMC will have access to unblinded information for the double-blind treatment for each patient. Members of the DMC will not be involved in other study-related tasks.

### 20 Interim Analyses

No interim analyses will be conducted for this study.

# 21 Sample Size Considerations



The 18331A sample size has been selected to ensure an appropriate power to detect a 40% slowing in MSA progression in the Lu AF82422 dose group compared to the placebo group on a 5% significance level evaluated 1-sided. Applying a repeated measures model with proportional treatment effect, yields an approximate 75% power when having N=60 patients allocated 2:1 in favour of Lu AF82422 treatment (i.e., 40 on Lu AF82422 versus 20 on

placebo) when using the NLMIXED procedure for simulating in SAS<sup>®</sup>. To account for differences in treatment duration due to the study design, approximately 50% of the patients are expected to contribute with 60 weeks data and 25% of the patients with full 72 weeks data. On top, an overall 20% drop-out rate has been accounted for. For comparison, it is expected that the frequentist repeated measures model used for simulation is quite similar in relation to performance to the primary Bayesian repeated measures model.

#### 22 Statistical Software

The statistical software used will be SAS®, version 9.4 or later, and R, version 3.12 or later, respectively. For R, the packages Jags and Coda would be required to run the MCMC procedures.

### 23 Changes to Analyses Specified in the Protocol

• According to SAP section 16.1.4, TEAEs will be assigned to two periods rather than four periods as described in Protocol section 16.10.1, the reason being that the safety follow up periods following the DBP and the OLEP, respectively, will be part of the reporting periods rather than individual periods. In this way the first safety follow up period following the DBP will be reported as part of the DBP, and the safety follow up period following the OLEP will be reported as part of the OLEP.

### 24 Details on Data Handling

#### 24.1 Derived Variables

Total scores which are (also) calculated by the investigator (e.g. the UMSARS part I score used for inclusion/exclusion), will be represented in two variables: one calculated directly from item scores (e.g. PARAMCD: UMSARSP1) and one with the same name and the extension 'I' containing the total score as calculated by the investigator (e.g. PARAMCD: UMSARSP1I).

#### 24.1.1 Missing Item Scores

Since all rating scales will be performed electronically missing single items should in principle not occur. However, if >20% of the items for a rating scale or subscale are missing, the total score or subdomain score will be set to missing. The maximum number of missing items is given for each in Panel 6.

If number of missing items in a scale does not exceed the maximum number, total scores and/or subdomain scores will be imputed for the UMSARS part I and part II, SE-ADL, and EQ-5D-5L. The general rule when imputing total scores or subdomain scores is that the score will be calculated using the SAS function ROUND:

ROUND ([(sum of scores in non-missing items) / (number of non-missing items) \* (total number of items)])

Derived scores including imputed items will be marked (DTYPE = 'EXTRAP').

Panel 6 Maximum Number of Missing Items on Rating Scales

| PARAMCD | Description | Maximum Number of<br>Missing Items |
|---|---|---|
| UMSARSP1 | UMSARS part I score, 12 items | 2 |
| UMSARSP2 | UMSARS part II score, 14 items | 2 |
| EQ5D5L | EuroQoL 5-dimension, 5 items | 1 |

An exception to this rule will be for patients dropping out due to death. In case of death, the total or domain score will be set to worst rank according to Panel 7 below at the visit following the date of death applying both a narrow and a broad visit windowing approach. Hereafter, scores will be set to missing.

In case of drop-out due to death, derived scores will be included for the imputed values marked with D TYPE = 'WC'.

Panel 7 Imputation of worst rank following events of death

| PARAMCD | Description | Imputed worst rank |
|---|---|---|
| UMSARSP1 | UMSARS part I score | 48 |
| UMSARSP2 | UMSARS part II score | 56 |
| UMSARSTS | UMSARS total score | 104 |
| mUMSARS | Modified UMSARS part I score | 48 |
| COMPS | COMPASS Select Change - Orthostatic Intolerance Score | -60 |
| COMPS | COMPASS Select Change – Secretomotor Score | -25 |
| COMPS | COMPASS Select Change – Bladder Score | -30 |
| COMPS | COMPASS Select Change – Vasomotor Score | -10 |
| COMPS | COMPASS Select Change – Sleep Score | -25 |
| SEADL | Schwab & England ADL score | 0% |
| CGIS | Clinical Global Impression score – Severity | 4 |
| PGIS | Patient Global Impression score - Severity | 4 |
| OGIS | Observer-reported Global Impression - Severity | 4 |
| EQ5D5L | EuroQoL 5-dimension, each single domain | 5 |

#### 24.1.2 UMSARS scale

The UMSARS scale consists of four part, i.e. part I-IV, where part I and part II are covering multiple domains with an associated score, whereas part III is covering an autonomic examination and part IV is a 1-dimensional disability scale. In addition, two moderated

UMSARS scores will be derived, i.e., a modified UMSARS part I (mUMSARS) score and an abbreviated UMSARS (aUMSARS) score, respectively.

Panel 8 UMSARS Scale Overview

| UMSARS | Total Score | | |
|---|---|---|---|
| PART 1 | PART 2 | PART 3 | PART 4 |
| Historical functional review of activities of daily living over the past two weeks | Motor examination scale | Autonomic<br>examination (supine<br>blood pressure after | |
| 1. Speech 2. Swallowing 3. Handwriting 4. Cutting food/handling utensils 5. Dressing 6. Hygiene 7. Walking 8. Falling (past month) 9. Orthostatic symptoms 10. Urinary function 11. Sexual function 12. Bowel function Scored from 0-104 | Facial expression Speech Ocular motor dysfunction Tremor at rest Action tremor Increased tone Rapid alternating hand movements Finger taps Leg agility Heel-knee-shin test Arising from chair Posture Body sway Gait with higher scores | 15 min rest, and standing blood pressure within 10 mins of standing, supine and standing heart rate, and presence of autonomic symptoms) | Global disability scale, ranging from 1 (completely independent) to 5 (totally independent) |
| indicating great | ater impairment | | |

#### **UMSARS** part I and mUMSARS

The UMSARS part I comprises 12 items rating the average functional situation for the past 2 weeks (unless specified) according to the patient and caregiver interview. It covers the following domains: speech, swallowing, handwriting, cutting food and handling utensils, dressing, hygiene, walking, falling, orthostatic symptoms, urinary function, sexual function, and bowel function; all rated 0 to 4, with 0 = not affected/normal; 1= mildly affected/impaired; 2= moderately affected/impaired; 3= severely affected/impaired; and 4 = helpless or entirely affected/impaired. The UMSARS part I total score ranges from 0 to 48.

If more than 2 items for the UMSARS part I are missing, the score will be set to missing. If no more than 2 items are missing, the score will be equal to the mean of the recorded items multiplied by the total number of items and then rounded to the first decimal place using the SAS function ROUND:

ROUND ([(sum of scores in non-missing items) / (number of non-missing items) \* (total number of items)]).

The modified UMSARS part I (mUMSARS) score is derived by collapsing the response option 0 and 1 within each item  $\{0 \& 1 = 1\}$ . Hence, the mUMSARS score ranges from 12 to 48. In case of missing items the same above rule will be applied using the ROUND function.

#### **UMSARS** part II

The UMSARS part II comprises 14 items rating different aspects of motor performance for the worst affected limb at the actual visit. It covers the following domains: Facial expression, speech, ocular motor dysfunction, tremor at rest, action tremor, increased tone, rapid alternating movements of hands, finger taps, leg agility, heel-knee-shin test, arising from chair, posture, body sway, gait; all rated 0 to 4, with 0 = not affected/normal; 1= mildly affected/ impaired; 2= moderately affected/impaired; 3= severely affected/impaired; and 4 = helpless or entirely affected/impaired. The UMSARS part II total score ranges from 0 to 56.

If more than 2 items for the UMSARS part II are missing, the score will be set to missing. If no more than 2 items are missing, the score will be equal to the mean of the recorded items multiplied by the total number of items and then rounded to the first decimal place using the SAS function ROUND:

ROUND ([(sum of scores in non-missing items) / (number of non-missing items) \* (total number of items)]).

#### **UMSARS** part III

The UMSARS part III comprises an autonomic examination of systolic blood pressure, diastolic blood pressure, heart rate, and orthostatic symptoms. Supine blood pressure and heart rate are measured after 2 minutes of rest and again after 2 minutes of standing. Orthostatic symptoms are assessed as 'yes'/'no' and may include lightheadedness, dizziness, blurred vision, weakness, fatigue, cognitive impairment, nausea, palpitations, tremulousness, headache, neck and "coat-hanger" ache. The UMSARS part III is not reported as a joint score.

Missing data from UMSARS part III will not be imputed.

#### **UMSARS** part IV

The UMSARS part IV comprises a global disability scale ranging from 1-5, with 1='Completely independent. Able to do all chores with minimal difficulty or impairment. Essentially normal. Unaware of any difficulty'; 2='Not completely independent. Needs help with some chores'; 3='More dependent. Help with half of chores. Spends a large part of the day with chores'; 4='Very dependent. Now and then does a few chores alone or begins alone. Much help needed'; and 5='Totally dependent and helpless. Bedridden'.

Missing data from UMSARS part IV will not be imputed.

The UMSARS TS is derived as the sum of part I and part II, hence ranging from 0 to 104. The UMSARS TS will be missing in case either part I or part II would be missing at the same visit.

The UMSARS subscale scores are described in Panel 9.

Panel 9 Derivation of UMSARS total score and domain scores

| UMSARS total score and domain scores | Derivation | Range |
|---|---|---|
| UMSARS part I | Sum of part I items (1.1-1.12) | 0-48 |
| UMSARS part II | Sum of part items (2.1-2.14) | 0-56 |
| UMSARS part III | Individual part III items (3.1-3.4) | NA |
| UMSARS part IV | One item score 4.1 | 1-5 |
| UMSARS TS | Sum of part I and part II | 0-104 |
| Modified UMSARS (mUMSARS) | Sum of part I items with response option 0 and 1 collapsed (=1) | 12-48 |
| Abbreviated UMSARS (aUMSARS) | Sum of part I and part II selected items | 0-40 |

<sup>\*</sup> since the abbreviated UMSARS is still under development the final items will be amended at a later point.

#### 24.1.3 Composite Autonomic Symptom Score Select (COMPASS Select)

The COMPASS 31 is a refined, internally consistent, and markedly abbreviated quantitative measure of autonomic symptoms. It provides clinically relevant scores of autonomic symptom severity based on the well-established 169-item Autonomic Symptom Profile (ASP) and its validated 84-question scoring instrument, the Composite Autonomic Symptom Score (COMPASS). However, it applies a much-simplified scoring algorithm, and is suitable for widespread use in autonomic research and practice. COMPASS Select is a simplified version of the COMPASS 31 with selected items only.

Two versions of the COMPASS Select will be applied. At baseline, the COMPASS Select which is a 36-item questionnaire asking into autonomic symptoms within the past year. At subsequent visits, the COMPASS Select Change which is a 16-item questionnaire asking into changes in symptoms since last evaluation.

Since the COMPASS Select Change is licenced by the Mayo Clinic, they will be responsible for deriving the total scores to be used for further analysis. Patient-level single item data and the derived score will be included in sdtm format.

Panel 10 COMPASS Select Change domain scores

| COMPASS Change Select Domain* | Questions in domain | Range** |
|---|---|---|
| Orthostatic Intolerance domain Score (OI_domain) | Q1, 2, 3, 4, 5, 6 | -60-60 |
| Secretomotor domain score (Secretomotor_domain) | Q10, 11, 12 | -25-25 |
| Bladder domain score (Bladder_domain) | Q7, 8, 9 | -30-30 |
| Vasomotor domain score (Vasomotor_domain) | Q13 | -10-10 |
| Sleep domain score (Sleep_domain) | Q14, 15, 16 | -25-25 |
| COMPASS Change Select score (COMPASS_Change_Select) | Sum of all 5 domains | -150-150 |

<sup>\*</sup> COMPASS Select Change domain scores will be derived by Mayo Clinic

#### 24.1.4 Schwab & England Activity Daily Living Scale (SE-ADL)

The Schwab and England Activities of Daily Living (SE-ADL) scale is a method of assessing the capabilities of people suffering from impaired mobility. Originally presented at a Parkinson's disease conference, the scale assesses the difficulties patients have completing daily activities or chores. The scale uses percentages to represent how much effort and dependence on others, patients need to complete daily chores. The rating may be given by a professional or by the person being tested. Only the clinician reported part will be included in this study.

Panel 11 SE-ADL Scoring

| Percentage of independence | Degree of independence | Description |
|---|---|---|
| 100% | Completely independent | Able to do all chores without slowness, difficulty or impairment. |
| 90% | Completely independent | Able to do all chores, but with some degree of slowness, difficulty and/or impairment. One might take two times longer than normal to complete chores. |
| 80% | Usually completely independent | Takes two times longer than normal to complete chores. |
| 70% | Mostly independent | Faces more difficulty with some chores. One spends a large part<br>of the day with chores and might take three to four times longer<br>than normal. |
| 60% | Somewhat independent | Can do most chores, but exceedingly slowly and with much effort. Errors are possible during the chores. |
| 50% | Mostly dependent | Needs help with half of every chore. Everything is difficult to one. |
| 40% | Very dependent | Can assist with chores and can complete some alone. |

<sup>\*\*</sup> the lower score the more severe symptoms

| Percentage of independence | Degree of independence | Description |
|---|---|---|
| 30% | Very dependent | With help, can start chores. One can also complete few chores with effort and help. |
| 20% | Very dependent | Can slightly help with chores but cannot complete any alone. |
| 10% | Fully dependent | Is helpless and somewhat comatose. |
| 0% | Fully dependent | Is bedridden and helpless. One is almost completely comatose. |

#### 24.1.5 Clinical Global Impression Severity Scale (CGI-S)

The CGI-S is administered by an experienced neurologist familiar with MSA patients to make an expert clinical global judgement about the severity of the disease across various time points. The neurologist makes a judgement about the total picture of the patient at each visit: the disease severity, the patient's level of distress and other aspects of impairment, and the impact of disease on functioning. The rating is based upon observed and reported symptoms, behaviour, and function in the past seven days. Symptoms and behaviour may fluctuate over a week; the score should therefore reflect the average severity level across the seven days. The CGI-S is rated on a scale ranging from 0 to 4 (whereas the 0 = normal, not impaired; 1 = mildly impaired; 2 = moderately impaired; 3 = severely impaired; 4 = extremely impaired).

#### 24.1.6 Patient global Impression Scale (PGI-S)

The PGI-S is a self-reported single item to evaluate all aspects of patients' MSA symptoms. Patients are asked to choose the response that best describes the severity of their MSA symptoms over the past week. The question is rated on a 5-point scale ranging from 0 to 4 (0 = none; 1 = minor; 2 = moderate; 3 = severe; 4 = very severe). It takes approximately 1 minute to complete the PGI-S.

#### 24.1.7 Observer-reported Global Impression – Severity of Illness (OGI-S)

The OGI-S is a single-question carer/observer-reported outcome to evaluate all aspects of patients' MSA symptoms. Carer/observers are asked to choose the response that best describes the observed severity of MSA symptoms in the person they care for over the past week. The question is rated on a 5-point scale ranging from 0 to 4 (0 = none; 1 = minor; 2 = moderate; 3 = severe; 4 = very severe). It takes approximately 1 minute to complete the OGI-S.

#### 24.1.8 EuroQoL five-dimensional five-levels Scale (EQ-5D-5L)

The EQ-5D instrument comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS) that are cognitively undemanding, taking only a few minutes to complete. The questionnaire provides a simple descriptive profile of a respondent's health state. The EQ VAS provides an alternative way to elicit an individual's rating of their own overall current health. When the descriptive system profile is linked to a 'value set', a single

summary index value for health status is derived that can be used in economic evaluations of healthcare interventions.

The EQ-5D-5L covers five domains (i.e. MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION ) all evaluated using 5 response levels: 'having no problems', 'having slight problems', 'having moderate problems', 'having severe problems' and 'being unable to do/having extreme problems'.

Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state; for instance, 21111 means slight problems in the mobility dimension and no problems in any of the other dimensions. An EQ-5D summary index is derived by applying a formula that attaches values (weights) to each of the levels in each dimension. The index is calculated by deducting the appropriate weights from 1, the value for full health (i.e. state 11111).

The EQ VAS records the respondent's overall current health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.

#### 24.1.9 FeetMe® gait parameters

The FeetMe® Monitor sole combines pressure sensors, inertial control units and on-board computing capacity for real-time measurement of walking parameters and plantar pressures, which will be applied periodically for a subgroup according to study procedure (See Appendix IV). The patients receive insoles during scheduled visits and are asked to wear the insoles continuously for 10 days in their home environment in the 5 pre-defined periods (baseline and 4 post-dose assessments).

Equipped with inertial units and plantar pressure sensors, the soles provide quantitative and real time readings of the following gait parameters: heel attack, heel lift, swing duration and duration, single and double support, oscillation time, distance and walking speed, cadence, plantar pressure peak map. These parameters are measured on both feet and thus provide the asymmetries relative to these parameters.

Individual parameters of gait will be derived by-step for each home-based assessment period. For analysis purpose, parameters will be further collapsed using both the median and the 95<sup>th</sup> percentiles for each day and period, respectively. Additional percentiles will be derived for exploratory purposes. Panel 12 below contains a list of available parameters and endpoint description.

Panel 12 Derivation of gait parameters, by-step

| Technology | Parameter | Unit | Endpoint Description |
|---|---|---|---|
| FeetMe® insoles | Gait velocity | m/s | - The median and the 95 <sup>th</sup> percentiles for all gait parameters will be derived for each |
| | Stride length | m | subject and home-based period For exploratory purpose, the 95 <sup>th</sup> , the 75 <sup>th</sup> and the 50 <sup>th</sup> percentiles (median) will be |
| | Stride duration | s derived on an hourly basis for all he | derived on an hourly basis for all home-<br>based gait parameters |
| Swing duration s | | | |
| | Stance duration | S | |
| | Cadence | steps/min | |
| | Distance travelled per hour | m | |

FeetMe parameters calculated at each stride: strideLength (m), widthMotion (m), timeHeelStrike1 (ms), timeHeelStrike2 (ms), timeToeOff (ms), strideDuration (ms), velocity (m/s), cadence (stride/min), swingDuration (ms), stanceDuration (ms), swingPercentage (%), stancePercentage (%), stepTime (ms), stepLength (m), asymmetryParamStepTime (ms), asymmetryParamStepLength (m), singleSupportDuration (ms), doubleSupportDuration (ms), singleSupportPercentage (%), doubleSupportPercentage (%), asymmetryParamStrideDuration (ms), asymmetryParamStrideLength (m), asymmetryParamSingleSupportPercentage (%), strideElevation(cm), Capacitive measures of the 18 pressure sensors (in atmel unity), Centers of pressure (in cm, to confirm)

In case of large amount of missing data for a subject within a given period consisting of 10 days, the percentiles will not be derived and hence these will be set to missing. Data cleaning, population classification and confirmation of decision rules for derivation of percentiles will take place prior to database lock and will be documented as part of the classification meeting.

Additionally, raw data will be made available as sdtm format.

#### 24.1.10 BioSensics<sup>TM</sup> PAMSys sensor

PAMSys (Physical activity and posture) is a clinical-grade wearable sensor for continuous remote monitoring of physical activity, sleep, posture, gait parameters and falls, which will be applied periodically for a subgroup according to study procedure (See Appendix IV).

Panel 13 below contains a list of available parameters and endpoint description.

| Panel 13 | Derivation | of PAMSys | parameters |
|----------|------------|-----------|------------|
|----------|------------|-----------|------------|

| Posture and postural transition | Gait parameters |
|---|---|
| <ul> <li>Posture classification (sitting, standing, walking and lying down)</li> <li>Postural transition (duration and number of occurrence)</li> <li>Sedentary behavior</li> </ul> | <ul> <li>Number of steps (for example per hour)</li> <li>Walking duration (for example per hour)</li> <li>Time stamp of individual steps</li> <li>Cadence</li> <li>Cadence variability</li> <li>Number of episodes of walking (for example per day)</li> <li>Number of steps per walking episode</li> </ul> |
| Sleep and sleep quality | Falls and fall risk |
| <ul> <li>Start- and end-time of periods of lying down</li> <li>Sleep onset latency (i.e., time lying down before sleep onset)</li> <li>Wake time after sleep onset</li> <li>Total sleep time</li> </ul> | <ul> <li>Falls (number of falls and time of occurrence)</li> <li>Continuous fall risk monitoring</li> </ul> |

In case of large amount of missing data for a subject within a given period, endpoints might not be derived according to BioSensics procedure and hence the data will be set to missing. Data cleaning and classification will take place prior to database lock.

Additionally, raw data will be made available as sdtm format.

#### **24.1.11** Fall Diary

Assessment of falls during the course the trial will be done using a dedicated MSA fall diary developed by Lundbeck. The diary consists of 12 questions with response options as seen below in Panel 14, with number of falls within the last 24 hours (Q2) being the key outcome for further analysis.

Question 10, 11 and 12 are only to be filled out on a weekly basis and should only occur once a week in the e-diary. However, due to an initial mistake in the set-up, the weekly questions appeared daily and hence several assessments will be available within the same week. In those cases, the Day 7 assessment (related to the Day 1 being the first day an individual fills out the diary within a period) will be the applicable one used for the analysis; meaning that remaining assessments within the same period will be disregarded. The e-diary will be updated and hence this rule will only apply for early patients having multiple entries for the weekly questions within the same week.

Panel 14 Derivation of Fall Diary parameters

| Fall Diary question | Specific wording | Response option |
|---|---|---|
| Q1 | Did you fall in the past 24 hours? (A fall is defined as UNEXPECTANTLY coming to rest on the ground, floor or just a lower level than where you started.) | Yes/No |
| Q2 | How many times did you fall in the past 24 hours? | Number |
| Q3 | What time did you fall? | Time point |
| Q3<br>Q4 | Where were you when you fell? | Indoors /<br>Outdoors |
| Q5 | Was it in a place you know well? | Yes/No |
| Q6 | Did you experience any dizziness, light-headedness, feeling faint or blurred vision before falling? | Yes/No |
| Q7 | Did you experience freezing of gait/movement locking before falling? (Freezing of gait: feeling like your feet were stuck to the ground) | Yes/No |
| Q8 | Did you need somebody's help to get up after you fell? | Yes/No |
| Q9 | Did the fall cause any physical injury? | Yes/No |
| Q10 | During the last week, how many times did you consult a healthcare professional due to a fall? (consider any past falls / whenever the fall happened) | Number |
| Q11 | During the last week, how many times did you visit a hospital due to a fall? (consider any past falls / whenever the fall happened) | Number |
| Q12 | During the last week, how many times did you have an x-ray due to a fall? (consider any past falls / whenever the fall happened) | Number |

#### Number of falls per period

Within each dispense/observation period (BL, V9, V12, V15, and V18) the defined visit windows will be applied to identify valid data entries. Within each period, the total number of falls will be calculated as the sum of the Q2 responses. In addition, an adjusted total number of falls per period will be calculated as the total number of falls divided by the number of days where the Fall Diary was filled out (Q1 NOT missing). The adjusted number of falls per period will be the primary endpoint for further analysis of falls.

#### 24.1.12 Magnetic Resonance Imaging (MRI)

MRI at Screening will be performed for eligibility and, in addition, the presence of MRI abnormalities supporting the diagnosis of MSA (putaminal atrophy, pontine atrophy, cerebellar and middle cerebellar peduncle atrophy, presence of putaminal hyperintense rim, putaminal signal hypointensity and/or hot cross bun sign) will also be recorded.

In addition, MRI scans will be performed for evaluation of biomarkers of disease progression and safety. The scans will be evaluated by a central reader, as pre-specified in the study-specific *Imaging Charter*.

Panel 15 contains an overview for the MRI sequences and derived parameters used for evaluation of disease progression.

Panel 15 Derivation of MRI parameters

| MRI sequencing | Description | Regions of interest |
|---|---|---|
| Volumetric MRI (vMRI) | Quantification of atrophy<br>measures in brain ROIs | <ul><li>caudate nucleus</li><li>putamen</li><li>striatum</li></ul> |
| | | <ul><li>pons</li><li>brain stem</li><li>cerebellum</li></ul> |
| Diffusion-tensor imaging (DTI) | Quantification of diffusivity measures in brain ROIs | <ul> <li>caudate nucleus</li> <li>putamen</li> <li>globus pallidus</li> <li>pons</li> <li>cerebellar white matter</li> <li>middle cerebellar peduncle</li> </ul> |
| Arterial spin label (ASL) | Quantification of cerebral blood<br>flow (CBF) in selected brain<br>regions | <ul><li>putamen</li><li>cerebellum</li></ul> |

Additional MRI sequences will be performed for assessment of safety, including 2D T2-weighted, 3D T2 FLAIR, diffusion-weighted imaging and gradient-recalled echo (GRE) sequence. The last will be used to assess the presence of cerebral microhaemorrhages.

The primary analysis for the volumetric parameters will be the percentage-wise change from baseline in each region-of-interest in the actual numbers, whereas numbers normalized by the intercranial volume (head size) will be secondary.

In some instances, an alternative workflow was performed to ensure quality of data. In case where both the original and the re-analyzed value would be present, the re-analyzed value would be the one used for further analyses.

#### 24.2 Assigning Data to Visits

*Invalid assessments* will be assigned AVISTN = 888. If the date of last dose is missing, assessments will be considered valid. If multiple assessments are taken the same day, only the last assessment will be valid. Invalid assessments will not be considered in descriptive statistics or statistical analyses but will be included in listings of safety variables.

Assessments at *unscheduled and withdrawal visits* will be assigned to a target day (AWTARGET) based on days after baseline visit, and to an analysis week (AVISTN = AWTARGET/7). Assessments falling outside a defined visit window will be evaluated and will be deemed invalid (AVISTN = 888) for that specific windowing approach in case no obvious week can be identified.

#### 24.2.1 UMSARS and additional efficacy COAs

For UMSARS, both a narrow and a broad approach will be applied for assigning observations to a visit: 1) observations will be mapped to the nearest official clinical visit in 4-weeks intervals, independent whether UMSARS originally was scheduled for this visit, and 2)

observations will be mapped to the nearest official UMSARS visit in 12-weeks intervals according to protocol.

Panel 16 Visit Windows for UMSARS

| Nominal Vis Number (DB-Period) | Nominal<br>Vis Week | Nominal<br>Vis Day | Time Window<br>narrow <sup>1</sup> | Time Window<br>broad <sup>1</sup> |
|---|---|---|---|---|
| V1 (Screening Visit) | -6 | -42 | NA | NA |
| V3 (Baseline Visit) | 0 | 0 | -7 to 7 | -7 to 7 |
| V5 (WD Visit) | 4 | 28 | 15 to 42 | NA |
| V7 (WD Visit) | 8 | 56 | 43 to 69 | NA |
| V9 (planned UMSARS/WD Visit) | 12 | 84 | 70 to 98 | 15 to 126 |
| V10 (WD Visit) | 16 | 112 | 99 to 126 | NA |
| V11 (WD Visit) | 20 | 140 | 127 to 154 | NA |
| V12 (planned UMSARS/WD Visit) | 24 | 168 | 155 to 182 | 127 to 210 |
| V13 (WD Visit) | 28 | 196 | 183 to 210 | NA |
| V14 (WD Visit) | 32 | 224 | 211 to 238 | NA |
| V15 (planned UMSARS/WD Visit) | 36 | 252 | 239 to 266 | 211 to 294 |
| V16 (WD Visit) | 40 | 280 | 267 to 294 | NA |
| V17 (WD Visit) | 44 | 308 | 295 to 322 | NA |
| V18 (planned UMSARS/EoTDBP/WD Visit) | 48 | 336 | 323 to 350 | 295 to 378 |
| V19 (EoTDBP/WD Visit) | 52 | 364 | 351 to 378 | NA |
| V20 (EoTDBP/WD Visit) | 56 | 392 | 379 to 406 | NA |
| V21 (planned UMSARS/EoTDBP/WD Visit) | 60 | 420 | 407 to 434 | 379 to 462 |
| V22 (EoTDBP/WD Visit) | 64 | 448 | 435 to 462 | NA |
| V23 (EoTDBP/WD Visit) | 68 | 476 | 463 to 490 | NA |
| V24 (planned UMSARS/EoTDBP Visit) | 72 | 504 | 491 to 518 | 463 to 518 |
| Nominal Visit Number (OLE-Period) | | | | |
| V1E (baseline OLEP Visit) <sup>2</sup> | 0E | 0 | -7 to 7 | -7 to 7 |
| V2E (WD Visit) | 4E | 28 | 15 to 42 | NA |
| V3E (WD Visit) | 8E | 56 | 43 to 69 | NA |
| V4E (planned UMSARS/WD Visit) | 12E | 84 | 70 to 98 | 15 to 126 |
| V5E (WD Visit) | 16E | 112 | 99 to 126 | NA |
| V6E (WD Visit) | 20E | 140 | 127 to 154 | NA |
| V7E (planned UMSARS/WD Visit) | 24E | 168 | 155 to 182 | 127 to 210 |
| V8E (WD Visit) | 28E | 196 | 183 to 210 | NA |
| V9E (WD Visit) | 32E | 224 | 211 to 238 | NA |
| V10E (planned UMSARS/WD Visit) | 36E | 252 | 239 to 266 | 211 to 294 |
| V11E (WD Visit) | 40E | 280 | 267 to 294 | NA |
| V12E (WD Visit) | 44E | 308 | 295 to 322 | NA |
| V13E (planned EoTOLE Visit) | 48E | 336 | 323 to 350 | 295 to 350 |

All post-baseline visits (except EoT visits) can be converted into a Withdrawal (WD) Visit.

Records to be used in descriptive statistics or statistical analyses will be flagged with ANL01FL=Y and ANL02FL=Y. ANL01FL = Y and ANL02FL=Y will be assigned to all valid assessments (NOMWEEK not equal to 888) unless an assessment at the Withdrawal Visit or an Unscheduled Visit is assigned to the same analysis week as a scheduled visit (having the same NOMWEEK). In this case, ANL01FL = Y will be assigned to one valid visit prioritized in the following order: Scheduled Visit, Unscheduled Visit, and Withdrawal Visit.

CGI-S, PGI-S, and OGI-S will follow the same windowing principles since these were administered at the exact same visits as the UMSARS. The remaining COAs, i.e., SE-ADL, COMPASS Select Change and EQ-5L-5D were only administered at Week 24, 48 and 72 (Visit 12, 18, and 24) post-baseline in the DBP, and hence the broad windowing will only contain these visits using the above intervals, meaning that some observations might be deemed invalid for this mapping. However, they will be mapped into the above narrow windows as well using the continuous windowing approach. The same principles will be applied for the OLEP.

Remission in the CGI-S, PGI-S or OGI-S score (defined as a score of 1 or 2) at each analysis week following a baseline will be included as new parameters (PARAM=*Remission*).

#### 24.2.2 MRI parameters

MRI parameters (volumetric, DTI and ASL) are assessed at the following visits, and hence a broad windowing will only be applied for these visits. A narrow window will also be defined using all per-protocol defined efficacy visits as scheduled in Panel 16 above. Only MRI volumetric will be evaluated in the OLEP.

Panel 17 Visit Windows for MRI

| Nominal Vis Number (DB-Period) | Nominal<br>Vis Week | Nominal<br>Vis Day | Time Window<br>narrow <sup>1</sup> | Time Window<br>broad <sup>1</sup> |
|---|---|---|---|---|
| V3 (Baseline Visit) | 0 | 0 | -7 to 7 | -7 to 7 |
| V9 (planned MRI Visit) | 12 | 84 | 70 to 98 | 15 to 126 |
| V12 (planned MRI Visit) | 24 | 168 | 155 to 182 | 127 to 210 |
| V18 (planned MRI Visit) | 48 | 336 | 323 to 350 | 295 to 378 |
| V24 (planned UMSARS/EoTDBP Visit) | 72 | 504 | 491 to 518 | 463 to 518 |
| Nominal Visit Number (OLE-Period) | | | | |
| V1E (baseline OLEP Visit) <sup>2</sup> | 0E | 0 | -7 to 7 | -7 to 7 |
| V13E (planned EoTOLE Visit) | 48E | 336 | 323 to 350 | 295 to 350 |

 $<sup>^1</sup>$  For DBP and OLEP, respectively, the applied narrow window will be continuous (i.e.,  $\pm 14$  days) to avoid invalid assessments (protocol text  $\pm 3$  days). The broad window is set up as continuous as well to match.

<sup>&</sup>lt;sup>2</sup> EoTDBP Visit will work as Baseline Visit for the OLEP if done within the acceptable window.

#### 24.2.3 Blood sampling parameters

For blood sampling for IMP, safety lab (only one performed also at screening),  $\alpha$ -synuclein and ADA the following windowing will be applied with the addition of the Visit 6 and the Safety follow-up Visit (SFU).

Panel 18 Visit Windows for Blood Sampling Parameters

| Nominal Vis Number (DB-Period) | Nominal<br>Vis Week | Nominal<br>Vis Day | Time Window<br>narrow <sup>1</sup> | Time Window<br>broad <sup>1</sup> |
|---|---|---|---|---|
| V1 (Screening Visit – planned sampling) | -6 | -42 | NA | NA |
| V3 (Baseline Visit – planned sampling) | 0 | 0 | -7 to 7 | -7 to 7 |
| V5 (planned sampling Visit) | 4 | 28 | 21 to 35 | 21 to 35 |
| V6 (planned sampling Visit) | 6 | 42 | 36 to 49 | 36 to 49 |
| V7 (planned sampling Visit) | 8 | 56 | 50 to 69 | 50 to 69 |
| V9 (planned sampling Visit) | 12 | 84 | 70 to 98 | 70 to 126 |
| V10 (WD Visit) | 16 | 112 | 99 to 126 | NA |
| V11 (WD Visit) | 20 | 140 | 127 to 154 | NA |
| V12 (planned sampling Visit) | 24 | 168 | 155 to 182 | 127 to 210 |
| V13 (WD Visit) | 28 | 196 | 183 to 210 | NA |
| V14 (WD Visit) | 32 | 224 | 211 to 238 | NA |
| V15 (planned sampling Visit) | 36 | 252 | 239 to 266 | 211 to 294 |
| V16 (WD Visit) | 40 | 280 | 267 to 294 | NA |
| V17 (WD Visit) | 44 | 308 | 295 to 322 | NA |
| V18 (planned sampling Visit) | 48 | 336 | 323 to 350 | 295 to 378 |
| V19 (EoTDBP/WD Visit) | 52 | 364 | 351 to 378 | NA |
| V20 (EoTDBP/WD Visit) | 56 | 392 | 379 to 406 | NA |
| V21 (planned sampling Visit) | 60 | 420 | 407 to 434 | 379 to 462 |
| V22 (EoTDBP/WD Visit) | 64 | 448 | 435 to 462 | NA |
| V23 (EoTDBP/WD Visit) | 68 | 476 | 463 to 490 | NA |
| V24 (planned sampling EoTDBP/WD Visit) | 72 | 504 | 491 to 518 | 463 to 518 |
| V25 (planned sampling SFU Visit) | 88 | 616 | 609 to 623 | 595 to 630 |

All post-baseline visits (except EoT visits) can be converted into a Withdrawal (WD) Visit.

<sup>&</sup>lt;sup>1</sup> For DBP and OLEP, respectively, the applied narrow window will be continuous (i.e.,  $\pm 14$  days) to avoid invalid assessments (protocol text  $\pm 3$  days). The broad window is set up as continuous as well to match.

<sup>&</sup>lt;sup>2</sup> EoTDBP Visit will work as Baseline Visit for the OLEP if done within the acceptable window.

| Nominal Visit Number (OLE-Period) | | | | |
|---|---|---|---|---|
| V1E (BL OLEP Visit – planned sampling) <sup>2</sup> | 0E | 0 | -7 to 7 | -7 to 7 |
| V2E (WD Visit) | 4E | 28 | 15 to 42 | NA |
| V3E (WD Visit) | 8E | 56 | 43 to 69 | NA |
| V4E (WD Visit) | 12E | 84 | 70 to 98 | NA |
| V5E (WD Visit) | 16E | 112 | 99 to 126 | NA |
| V6E (WD Visit) | 20E | 140 | 127 to 154 | NA |
| V7E (planned sampling Visit) | 24E | 168 | 155 to 182 | 127 to 210 |
| V8E (WD Visit) | 28E | 196 | 183 to 210 | NA |
| V9E (WD Visit) | 32E | 224 | 211 to 238 | NA |
| V10E (WD Visit) | 36E | 252 | 239 to 266 | NA |
| V11E (WD Visit) | 40E | 280 | 267 to 294 | NA |
| V12E (WD Visit) | 44E | 308 | 295 to 322 | NA |
| V13E (EoTOLE Visit – planned sampling) | 48E | 336 | 323 to 350 | 295 to 350 |
| SFU-E (planned sampling SFU Visit | 64E | 448 | 434 to 462 | 434 to 462 |

All post-baseline visits (except EoT visits) can be converted into a Withdrawal (WD) Visit.

Since CSF sampling for IMP, NfL, t-tau and  $\alpha$ -synuclein quantification only is planned for Visit 3 (Baseline), Visit 18 and Visit 72, the above broad windowing will only be applied around these visits. The above narrow windowing will be identical. CSF sampling will not be performed in the OLEP.

Blood sampling for NfL will be assessed at Screening Visit and Baseline Visit Pre-IMP and at Visit 9, 12, 15, 18, 24, 1E, 7E and 13E post-IMP, and hence the above broad windowing will only be applied around these visits. Again, the above narrow windowing will be fully applied in addition.

#### 24.2.4 Vital signs and C-SSRS

Vital signs and C-SSRS assessments will be performed at all DBP and OLEP post-baseline visits except the two Telephone visits (i.e., Visit 4 and Visit 8), and hence only the above narrow windowing will be applied. The C-SSRS will in addition be assessed at the Screening Visit.

#### 24.2.5 Weight

Weight assessments will be performed at the following visits, and hence a broad windowing will only be applied for these visits. A narrow window will also be defined using all perprotocol defined visits as scheduled in Panel 18 above. Weight is not collected in the OLEP.

 $<sup>^{1}</sup>$  For DBP and OLEP, respectively, the applied narrow window will be continuous (i.e.,  $\pm 14$  days) to avoid invalid assessments (protocol text  $\pm 3$  days). The broad window is set up to allow additional flexibility.

<sup>&</sup>lt;sup>2</sup> EoTDBP Visit will work as Baseline Visit for the OLEP if done within the acceptable window.

Panel 19 Visit Windows for Weight

| Nominal Vis Number (DB-Period) | Nominal<br>Vis Week | Nominal<br>Vis Day | Time Window<br>narrow <sup>1</sup> | Time Window<br>broad <sup>1</sup> |
|---|---|---|---|---|
| V1 (Screening Visit – planned eval) | -6 | -42 | See Panel 16 | NA |
| V3 (Baseline Visit – planned eval) | 0 | 0 | | -7 to 7 |
| V9 (planned eval Visit) | 12 | 84 | | 50 to 126 |
| V12 (planned eval Visit) | 24 | 168 | | 127 to 210 |
| V15 (planned eval Visit) | 36 | 252 | | 211 to 294 |
| V18 (planned eval Visit) | 48 | 336 | | 295 to 378 |
| V24 (planned eval EoTDBP/WD Visit) | 72 | 504 | | 463 to 518 |

All post-baseline visits (except EoT visits) can be converted into a Withdrawal (WD) Visit.

#### 24.2.6 ECG

ECG assessments will be performed at the following visits, and hence a broad windowing will only be applied for these visits. A narrow window will also be defined using all per-protocol defined visits as scheduled in Panel 18. ECG is not collected in the OLEP.

Panel 20 Visit Windows for ECG

| Nominal Vis Number (DB-Period) | Nominal<br>Vis Week | Nominal<br>Vis Day | Time Window<br>narrow <sup>1</sup> | Time Window<br>broad <sup>1</sup> |
|---|---|---|---|---|
| V1 (Screening Visit – planned eval) | -6 | -42 | See Panel 16 | NA |
| V3 (Baseline Visit – planned eval) | 0 | 0 | | -7 to 7 |
| V6 (planned sampling Visit) | 6 | 42 | | 36 to 49 |
| V12 (planned eval Visit) | 24 | 168 | | 127 to 210 |
| V18 (planned eval Visit) | 48 | 336 | | 295 to 378 |
| V24 (planned eval EoTDBP/WD Visit) | 72 | 504 | | 463 to 518 |

All post-baseline visits (except EoT visits) can be converted into a Withdrawal (WD) Visit.

#### 24.2.7 Fall Diary

Each Fall Diary period will be defined as the period between the two visits where the diary was supposed to be filled out according to the protocol. Hence, even though this per protocol has been defined as a two-week period for the baseline period and a four-week period for the subsequent periods, the length of each individual period will slightly vary depending on the visit structure for each individual patient. Hence, the following rules will be applied for mapping data into the periods:

<sup>&</sup>lt;sup>1</sup> For DBP the applied narrow window will be continuous (i.e.,  $\pm 14$  days) to avoid invalid assessments (protocol text  $\pm 3$  days). The broad window is set up to allow additional flexibility.

<sup>&</sup>lt;sup>1</sup> For DBP the applied narrow window will be continuous (i.e.,  $\pm 14$  days) to avoid invalid assessments (protocol text  $\pm 3$  days). The broad window is set up to allow additional flexibility.

Panel 21 Windows for Fall Diary (Periods)

| Period (DB-Period) | Start visit | End visit | Planned duration | window around<br>both visits* |
|---|---|---|---|---|
| Period 0 (Baseline) | Visit 2 (R. visit) | Visit 3 (BL visit) | 2 weeks | +/- 3 days |
| Period 1 (post-IMP) Visit 7 | | Visit 9 | 4 weeks | +/- 3 days |
| Period 2 (post-IMP) | Visit 11 | Visit 12 | 4 weeks | +/- 3 days |
| Period 3 (post-IMP) | Visit 14 | Visit 15 | 4 weeks | +/- 3 days |
| Period 4 (post-IMP) | Visit 17 | Visit 18 | 4 weeks | +/- 3 days |

For each period, the data will be mapped into the end visit. Only one windowing approach will be defined around the relevant visits. The Fall Diary data is not collected in the OLEP.

Visit windows for FeetMe and PAMSys devices will be defined on a similar way for consistency.

#### 24.3 Assigning Adverse Events to Analysis Phases

Adverse events will be assigned to an analysis period as follows:

- Adverse events prior to treatment Records not classified as TEAEs will have APHASE= PRETREAT
- Adverse events in the double-blind period (DBP) all TEAEs with date of onset or worsening of intensity/seriousness after first dose of IMP in the DBP and until first dose of IMP in the OLE period (planned for Visit 1E for patients entering the OLE) or the Safety Follow up visit for the DBP (SFU Visit 25 for patients NOT entering the OLE) (assigned APHASE = DOUBLE BLIND).
- Adverse events in the Open-Label Extension period TEAEs with date of onset or worsening of intensity/seriousness after first dose of IMP in the OLE period (Visit 1E) and until the final Safety Follow up visit for the OLE (Visit 64E) (assigned APHASE = OLE).

If the start date is missing/incomplete and not eligible for imputation, the TEAE will be assigned to the DOUBLE BLIND phase.

#### 24.4 Handling Missing or Incomplete Dates/Times

#### 24.4.1 IMP Start and Stop Dates

For deriving variables for adverse events and concomitant medication:

- Missing IMP start date will be imputed for enrolled patients by the date of the baseline visit
- Missing IMP stop date will be imputed for enrolled patients by the date of the latest attended visit (scheduled/unscheduled/withdrawal)

For evaluating validity of efficacy assessments:

• Missing IMP stop date will be imputed for enrolled patients by the date of the latest attended visit (scheduled/unscheduled/withdrawal) before the safety follow-up

Exposure will not be calculated for patients with missing IMP start and/or stop dates.

#### 24.4.2 Withdrawal Date

For withdrawn patients with a missing Withdrawal Visit, the date of the last attended visit before safety follow-up will be used in the calculation of time to withdrawal from treatment.

#### 24.4.3 Medication Start and Stop Dates

Concomitant medications with missing start and stop dates will be classified according to the following rulesas determined from the IMP start date. Incomplete dates will be evaluated and compared to IMP start date by imputing the missing information as follows:

- If Day is missing (DD): for start dates, 1 will be used; for end dates, the last day in that respective month, i.e., 28/29/30/31
- If Month is missing (MMM): for start dates: January will be used; for end dates, December will be used
- If Year is missing (YYYY): for start dates: year will be set to the year before IMP start; for end dates, year will be set to the year after last IMP

No duration will be calculated for ongoing medications and for medications with missing/incomplete start date and/or stop date.

#### 24.4.4 Adverse Event Start and Stop Dates

If the start date is missing/incomplete for an adverse event and the stop date is prior to the first dose of IMP, the adverse event will be classified as a pre-treatment adverse event. In all other cases of an adverse event with a missing/incomplete start and/or stop date, the adverse event will be classified as a TEAE. No imputation of start/stop dates will be done, except in the case of adverse events which change in intensity/seriousness. For details on deriving multiple events from change in intensity/seriousness, and corresponding stop- and start dates, see section 24.5.2.

For adverse events ongoing at the end of the study, the date of the last study contact will be used as the stop date for the adverse event in the calculation of duration. For other adverse events with a missing/incomplete start or stop date, the duration will not be calculated.

#### 24.4.5 Diagnosis and Symptom onset Start Dates

Missing start dates for diagnosis and symptom onset will be imputed according to the following rules:

• If Day is missing (DD): The first day of the month will be used, i.e., 01

• If Month is missing (MMM): January will be used, i.e., 01

If both dates are missing hence 01-01 should be used. After imputation, the calculation of both 'time-since-diagnosis' and 'time-since-symptom-onset' should be done in relation to treatment start date (i.e., TRTSDT – DIAGDTC, TRTSDT – SYMPDTC), meaning that if the diagnosis was done within the same year of treatment start, then time-since-diagnosis should be <1.

#### 24.5 Data with Multiple Records

#### 24.5.1 Dose Changes in Medication

Dose changes in medications are recorded on multiple rows in the dataset, with different start and stop dates. When classifying medications into periods (prior to IMP, continued after first dose of IMP, started at or after first dose of IMP), each dose is considered a separate medication, and the same medication can be assigned to several periods for the same patient. Within a period, multiple entries contribute as a single count.

#### 24.5.2 Changes in Intensity or Seriousness of Adverse Events

Changes in adverse event intensity or seriousness are recorded on multiple rows in the dataset. An adverse event that changes in intensity or seriousness will contribute to the count of events as a single event.

In summaries of adverse events presented by intensity, the maximum intensity of the adverse event will be used. The maximum intensity is searched for in events with changes, as well as over repeated events based on the preferred term. For TEAEs and causally related TEAEs, the record(s) with the maximum intensity and maximum related intensity within an analysis phase will be flagged in ADaM data with ASEVMAX=Y and ARSEVMAX=Y, respectively. Adverse events for which information on intensity is missing will be classified as *severe*. Adverse events for which information on seriousness is missing will be classified as *serious*.

During the course of an event, information about all changes in intensity are collected (intensity and start date of intensity change). In ADaM data, changes in intensity are included as additional records (rows) to the originally reported adverse event reflecting the way data are collected. For instance, an adverse event that changes from mild to moderate will have two records, one with intensity mild and one with intensity moderate. Start date for the first intensity will be the start date for the originally reported event. The stop date for the last intensity will be the stop date for the originally reported event, and for the preceding intensities the stop date will be set to the date of reported change in intensity minus 1, or the date of reported change if a change occurring on the same day as the originally reported event, or if there is more than one change on a day.

If an adverse event changes from non-serious to serious, in addition to the originally reported adverse event start date, the start date for the seriousness is reported. However, the event is only reported as serious in the adverse event eCRF. In ADaM data, adverse events that change

from non-serious to serious will be included as two records, one with seriousness non-serious and one with seriousness serious. The start date for the non-serious event will be the start date for the originally reported adverse event, and the stop date will be set to the start date of the seriousness minus 1. The stop date for the serious event will be the stop date for the originally reported adverse event. If an intensity and seriousness is reported on the same date, record will be added reflecting both the change in intensity and seriousness (e.g. for an adverse event originally reported as being mild and non-serious is reported as having changed to severe and serious on the same date, there will be one additional record in data).

Duration (days) will be calculated for each intensity/seriousness based on the intensity/seriousness start-and stop dates. No duration will be calculated for adverse events with incomplete or missing start-or stop date, or for events ongoing at the end of the study.

#### 24.6 Handling Exposure Data

Exposure across the whole study period will be assigned PARAM = 'Study' and exposure within visit intervals will be assigned PARAM = 'V1\_V2', PARAM = 'V2\_V3', and PARAM = 'V3\_V4', etc., for intervals between V1 and V2, V2 and V3, V3 and V4, etc., respectively.

Exposure to dose of Lu AF82422 in the study period is calculated as:

(Date of last dose +28) – (Date of first dose +1)

Exposure in days will be given in variables EXP1D, EXP2D, EXP3D. Corresponding exposure in years will be given in variables EXP1Y, EXP2Y, EXP3Y derived as exposure in days divided by 365.25.

The average dose in the full study period will be derived.

For the study time-interval the duration of exposure to dose will be categorized into the intervals 1-7 days, 8-14 days, ..., etc.

#### 24.7 Handling digital-device data

Data from two digital devices, i.e., FeetMe shoe insoles and BioSensics PAMSys wearable, will be collected throughout the study according to study procedure. Both data sources will have been curated by the vendor prior to integrating into sdtm and hence, relevant parameters have already been derived for the specific periods.

#### Reference

- 1 The natural history of multiple system atrophy: a prospective European cohort study, G.K. Wenning et al, Lancet Neurol 2013; 12: 264–74; US ref: Natural history of multiple system atrophy in the USA: a prospective cohort study, P.A. Law et al, Lancet Neurol 2015; 14: 710–19
- The DIAN-TU Next Generation Alzheimer's prevention trial: Adaptive design and disease progression model, R. J. Bateman et al., Alzheimer's & Dementia 13 (2017) 8-19.
- A novel cognitive disease progression model for clinical trials in autosomal-dominant Alzheimer's disease, G. Wang et al., Statistics in Medicine. 2018;1–9.
- Developing a Natural History Progression Model for Duchenne Muscular Dystrophy Using the Six-Minute Walk Test, L. Hamuro et al., CPT Pharmacometrics Syst. Pharmacol. (2017) 6, 596–603.
- 5 Bayesian model of disease progression in GNE myopathy, M. Quintana et al., Statistics in Medicine. 2019; 38:1459–1474.
- 6 Natural cubic splines for the analysis of Alzheimer's clinical trials, M. Donohue et al, Pharmaceutical Statistics. 2023;1-12.

# Appendix I Statistical Analysis Plan Authentication and Authorization

# **Statistical Analysis Plan Authentication and Authorization**

Trial title: Interventional, randomized, double-blind, parallel-group, placebo-controlled, multi-centre study to assess the efficacy, safety and tolerability of Lu AF82422 in patients with Multiple System Atrophy

Trial No.: 18331A

SAP date: 20 December 2023

This document has been signed electronically. The signatories are listed below.

Authentication

Biostatistician: PPD

Clinical research: PPD

Authorization

Head of Biostatistics:

PPD

# Appendix II SAS® Code

# SAS® Code



Study 18331A – Statistical Analysis Plan



# Appendix III 'R' code

# 'R' Code





# Appendix IV Study Flow Chart

# **Study Flow Chart**

Table 1 Study Procedures and Assessments - Double-blind Treatment Period

| Visit Name | Screening | Randomization | Baseline + IMP | Telephone Visit | IMP | Site Visit | IMP | Telephone Visit | IMP | IMP | IMP | IMP | IMP | IMP | IMP | IMP | IMP | IMP/EoT <sup>a</sup> | IMP/EoTª | IMP/EoT <sup>a</sup> | IMP/EoT <sup>a</sup> | IMP/EoT <sup>a</sup> | IMP/EoT <sup>a</sup> | EoT/Withdrawal <sup>b</sup> | ${\rm SFU}^c$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 |
| Week <sup>d</sup> | 6 | -2 | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 88 |
| Visit Window <sup>e</sup> (days relative to nominal visit) | | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>7 |
| Screening/Randomization | Screening/Randomization Procedures and Assessments | | | | | | | | | | | | | | | | | | | | | | | | |
| Signed informed consent | | | | | | | | | | | | | | | | | | | | | | | | | П |
| Demographics (age, sex, race) | 1 | | | | | | | | | | | | | | | | | | | | | | | | |
| MSA diagnostic criteria:<br>Possible or probable,<br>MSA-P or MSA-C | 1 | | | | | | | | | | | | | | | | | | | | | | | | |
| MSA History | 1 | | | | | | | | | | | | | | [ <u>-</u> | | | | | | | | | | |
| MoCA | √ | | | | | | | | | | | | | | | | | | | | | | | | $\Box$ |
| Relevant medical history<br>(e.g., psychiatric, neurological) | √ | | | | | | | | | | | | | | | | | | | | | | | | <br> |
| Recent and on-going medication | √ | | | | | | | | | | | | | | | | | | | | | | | | |
| Height | √ | | | | | | | | | | | | | | | | | | | | | | | | |
| Blood sampling for preg-<br>nancy test | √ | | | | | | | | | | | | | | | | | | | | | | | | |
| MRI scan for eligibility <sup>f</sup> | 1 | | | | | | | | | | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | 1 | <b>√</b> | | | | | | | | | | | | | | | | | | | | | | | <b> </b> |
| Signs and symptoms present at SCR, Randomization and/or BL (before IMP administration; recorded on an Adverse Event Form) | 1 | √ | √ | | | | | | | | | | | | | | | | | | | | | | |
| Randomization | | $\sqrt{}$ | | | | | | | | | | | | | | | | | | | | | | | |
| <b>Efficacy Assessments</b> | | | | | | | | | | | | | | | | | | | | | | | | | |
| UMSARS | 1 | | $\sqrt{}$ | | | | | | 1 | | | $\sqrt{}$ | | | 1 | | | $\sqrt{}$ | | | <b>V</b> | | | $\sqrt{}$ | |
| SE-ADL | ļ | | | | | | | | | | | $\checkmark$ | | | | | | √ | | | | | | $\sqrt{}$ | |
| COMPASS Select | [ | | | | | | | | | | | | | | [ | | | | | | | | | | [ ] |
| COMPASS Select Change | [ ] - | | | | | | | | | | | $\sqrt{}$ | | | | | | 1 | | | | | | √ | |
| CGI-S | | | | | | <u> </u> | | | $\sqrt{}$ | | | $\sqrt{}$ | | <u> </u> | $\sqrt{}$ | | | √ | | | √ | | | $\sqrt{}$ | |
| PGI-S<br>OGI-S | | | √<br>√ | | | | | | √<br>√ | | | √<br>√ | | | √<br>√ | | | √<br>√ | | | √<br>√ | | | $\sqrt{}$ | [] |
| | L | i i | الاناما | L J | I | i | L J | | L _ <u>`</u> _ | L J | | LLLI | I | i | L _ <u>'</u> _ J | | L | L _'_ J | 1 ! | L | '_ | ـــ | L | | L l |
| Visit Name | Screening | Randomization | Baseline + IMP | Telephone Visit | IMP | Site Visit | IMP | Telephone Visit | IMP | IMP | IMP | IMP | IMP | IMP | IMP | IMP | IMP | IMP/EoT <sup>a</sup> | IMP/EoT <sup>a</sup> | IMP/EoT <sup>a</sup> | IMP/EoT <sup>a</sup> | IMP/EoT <sup>a</sup> | IMP/EoT <sup>a</sup> | EoT/Withdrawal <sup>b</sup> | ${\rm SFU}^c$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 |
| Week <sup>d</sup> | 6 | -2 | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 88 |
| Visit Window <sup>e</sup> (days relative to nominal visit) | | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>7 |
| Fall diary, daily recording | | √g | $\sqrt{h}$ | | | | √g | | $\sqrt{h}$ | | √g | $\sqrt{h}$ | | √g | $\sqrt{h}$ | | √g | $\sqrt{h}$ | | | | | | | |
| FeetMe® (subset) optional <sup>x</sup> | <br> <br> | √i | ! | | | | √i | | √j | | √i | √j | | √i | √j | | √i | √j | | | | | | | |
| PAMSys (subset) optional <sup>x</sup> | | √i | √j | | | | √i | | √j | | √i | √j | | √i | √j | | $\sqrt{i}$ | √j | | | | | | | |
| MRI scan: vMRI, DTI and ASL measures <sup>v,w</sup> | <br> <br> <br> <br> <br> | <br> <br> | 1 | | | | | | 1 | <br> <br> | | 1 | | | | | | <b>V</b> | | | | | | √t | · |
| CSF sampling <sup>k</sup> for NfL and t-tau | <br> <br> <br> <br> | | 1 | | | | | | <br> <br> <br> <br> <br> | <br> <br> | | | | | | | | <b>V</b> | | | | | | √u | |
| Blood sampling for NfL | | | | | | | | | 1 | | | $\sqrt{}$ | | | <b>V</b> | | | | | | | | | $\sqrt{}$ | |
| Quality of Life Assessment | s | | | | | | | | | | | | | | | | | | | | | | | | |
| EQ-5D-5L | | | 1 | | | | | | | | | | | | | | | | | | | | | $\sqrt{}$ | |
| Pharmacokinetic Assessme | ents | | | | | | | | | | | | | | | | | | | | | | | | |
| Blood sampling for IMP quantification <sup>1</sup> | | | √l | | 1 | <b>V</b> | <b>V</b> | | $\sqrt{l}$ | | | 1 | | | √l | | | 1 | | | 1 | | | √ | <b>V</b> |
| CSF sampling <sup>k</sup> for IMP quantification | [<br> | | 1 | | | | | | | | | | | | | | | 1 | | | | | | √u | |
| Target Engagement Assess | mei | nts | | | | | | | | | | | | | | | | | | | | | | | |
| CSF sampling <sup>k</sup> for α-synuclein and pathological species of α-synuclein | | | 1 | | | | | | | | | | | | | | | 1 | | | | | | √u | |
| Blood sampling for α-synuclein <sup>l</sup> | | | √l | | √ | 1 | 1 | | √l | | | 1 | | | √l | | | <b>V</b> | | | <b>V</b> | | | <b>V</b> | V |
| Safety Assessments | | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse events | | | V | | | 1 | 1 | 1 | V | V | V | $\sqrt{}$ | <b>V</b> | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | <b>V</b> | $\sqrt{}$ | <b>V</b> | 1 | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | |
| Follow-up of adverse<br>events on-going at EoT or<br>withdrawal, and new AEs<br>and SAEs | | | | | | | | | | | | | | | | | | | | | | | | | <b>V</b> |
| Blood and urine sampling<br>for clinical safety labora-<br>tory tests | 1 | | √ | | √ | √ | <b>V</b> | | 1 | | | 1 | | | 1 | | | <b>V</b> | | | √ | | | √ | 1 |
| Blood sampling for ADAs | | | | | | | | | 1 | | | $\sqrt{}$ | | | $\sqrt{}$ | | | | | | 1 | | | $\sqrt{}$ | $\sqrt{}$ |
| Vital signs <sup>m</sup> | <br> | j | | | | <b>√</b> | | | 1 | 1 | | $\sqrt{}$ | <b>V</b> | √ | $\sqrt{}$ | √ | <b>√</b> | | <b>√</b> | <b>V</b> | 1 | √ | <b>V</b> | $\sqrt{}$ | 1 |
| Weight | 1 | [ | $\sqrt{}$ | [ | [ | | | | 1 | [· | | 1 | | | $\sqrt{}$ | | | | | | | | | $\sqrt{}$ | : <br> |
| Examinations (physical, neurological) <sup>n</sup> | 1 | | 1 | | √ | √ | | | 1 | | | 1 | | | <b>V</b> | | | √ | | | | | | √ | |
| ECG | 1 | | | | | | | | | | | √ | | | | | | √ | | | | | | $\sqrt{}$ | |
| MRI scan for safetyw | [ | | | | | | | | 1 | | | 1 | | | | | | √ | | | | | | $\sqrt{t}$ | |
| C-SSRS° | 1 | | | | | <b>V</b> | √ | | | | | √ | | $\sqrt{}$ | √ | $\sqrt{}$ | | | | | √ | √ | | $\sqrt{}$ | $\sqrt{}$ |

| | | | | | | | | | | | | | | | | | | | | | | | | | <del></del> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Name | Screening | Randomization | Baseline + IMP | Telephone Visit | IMP | Site Visit | IMP | Telephone Visit | IMP | IMP | IMP | IMP | IMP | IMP | IMP | IMP | IMP | $\mathrm{IMP/EoT}^{\mathrm{a}}$ | $\mathrm{IMP/EoT}^{\mathrm{a}}$ | $\mathrm{IMP/EoT}^{\mathrm{a}}$ | IMP/EoT <sup>a</sup> | $\mathrm{IMP/EoT}^{\mathrm{a}}$ | $\mathrm{IMP/EoT}^{\mathrm{a}}$ | EoT/Withdrawal <sup>b</sup> | ${\rm SFU}^c$ |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 |
| Week <sup>d</sup> | 6 | -2 | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | 56 | 60 | 64 | 68 | 72 | 88 |
| Visit Window <sup>e</sup> (days relative to nominal visit) | | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>3 | ±<br>7 |
| Biobanking | | | | | | | | | | | | | | | | | | | | | | | | | |
| Blood sampling for gene expression profiling (RNA) <sup>p</sup> | | | V | | | | | | | | | 1 | | | | | | 1 | | | | | | | |
| Blood sampling for metabolomics/proteomics (plasma) <sup>p</sup> | | | V | | | | | | | | | V | | | | | | V | | | | | | | |
| Blood sampling for pharmacogenetics (DNA) (optional) <sup>q</sup> | | | V | | | | | | | | | | | | | | | | | | | | | | |
| Blood sampling for ADA | | | √ | | √ | $\sqrt{}$ | 1 | | √ | | | $\sqrt{}$ | | | 1 | | | √ | | | √ | | | $\sqrt{}$ | 1 |
| CSF sampling <sup>k</sup> | | | $\sqrt{}$ | | | | | | | | | | | | | | | $\sqrt{}$ | | | | | | $\sqrt{u}$ | |
| Other Study Procedures a | nd A | Asse | ssm | ents | 5 | | | | | | | | | | | | | | | | | | | | |
| IMP administration <sup>m</sup> | | | 1 | | √ | | 1 | | <b>√</b> | ! | | 1 | | 1 | 1 | <b>√</b> | 1 | $\sqrt{}$ | 1 | 1 | √ | 1 | 1 | | |
| Concomitant medication (prescription and non-prescription) | √ | 1 | √ | 1 | <b>V</b> | 1 | 1 | 1 | <b>V</b> | 1 | 1 | 1 | √ | 1 | 1 | √ | 1 | √ | √ | 1 | √ | <b>V</b> | √ | √ | 1 |
| Pregnancy test, urine dip-<br>stick <sup>r</sup> | | 1 | √ | | √ | | 1 | | 1 | √ | √ | 1 | √ | 1 | 1 | √ | 1 | √ | √ | √ | √ | √ | 1 | √ | √ |
| Exit interview (subset)s | | | | | | | | | | | | | | | | | | | | | | _ | | $\sqrt{}$ | |

ADA = Anti-Drug Antibody; AE = adverse event; ASL = arterial spin label; BL = baseline; CGI-S = Clinical Global Impression – Severity of Illness; CSF = cerebrospinal fluid; C-SSRS = Columbia-Suicide Severity Rating Scale; COMPASS = Composite Autonomic System Score; DNA = deoxyribonucleic acid; DTI = diffusion-tensor imaging; ECG = electrocardiogram; EoT = End-of-Treatment; EQ-5D-5L = Euroqol 5 Dimensions-5 Levels; IMP = investigational medicinal product; IRT = Interactive Response Technology; MoCA = Montreal Cognitive Assessment; MSA-C = Multiple System Atrophy with predominant cerebellar features; MSA-P = Multiple System Atrophy with predominant parkinsonism; MRI = magnetic resonance imaging; NfL = Neurofilament Light chain; OGI-S = Observer-rated Global Impression-Severity of Illness; PGI-S = Patient Global Impression-Severity of Illness; SAE = serious adverse event; SE-ADL = Schwab & England Activities of Daily Living; SFU = Safety Follow-up of DBP; SCR = screening; T-tau = total tau; UMSARS = Unified Multiple System Atrophy Rating Scale; vMRI = volumetric magnetic resonance imaging

a. When the last patient randomized reaches Visit 18/Week 48, the remaining patients in the double-blind treatment period will have their next scheduled visit converted to an EoT Visit (assessments as listed for Visit 24, no IMP administration).

b. Patients who withdraw, except for those who withdraw their consent, will be asked to attend a Withdrawal Visit as soon as possible.

c. The Safety Follow-up Visit will take place 20 weeks after last IMP administration. This will apply only to patients who do not enter the OLE or if timing of the safety FU will be before their first visit in the OLE.

- d. All assessments may be completed over a maximum of 2 consecutive days (except for MRI, see footnote w); if so, the first day is considered the "visit" day according to the schedule and at IMP Visits, IMP must be registered in IRT and administered on the second day. The Screening Visit can be performed over 2 days during the first week of the Screening Period.
- e. If the date of a visit does not conform to the schedule, subsequent visits should be planned to maintain the visit schedule relative to screening for Visit 2 and Visit 3 and relative to baseline for visits after baseline.
- f. MRI scan for eligibility can be performed between Visit 1 and Visit 2. The MRI scan should be uploaded for central reading no later than ten calendar days before the Randomization Visit.
- g. Dispense fall diary. This does not apply to a patient who scores 4 on UMSARS Part I item 7 (walking) or if the patient is wheelchair bound for unrelated disorders. This needs to be evaluated at each visit, where the fall diary is dispensed.
- h. Return of the fall diary. Patients who withdraw during a period with fall diary entries must return the diary at the Withdrawal Visit.
- i. Sensor subset: at the US sites, the patients can participate in an optional objective sensor-based assessments subset. The patients undergoing the additional objective sensor-based assessments must provide specific consent as part of the main *Informed Consent Form*. The patient does not have to consent to both objective sensor-based assessments to participate. The sensor(s) will be applied during the clinic visit. The use of the sensors does not apply to a patient who scores 4 on UMSARS Part I item 7 (walking) or if the patient is wheelchair bound for unrelated disorders. This needs to be evaluated at each visit, where the sensors are dispensed.
- j. Return of the sensor(s). Patients who withdraw during a period with objective sensor-based assessments must return the sensor(s) at the Withdrawal Visit.
- k. CSF sampling not applicable for patients with contraindications of lumbar puncture, history of severe post-lumbar puncture headache, on-going skin infection at the lumbar puncture injection site or documented history of vertebral deformities, major lumbar back surgery, clinically significant back pain, clinically significant abnormal x-ray, and/or injury that, in the opinion of the investigator, would preclude CSF collection. CSF sampling, when performed at baseline, should be completed prior to IMP administration.
- l. Multiple samples to be taken relative to IMP infusion: before infusion (at the same time as sampling for clinical safety laboratory tests), immediately after the end of infusion (EOI), 1 and 2 hours after EOI at baseline, Week 12 and Week 36. At all other visits with blood PK and  $\alpha$ -synuclein sampling, samples will be taken before infusion.
- m. Blood pressure and pulse will be measured immediately prior to IMP administration and patients will be monitored after IMP administration for immediate drug reactions for a minimum of 2 hours with vital signs taken every 30 minutes (±5 minutes) or until stable, whichever is later.
- n. Including recording of use of feeding tube and/or wheelchair.
- o. Different versions will be used: 'Baseline/Screening' version at Visit 1 and at Visit 3 and 'Since last visit' version at subsequent visits.
- p. Exploratory gene expression profiling (RNA) and metabolomics/proteomics are an integrated part of the study and are covered by the main *Informed Consent Form*.
- q. Sampling for pharmacogenetics is optional and a separate signed *Informed Consent Form* must be in place to cover this analysis.
- r. If positive, confirm with serum pregnancy test.
- s. Exit Interview subset: at the US sites, the patients and caregivers will undergo the Exit interviews via telephone or web conferencing platform (e.g., Microsoft Teams). The Exit interview will be conducted within 3 weeks after the EoT Visit or within 3 weeks after the Withdrawal Visit for patients who reach a 48-week treatment period but withdraw prior to the EoT Visit. Study Experience Interview subset: at US sites, a subset of patients and caregivers may be contacted to participate in a Study Experience interview by telephone or web conferencing platform (e.g., Microsoft Teams). The Study Experience interview will be conducted within 6 weeks after the completed Exit interview for patients who consent.
- t. MRI scanning only to be performed as EoT/withdrawal procedure if not performed within the last 8 weeks.
- u. CSF sampling only to be performed as withdrawal procedure in case of withdrawal prior to Visit 18/Week 48 and for patients with EoT at Visit 18/Week 48. Patients with EoT after Visit 18/Week 48 will not undergo CSF sampling as part of the EoT procedures.

- v. DTI and ASL measures where available. If Visit 3 MRI scanning is performed without DTI and/or ASL sequences and these sequences are implemented in the scanner at a later stage, DTI and ASL should not be performed at subsequent visits with MRI measurements.
- w. MRI scan can be performed any day within the Visit Window, except for Visit 3 where it must be performed before IMP administration. Date of MRI scan will not define Day 1 or Day 2 of a visit and will not be regarded as a separate visit.
- x. Participation in FeetMe® and PAMSys subsets are optional, but informed consent for these are part of the main informed consent. The use of the sensors does not apply to a patient who scores 4 on UMSARS Part I item 7 (walking) or if the patient is wheelchair bound for unrelated disorders. This needs to be evaluated at each visit, where the sensors are to be dispensed.

Table 2 Optional Open-label Long-term Extension Treatment Period

| <u>Visit Name</u> | Base<br>line -<br>IMP | <u>IMP</u> | <u>IMP</u> | <u>IMP</u> | <u>IMP</u> | <u>IMP</u> | <u>IMP</u> | <u>IMP</u> | <u>IMP</u> | <u>IMP</u> | <u>IMP</u> | <u>IMP</u> | End of Ope n- La- bel Trea tmen | | Safet Y Fol- low- up <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | <u>1E</u> | <u>2E</u> | <u>3E</u> | <u>4E</u> | <u>5E</u> | <u>6E</u> | <u>7E</u> | <u>8E</u> | <u>9E</u> | <u>10E</u> | <u>11E</u> | <u>12E</u> | <u>13E</u> | <u>WD</u> | SFU-<br>E |
| Week <sup>c</sup> | <u>0E</u> | <u>4E</u> | <u>8E</u> | <u>12E</u> | <u>16E</u> | <u>20E</u> | <u>24E</u> | <u>28E</u> | <u>32E</u> | <u>36E</u> | <u>40E</u> | <u>44E</u> | <u>48E</u> | | <u>64E</u> |
| Visit Window <sup>d</sup> (days relative to nominal visit) | | <u>±3</u> | <u>±3</u> | <u>±3</u> | <u>±3</u> | <u>±3</u> | <u>±3</u> | <u>±3</u> | <u>±3</u> | <u>±3</u> | <u>±3</u> | <u>±3</u> | <u>±3</u> | | <u>±7</u> |
| Signed informed consent | _√ | | | i<br>I | ! | | | | | İ | | | | | i . |
| Efficacy Assessments | | | | | | | | | | | | | | | |
| UMSARS | <u>√e</u> | l | l | _√ | -<br>!<br>! | | 1/2 | | <br> | √ | <br> | | 1 √ | √ | i<br>i |
| <u>CGI-S</u> | √e | | | √ | 7<br>! | | √ | | i | √ | | ; | $\sqrt{}$ | √ | î<br>! |
| <u>PGI-S</u> | <u>√</u> e | - | - | √ | - | | √ | - | - | √ | - | | √ | √ | +<br>!<br>! |
| SE-ADL | <u>√e</u> | - | - | | <br> | <br> | √_ | <br> | | ·<br> | | <br> | 1 √ | _√ | f<br>' |
| EQ-5D-5L | <u>√e</u> | - | - | <br>! | <br>! | : | √ | :<br> | - | ·<br> <br> | <br> <br> | <br> <br> | √ | _√ | t<br>! |
| MRI scans: vMRIf | $\sqrt{e,g}$ | - | <br> | <br> | <br> <br> | | | - | - | - | <br> | | _√ | _√ | †<br>! |
| Blood sampling for NfL | √ | | | | <del> </del><br> | | <u>√</u> | | | | | | √ | √ | !<br>! |
| Pharmacokinetic Assessme | <u>ents</u> | | | | | | | | | | | | | | <u>. </u> |
| Blood sampling for IMP quantification | <u>√</u> e | | | l<br>I | | | <u>√</u> | | | l<br>I | <br> | <br> | √_ | √ | <u>√</u> |
| Pharmacodynamic Assessi | <u>ments</u> | | | | | | | | | | | | | | |
| Blood sampling for α-<br>synuclein | <u>√</u> e | <br> | <br> | | Ī | | √ | <br> | | | | | √ | √ | √ |
| Safety Assessments | | | | | | | | | | | | | | | |
| Adverse events | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ |

| Blood and urine sampling<br>for clinical safety labora-<br>tory tests | <u>√e</u> | <br> <br> <br> | <b></b><br> - | <br> <br> <br> | | | <u>√</u> | :<br>! : : | | <b></b> 1 | | <br> <br> <br> | $\sqrt{}$ | √_ | ( 7<br>! ! |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <u>Vital signs<sup>h</sup></u> | _ √ | √ | <u>√</u> | √ | √ | √ | _√ | √ | √ | √ | √ | _√ | √ | √ | , |
| Examinations <sup>i</sup> (physical, neurological) | <u>√</u> e | <br> <br> | - | | <br>i<br>i | | √ | | | | | <b>; </b> | √ | √ | ; |
| C-SSRS since last visit | <u>√</u> e | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ |
| Biobanking | | | | | | | | | | | | | | | |
| Blood sampling for ADA | √e | | ]<br>] | | | | √ | l<br>! | | | | | √ | $\sqrt{}$ | √ |
| Other Study Procedures a | nd Ass | sessme | ents | <b></b> ' | | | | | | | | | | | |
| IMP administration <sup>h</sup> | _√ | √ | _√ | √ | √ | √_ | √ | <u>√</u> | √ | √ | √ | √ | | i<br>I I | |
| Concomitant medication | √ | √ | <u>√</u> | √ | √_ | $\underline{\checkmark}$ | $\underline{\checkmark}$ | √_ | $\underline{\checkmark}$ | $\underline{\checkmark}$ | $\underline{\checkmark}$ | √ | $\underline{\checkmark}$ | $\underline{\checkmark}$ | √ |
| Urine pregnancy test <sup>j</sup> | | √ | _√ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | √ | |

ADA = Anti-Drug Antibody; CGI-S = Clinical Global Impression – Severity of Illness; C-SSRS = Columbia-Suicide Severity Rating Scale; EQ-5D-5L = Euroqol 5 Dimensions-5 Levels; IMP = investigational medicinal product; PGI-S = Patient Global Impression-Severity of Illness; SE-ADL: Schwab & England Activities of Daily Living; SFU-E = Safety Follow-up OLE; UMSARS = Unified Multiple System Atrophy Rating Scale; vMRI = volumetric magnetic resonance imaging; WD = withdrawal

- a Participants who withdraw, except for those who withdraw their consent, will be asked to attend a Withdrawal Visit as soon as possible.
- b The Safety Follow-up Visit will take place 16 weeks after Visit 13E / 20 weeks after last IMP administration in case of withdrawal (follow-up of adverse events on-going at EoT or withdrawal, and new AEs and SAEs).
- b All assessments may be completed over a maximum of 2 days (except for MRI, see footnote e); if so, the first day is considered the "visit" day according to the schedule and at IMP visits, IMP must be registered in IRT and administered on the second day.
- d If the date of a visit does not conform to the schedule, subsequent visits should be planned to maintain the visit schedule relative to Visit 1E. o
- e Only applicable for patients who enter the OLE more than 1 week later as the EoT Visit in the double-blind treatment period.
- f MRI scan can be performed any day within the Visit Window. Date of MRI scan will not define Day 1 or Day 2 of a visit and will not be regarded as a separate visit.
- g MRI scanning only to be performed as Visit 1E if not performed within the last 8 weeks.
- h Blood pressure and pulse will be measured immediately prior to IMP administration and patients will be monitored after IMP administration for immediate drug reactions for a minimum of 2 hours with vital signs taken every 30 minutes (±5 minutes) or until stable, whichever is later.
- i Including recording of use of feeding tube and/or wheelchair.
- j Only for women of childbearing potential. If positive, confirm with serum pregnancy test.

### Appendix V PCS Criteria

#### **PCS** Criteria

 Table 3
 PCS Criteria for Clinical Safety Laboratory Tests

| Laboratory Test | CDISC Term | Unit | PCS Low | PCS High |
|---|---|---|---|---|
| Haematology / Coagulation | | | | |
| B-haemoglobin | HGB | g/L | ≤ 95 (women) | ≥ 165 (women) |
| | | | ≤ 115 (men) | ≥ 185 (men) |
| B-erythrocytes (red cell count) | RBC | x 10E12/L | $\leq$ 3.5 (women) | $\geq$ 6.0 (women) |
| | | | $\leq$ 3.8 (men) | $\geq 7.0 \text{ (men)}$ |
| B-haematocrit (packed cell volume) | HCT | V/V | ≤ 0.32 (women) | ≥ 0.50 (women) |
| | | | $\leq$ 0.37 (men) | $\geq 0.55 \text{ (men)}$ |
| B-MCV (mean cell volume) | MCV | fL | $\leq$ 0.8 x LLN | ≥ 1.2 x ULN |
| B-total leucocyte (white cell count) | WBC | x 10E9/L | ≤ 2.8 | ≥16 |
| B-neutrophils/leucocytes | NEUTLE | % | $\leq$ 20 | ≥ 85 |
| B-eosinophils/leucocytes | EOSLE | % | | ≥ 10 |
| B-basophils/leucocytes | BASOLE | % | | ≥ 10 |
| B-lymphocytes/leucocytes | LYMLE | % | ≤ 10 | ≥ 75 |
| B-monocytes/leucocytes | MONOLE | % | | ≥ 15 |
| B-thrombocytes (platelet count) | PLAT | x 10E9/L | ≤ 75 | $\geq 600$ |
| P-INR (prothrombin ratio) | INR | Ratio | | $\geq 2.0$ |
| B-prothrombin time | PT | Sec | | ≥ 18 |
| Liver | | | | |
| S-aspartate aminotransferase | AST | U/L | | $\geq$ 3 × ULN |
| S-alanine aminotransferase | ALT | U/L | | $\geq$ 3 × ULN |
| S-bilirubin | BILI | μmol/L | | ≥ 34 |
| S-bilirubin, direct | BILDIR | μmol/L | | ≥ 12 |
| S-bilirubin, indirect | BILIND | μmol/L | | ≥ 22 |
| S-alkaline phosphatase | ALP | U/L | | $\geq$ 3 × ULN |
| S-gamma glutamyl transferase | GGT | U/L | | $\geq 200$ |
| S-alpha-glutathione S-transferase (alpha-GST) | GSTAL | μg/L | | ≥ 20 |
| Kidney | | | | |
| S-creatinine | CREAT | μmol/L | | ≥ 1.5 x ULN |
| B-urea nitrogen (BUN) | BUN | mmol/L | | ≥ 11 |
| S-uric acid (urate) | URATE | μmol/L | | ≥ 510 (women) |
| | | | | ≥ 630 (men) |
| Electrolytes | | | | |
| S-sodium (natrium) | SODIUM | mmol/L | ≤ 125 | ≥ 155 |
| S-potassium (kalium) | K | mmol/L | $\leq$ 3.0 | $\geq 6.0$ |

| <b>Laboratory Test</b> | CDISC Term | Unit | PCS Low | PCS High |
|---|---|---|---|---|
| S-calcium | CA | mmol/L | ≤ 1.8 | ≥ 3.0 |
| S-chloride | CL | mmol/L | ≤ 90 | ≥ 117 |
| S-magnesium | MG | mmol/L | $\leq 0.6$ | ≥ 1.3 |
| S-phosphate (phosphorus, (inorganic) | PHOS | mmol/L | ≤ 0.65 | ≥ 1.95 |
| S-bicarbonate | BICARB | mmol/L | ≤ 12 | ≥38 |
| Endocrine / Metabolic | | | | |
| B-glucose, non-fasting/unknown | GLUC | mmol/L | ≤ 3.4 | ≥ 9.4 |
| B-glucose, fasting | GLUC | mmol/L | $\leq$ 3.0 | $\geq 6.0$ |
| S-glucose, non-fasting/unknown | GLUC | mmol/L | ≤ 3.9 | ≥ 11.1 |
| S-glucose, fasting | GLUC | mmol/L | ≤ 3.5 | $\geq 7.0$ |
| B-glycosylated haemoglobin, fasting | HBA1C | Hb fract. | | ≥ 0.065 |
| S-prolactin | PROLCTN | mIU/L | | ≥ 1350 |
| S-thyrotropin/TSH | TSH | mIU/L | $\leq 0.3$ | ≥ 5.5 |
| S-protein (total) | PROT | g/L | ≤ <b>4</b> 5 | ≥ 95 |
| S-albumin | ALB | g/L | ≤ 27 | |
| Lipids | | | | |
| S-cholesterol total, non-fasting/unknown | CHOL | mmol/L | | ≥ 7.8 |
| S-cholesterol total, fasting | CHOL | mmol/L | | $\geq$ 6.2 |
| S-triglycerides, non-<br>fasting/unknown | TRIG | mmol/L | | ≥ 5.65 |
| S-triglycerides, fasting | TRIG | mmol/L | | ≥ 4.2 |
| S-LDL cholesterol, non-fasting/unknown | LDL | mmol/L | | ≥ 5.3 |
| S-LDL cholesterol, fasting | LDL | mmol/L | | ≥ 4.9 |
| S-HDL cholesterol, non-fasting/unknown | HDL | mmol/L | ≤ 0.8 | |
| S-HDL cholesterol, fasting | HDL | mmol/L | $\leq 0.9$ | |
| Cardiac/Skeletal/Muscle | | | | |
| S-creatine kinase (total) | CK | U/L | | ≥ 400 (women)<br>≥ 750 (men) |
| S-creatine kinase MB isoenzyme | CKMB | μg/L | | $\geq 8.5$ or |
| • | CKMBCK | % | | $\geq$ 3.5% of total CK |
| S-lactate dehydrogenase (total) | LDH | IU/L | | ≥ 750 |
| S-troponin I | TROPONI | μg/L | | ≥ 1.5 |
| S-troponin T | TROPONT | μg/L | | $\geq 0.4$ |
| Infection | | | | |
| S-C-reactive protein | CRP | mg/L | | ≥ 25 |
| S-globulin (total) | GLOBUL | g/L | ≤ 15 | ≥ 55 |
| Urine Urine | • | | <del>-</del> - | · |

| Laboratory Test | CDISC Term | Unit | PCS Low | PCS High |
|-----------------|------------|------|------------|----------|
| Urinary pH | PH | | ≤ <b>4</b> | ≥ 9 |

S=serum; B=whole blood; U=urine

Table 4 PCS Criteria for Vital Signs, Weight/BMI, and Waist Circumference

| Variable | CDISC Term | Unit | PCS Low | PCS High |
|---|---|---|---|---|
| Waist circumference | WSTCIR | Cm | decrease ≥ 7% | increase ≥ 7% |
| Weight | WEIGHT | Kg | $decrease \geq 7\%$ | increase $\geq 7\%$ |
| Body Mass Index | BMI | kg/m2 | $decrease \geq 7\%$ | increase $\geq 7\%$ |
| Pulse rate,<br>supine/sitting/unknown | PULSE | beats/min | $<$ 50 and decrease $\ge$ 15 | $\geq$ 120 and increase $\geq$ 15 |
| Diastolic blood pressure, supine/sitting/unknown | DIABP | mmHg | $\leq$ 50 and decrease $\geq$ 15 | $\geq$ 105 and increase $\geq$ 15 |
| Systolic blood pressure, supine/sitting/unknown | SYSBP | mmHg | $\leq$ 90 and decrease $\geq$ 20 | $\geq$ 180 and increase $\geq$ 20 |
| Orthostatic systolic blood pressure | OBP | mmHg | ≤ -30 | |
| Orthostatic pulse rate | OPR | beats/min | | ≥ 20 |
| Temperature | TEMP | °C | decrease $\geq 2$ | $\geq$ 38.3 and increase $\geq$ 2 |

Increase/decrease is relative to the baseline value.

**Table 5** PCS Criteria for ECG Parameters

| ECG Parameter | CDISC Term | Unit | PCS Low | PCS High |
|---|---|---|---|---|
| Absolute Time Interval | | | | |
| PR interval | PRAG | Msec | | ≥ 260 |
| QRS interval | QRSAG | Msec | | ≥ 150 |
| QT interval | QTAG | Msec | | ≥ 500 |
| <b>Derived Time Interval</b> | | | | |
| Heart rate | EGHRMN | beats/min | $<$ 50 and decrease $\ge$ 15 | $\geq$ 120 and increase $\geq$ 15 |
| QTcB interval | QTCBAG | Msec | < 300 | > 500 or increase > 60 |
| QTcF interval | QTCFAG | Msec | < 300 | > 500 or increase > 60 |

Increase/decrease is relative to the baseline value.

# Appendix VI Definition of Hypersensitivity related reactions

### **Definition of Hypersensitivity related reactions**

Type I hypersensitivity reaction: Anaphylaxis

SEARCH: TEAEs with a PT within the SMQ of Hypersensitivity (narrow scope)

| Hypersensitivity (SMQ): | |
|--------------------------------------------|----------|
| Acquired C1 inhibitor deficiency | 10081035 |
| Acute generalised exanthematous pustulosis | 10048799 |
| Administration related reaction | 10069773 |
| Administration site dermatitis | 10075096 |
| Administration site eczema | 10075099 |
| Administration site hypersensitivity | 10075102 |
| Administration site rash | 10071156 |
| Administration site recall reaction | 10075964 |
| Administration site urticaria | 10075109 |
| Administration site vasculitis | 10075969 |
| AGEP-DRESS overlap | 10089003 |
| Allergic bronchitis | 10052613 |
| Allergic colitis | 10059447 |
| Allergic cough | 10053779 |
| Allergic cystitis | 10051394 |
| Allergic eosinophilia | 10075185 |
| Allergic gastroenteritis | 10075308 |
| Allergic hepatitis | 10071198 |
| Allergic keratitis | 10057380 |
| Allergic lymphangitis | 10086007 |
| Allergic oedema | 10060934 |
| Allergic otitis externa | 10075072 |
| Allergic otitis media | 10061557 |
| Allergic pharyngitis | 10050639 |
| Allergic reaction to excipient | 10078853 |
| Allergic respiratory disease | 10063532 |
| Allergic respiratory symptom | 10063527 |
| Allergic sinusitis | 10049153 |
| Allergic stomatitis | 10079554 |
| Allergic transfusion reaction | 10066173 |
| Allergy alert test positive | 10075479 |
| Allergy test positive | 10056352 |
| Allergy to immunoglobulin therapy | 10074079 |
| Allergy to surgical sutures | 10077279 |
| Allergy to vaccine | 10055048 |

| Anal eczema | 10078682 |
|----------------------------------------------------------|----------|
| Anaphylactic reaction | 10002198 |
| Anaphylactic shock | 10002199 |
| Anaphylactic transfusion reaction | 10067113 |
| Anaphylactoid reaction | 10002216 |
| Anaphylactoid shock | 10063119 |
| Anaphylaxis treatment | 10002222 |
| Angioedema | 10002424 |
| Antiallergic therapy | 10064059 |
| Antiendomysial antibody positive | 10065514 |
| Anti-neutrophil cytoplasmic antibody positive vasculitis | 10050894 |
| Application site dermatitis | 10003036 |
| Application site eczema | 10050099 |
| Application site hypersensitivity | 10063683 |
| Application site rash | 10003054 |
| Application site recall reaction | 10076024 |
| Application site urticaria | 10050104 |
| Application site vasculitis | 10076027 |
| Arthritis allergic | 10061430 |
| Atopic cough | 10081492 |
| Atopy | 10003645 |
| Blepharitis allergic | 10005149 |
| Blood immunoglobulin E abnormal | 10005589 |
| Blood immunoglobulin E increased | 10005591 |
| Bone cement allergy | 10087325 |
| Bromoderma | 10006404 |
| Bronchospasm | 10006482 |
| Bullous haemorrhagic dermatosis | 10083809 |
| Catheter site dermatitis | 10073992 |
| Catheter site eczema | 10073995 |
| Catheter site hypersensitivity | 10073998 |
| Catheter site rash | 10052271 |
| Catheter site urticaria | 10052272 |
| Catheter site vasculitis | 10074014 |
| Chronic eosinophilic rhinosinusitis | 10071399 |
| Chronic hyperplastic eosinophilic sinusitis | 10071380 |
| Circulatory collapse | 10009192 |
| Circumoral oedema | 10052250 |
| Circumoral swelling | 10081703 |
| Conjunctival oedema | 10010726 |
| Conjunctivitis allergic | 10010744 |
| Contact stomatitis | 10067510 |
| Contrast media allergy | 10066973 |
| Contrast media reaction | 10010836 |

| Corneal oedema | 10011033 |
|-------------------------------------------------------|----------|
| Cross sensitivity reaction | 10011411 |
| Cutaneous vasculitis | 10011686 |
| Dennie-Morgan fold | 10062918 |
| Dermal filler reaction | 10086476 |
| Dermatitis | 10012431 |
| Dermatitis acneiform | 10012432 |
| Dermatitis allergic | 10012434 |
| Dermatitis atopic | 10012438 |
| Dermatitis bullous | 10012441 |
| Dermatitis contact | 10012442 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Dermatitis herpetiformis | 10012468 |
| Dermatitis infected | 10012470 |
| Dermatitis psoriasiform | 10058675 |
| Device allergy | 10072867 |
| Dialysis membrane reaction | 10076665 |
| Distributive shock | 10070559 |
| Documented hypersensitivity to administered product | 10076470 |
| Drug eruption | 10013687 |
| Drug hypersensitivity | 10013700 |
| Drug provocation test | 10074350 |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Eczema | 10014184 |
| Eczema infantile | 10014198 |
| Eczema nummular | 10014201 |
| Eczema vaccinatum | 10066042 |
| Eczema vesicular | 10058681 |
| Eczema weeping | 10055182 |
| Encephalitis allergic | 10056387 |
| Encephalopathy allergic | 10014627 |
| Eosinophilic granulomatosis with polyangiitis | 10078117 |
| Epidermal necrosis | 10059284 |
| Epidermolysis | 10053177 |
| Epidermolysis bullosa | 10014989 |
| Epiglottic oedema | 10015029 |
| Erythema multiforme | 10015218 |
| Erythema nodosum | 10015226 |
| Exfoliative rash | 10064579 |
| Eye allergy | 10015907 |
| Eye oedema | 10052139 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |

| Face oedema | 10016029 |
|--------------------------------------------|----------|
| Fixed eruption | 10016741 |
| Generalised bullous fixed drug eruption | 10084905 |
| Giant papillary conjunctivitis | 10018258 |
| Gingival oedema | 10049305 |
| Gingival swelling | 10018291 |
| Gleich's syndrome | 10066837 |
| Haemorrhagic urticaria | 10059499 |
| Hand dermatitis | 10058898 |
| Henoch-Schonlein purpura | 10019617 |
| Henoch-Schonlein purpura nephritis | 10069440 |
| Heparin-induced thrombocytopenia | 10062506 |
| Hypersensitivity | 10020751 |
| Hypersensitivity myocarditis | 10081004 |
| Hypersensitivity pneumonitis | 10081988 |
| Hypersensitivity vasculitis | 10020764 |
| Idiopathic urticaria | 10021247 |
| Immediate post-injection reaction | 10067142 |
| Immune thrombocytopenia | 10083842 |
| Immune tolerance induction | 10070581 |
| Implant site dermatitis | 10063855 |
| Implant site hypersensitivity | 10063858 |
| Implant site rash | 10063786 |
| Implant site urticaria | 10063787 |
| Incision site dermatitis | 10073168 |
| Incision site rash | 10073411 |
| Infusion related hypersensitivity reaction | 10082742 |
| Infusion related reaction | 10051792 |
| Infusion site dermatitis | 10065458 |
| Infusion site eczema | 10074850 |
| Infusion site hypersensitivity | 10065471 |
| Infusion site rash | 10059830 |
| Infusion site recall reaction | 10076085 |
| Infusion site urticaria | 10065490 |
| Infusion site vasculitis | 10074851 |
| Injection related reaction | 10071152 |
| Injection site dermatitis | 10022056 |
| Injection site eczema | 10066221 |
| Injection site hypersensitivity | 10022071 |
| Injection site rash | 10022071 |
| Injection site recall reaction | 10066797 |
| Injection site urticaria | 10000777 |
| Injection site vasculitis | 10022107 |
| Instillation site hypersensitivity | 10007993 |
| insulation site hypersonsitivity | 100/3012 |

| Instillation site rash | 10073622 |
|-------------------------------------------------|----------|
| Instillation site urticaria | 10073627 |
| Interstitial granulomatous dermatitis | 10067972 |
| Intestinal angioedema | 10076229 |
| Iodine allergy | 10052098 |
| Kounis syndrome | 10069167 |
| Laryngeal oedema | 10023845 |
| Laryngitis allergic | 10064866 |
| Laryngospasm | 10023891 |
| Laryngotracheal oedema | 10023893 |
| Limbal swelling | 10070492 |
| Lip oedema | 10024558 |
| Lip swelling | 10024570 |
| Mast cell activation syndrome | 10075217 |
| Mast cell degranulation present | 10076606 |
| Medical device site dermatitis | 10075572 |
| Medical device site eczema | 10075575 |
| Medical device site hypersensitivity | 10075579 |
| Medical device site rash | 10075585 |
| Medical device site recall reaction | 10076140 |
| Medical device site urticaria | 10075588 |
| Mouth swelling | 10075203 |
| Mucocutaneous rash | 10056671 |
| Multiple allergies | 10028164 |
| Nephritis allergic | 10029120 |
| Nikolsky's sign | 10029415 |
| Nodular rash | 10075807 |
| NSAID exacerbated respiratory disease | 10087423 |
| Nutritional supplement allergy | 10084049 |
| Oculomucocutaneous syndrome | 10030081 |
| Oculorespiratory syndrome | 10067317 |
| Oedema mouth | 10030110 |
| Oral allergy syndrome | 10068355 |
| Oropharyngeal blistering | 10067950 |
| Oropharyngeal oedema | 10078783 |
| Oropharyngeal spasm | 10031111 |
| Oropharyngeal swelling | 10031118 |
| Palatal oedema | 10056998 |
| Palatal swelling | 10074403 |
| Palisaded neutrophilic granulomatous dermatitis | 10068809 |
| Palpable purpura | 10056872 |
| Pathergy reaction | 10030872 |
| Penile dermatitis | 10074332 |
| Perioral dermatitis | 1008/419 |
| 1 Griorai definatio | 10057571 |

| Periorbital dermatitis | 10087203 |
|-----------------------------------|----------|
| Periorbital oedema | 10034545 |
| Periorbital swelling | 10056647 |
| Pharyngeal oedema | 10034829 |
| Pharyngeal swelling | 10082270 |
| Polymers allergy | 10086347 |
| Procedural shock | 10080894 |
| Pruritus allergic | 10063438 |
| Puncture site rash | 10087940 |
| Radioallergosorbent test positive | 10037789 |
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash follicular | 10037857 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |
| Rash neonatal | 10037871 |
| Rash papulosquamous | 10037879 |
| Rash pruritic | 10037884 |
| Rash pustular | 10037888 |
| Rash rubelliform | 10057984 |
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Reaction to azo-dyes | 10037973 |
| Reaction to colouring | 10037974 |
| Reaction to excipient | 10079925 |
| Reaction to flavouring | 10082681 |
| Reaction to food additive | 10037977 |
| Reaction to preservatives | 10064788 |
| Reaction to sweetener | 10086454 |
| Rhinitis allergic | 10039085 |
| Scleral oedema | 10057431 |
| Scleritis allergic | 10051126 |
| Scrotal dermatitis | 10083260 |
| Scrotal oedema | 10039755 |
| Serum sickness | 10040400 |
| Serum sickness-like reaction | 10040402 |
| Shock | 10040560 |
| Shock symptom | 10040581 |
| SJS-TEN overlap | 10083164 |
| Skin necrosis | 10040893 |
| Skin reaction | 10040914 |
| Skin test positive | 10040934 |

| Solar urticaria | 10041307 |
|----------------------------------------------------------------|----------|
| Solvent sensitivity | 10041316 |
| Stevens-Johnson syndrome | 10042033 |
| Stoma site hypersensitivity | 10074509 |
| Stoma site rash | 10059071 |
| Swelling face | 10042682 |
| Swelling of eyelid | 10042690 |
| Swollen tongue | 10042727 |
| Symmetrical drug-related intertriginous and flexural exanthema | 10078325 |
| Systemic contact dermatitis | 10087943 |
| Tattoo associated skin reaction | 10087549 |
| Tongue oedema | 10043967 |
| Toxic epidermal necrolysis | 10044223 |
| Toxic skin eruption | 10057970 |
| Tracheal oedema | 10044296 |
| Type I hypersensitivity | 10045240 |
| Type II hypersensitivity | 10054000 |
| Type III immune complex mediated reaction | 10053614 |
| Type IV hypersensitivity reaction | 10053613 |
| Urticaria | 10046735 |
| Urticaria cholinergic | 10046740 |
| Urticaria chronic | 10052568 |
| Urticaria contact | 10046742 |
| Urticaria papular | 10046750 |
| Urticaria physical | 10046751 |
| Urticaria pigmentosa | 10046752 |
| Urticaria vesiculosa | 10046755 |
| Urticarial dermatitis | 10082290 |
| Urticarial vasculitis | 10048820 |
| Vaccination site dermatitis | 10069477 |
| Vaccination site eczema | 10076161 |
| Vaccination site exfoliation | 10069489 |
| Vaccination site hypersensitivity | 10068880 |
| Vaccination site rash | 10069482 |
| Vaccination site recall reaction | 10076188 |
| Vaccination site urticaria | 10069622 |
| Vaccination site vasculitis | 10076191 |
| Vaccination site vesicles | 10069623 |
| Vaginal ulceration | 10046943 |
| Vancomycin infusion reaction | 10086737 |
| Vascular access site dermatitis | 10085938 |
| Vascular access site eczema | 10085939 |
| Vasculitic rash | 10047111 |
| Vernal keratoconjunctivitis | 10081000 |

| V1 | 10077117 |
|-------------------------------|----------|
| Vessel puncture site rash | 10077117 |
| Vessel puncture site vesicles | 10077813 |
| Vulval eczema | 10066273 |
| Vulval ulceration | 10047768 |
| Vulvovaginal rash | 10071588 |
| Vulvovaginal ulceration | 10050181 |
| Vulvovaginitis allergic | 10080783 |

Type II hypersensitivity reaction: Cytokine Release Syndrome (CRS)

SEARCH: TEAEs with the PT 'Cytokine release syndrome'

Type III hypersensitivity reaction: Immune-complex related reactions

SEARCH: TEAEs with a PT within the SMQ Vasculitis (narrow scope), or with the 15 defined PTs

| Vasculitis (SMQ): | |
|----------------------------------------------------------|----------|
| Acute haemorrhagic oedema of infancy | 10070599 |
| Administration site vasculitis | 10075969 |
| Anti-neutrophil cytoplasmic antibody positive vasculitis | 10050894 |
| Aortitis | 10002921 |
| Application site vasculitis | 10076027 |
| Arteritis | 10003230 |
| Arteritis coronary | 10003232 |
| Behcet's syndrome | 10004213 |
| Capillaritis | 10068406 |
| Central nervous system vasculitis | 10081778 |
| Cerebral arteritis | 10008087 |
| Chronic pigmented purpura | 10072726 |
| Cogan's syndrome | 10056667 |
| Cutaneous vasculitis | 10011686 |
| Diabetic arteritis | 10077357 |
| Diffuse vasculitis | 10012978 |
| Eosinophilic granulomatosis with polyangiitis | 10078117 |
| Erythema induratum | 10015213 |
| Giant cell arteritis | 10018250 |
| Granulomatosis with polyangiitis | 10072579 |
| Haemorrhagic occlusive retinal vasculitis | 10085070 |
| Haemorrhagic vasculitis | 10071252 |
| Henoch-Schonlein purpura | 10019617 |
| Henoch-Schonlein purpura nephritis | 10069440 |
| Hypersensitivity vasculitis | 10020764 |

| Infusion site vasculitis 10074851 Injection site vasculitis 10067995 Kawasaki's disease 10023320 Langerhans' cell histiocytosis 1006968 Lupus vasculitis 10058143 MAGIC syndrome 1007812 Medical device site vasculitis 10076146 Microscopic polyangiitis 10063344 Nodular vasculitis 10029491 Ocular vasculitis 1006926 Polyarteritis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 10036555 Pulmonary vasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10085059 Retinal vasculitis 10085059 Retinal vasculitis 10085059 Retinal vasculitis 10048628 Segmented hyalinising vasculitis 10047527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 1007517 Urticarial vascul | | |
|---|---|---|
| Kawasaki's disease 10023320 Langerhans' cell histiccytosis 1006968 Lupus vasculitis 10058143 MAGIC syndrome 10078132 Medical device site vasculitis 10063344 Nicroscopic polyangitis 10063344 Nodular vasculitis 10029491 Ocular vasculitis 10029491 Ocular vasculitis 10036026 Polyarteritis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 10065255 Pulmonary vasculitis 10037457 Rediation vasculitis 10038467 Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10085059 Retinal vasculitis 10048628 Segmented hyalinising vasculitis 10047327 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043097 Thromboangiitis obliterans 10043097 Urticarial vasculitis 10043097 Vascular pu | Infusion site vasculitis | 10074851 |
| Langerhans' cell histiocytosis 10069698 Lupus vasculitis 10078132 MAGIC syndrome 10076146 Microscopic polyangiitis 10063344 Nodular vasculitis 10029491 Ocular vasculitis 10029491 Ocular vasculitis 10036024 Polyarteritis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 10037457 Radiation vasculitis 10037457 Radiation vasculitis 10038373 Renal arteritis 10038373 Renial vasculitis 100385059 Retinal occlusive vasculitis 10038905 Retinal vasculitis 10038905 Retinal vasculitis 10048628 Segmented hyalinising vasculitis 1004802 Segmented hyalinising vasculitis 1004397 Thromboangiitis obliterans 1004397 Thromboangiitis obliterans 1004394 Type 2 lepra reaction 10070517 Urticarial vasculitis 10047097 Vascular purpura 10047097 Vasculitic | Injection site vasculitis | 10067995 |
| Lupus vasculitis 10058143 MAGIC syndrome 10078132 Medical device site vasculitis 10076146 Microscopic polyangiitis 10063344 Nodular vasculitis 10029491 Ocular vasculitis 10036024 Polyarretitis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10038505 Retinal vasculitis 10038905 Retinal vasculitis 10038905 Retinal vasculitis 10038905 Retinal vasculitis 10048628 Segmented hyalinising vasculitis 10048028 Segmented hyalinising vasculitis 1004797 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10047097 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10047115 Vasculitis necrotising | Kawasaki's disease | 10023320 |
| MAGIC syndrome 10078132 Medical device site vasculitis 10076146 Microscopic polyangiitis 10063344 Nodular vasculitis 10029491 Ocular vasculitis 10066926 Polyarteritis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 10037457 Radiation vasculitis 10037457 Renal arteritis 10038373 Renal vasculitis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10048628 Segmented hyalinising vasculitis 1004705 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043097 Type 2 lepra reaction 10070517 Urticarial vasculitis 10076191 Vascular purpura 10047097 Vascular purpura 10047011 Vasculitis gastrointestinal 10047115 Vasculitis pastrointestinal 10047115 | Langerhans' cell histiocytosis | 10069698 |
| Medical device site vasculitis 10076146 Microscopic polyangiitis 10063344 Nodular vasculitis 10029491 Ocular vasculitis 10066926 Polyarteritis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 10065255 Pulmonary vasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Retinal vasculitis 10048628 Segmented hyalinising vasculitis 10047527 Takayasu's arteritis 10043540 Type 2 lepra reaction 10043540 Type 2 lepra reaction 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10047097 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10047115 Vasculitis necrotising 10047124 | Lupus vasculitis | 10058143 |
| Microscopic polyangitis 10063344 Nodular vasculitis 10029491 Ocular vasculitis 10066926 Polyarteritis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 10065255 Pulmonary vasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043540 Type 2 lepra reaction 10043540 Type 2 lepra reaction 1007517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10047097 Vasculitic rash 10047011 Vasculitis gastrointestinal 10047115 Vasculitis pestrointestinal 10048319 Vasculitis necrotising 10047124 | MAGIC syndrome | 10078132 |
| Nodular vasculitis 10029491 Ocular vasculitis 10066926 Polyarteritis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 1005255 Pulmonary vasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10047527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 1004811 Vasculitis necrotising 10047115 | Medical device site vasculitis | 10076146 |
| Ocular vasculitis 10066926 Polyarteritis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 10065255 Pulmonary vasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10085059 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10047115 Vasculitis necrotising 100471124 | Microscopic polyangiitis | 10063344 |
| Polyarteritis nodosa 10036024 Polymyalgia rheumatica 10036099 Pseudovasculitis 10065255 Pulmonary vasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043997 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Nodular vasculitis | 10029491 |
| Polymyalgia rheumatica 10036099 Pseudovasculitis 10065255 Pulmonary vasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Ocular vasculitis | 10066926 |
| Pseudovasculitis 10065255 Pulmonary vasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 1004397 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Polyarteritis nodosa | 10036024 |
| Pulmonary vasculitis 10037457 Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10047097 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Polymyalgia rheumatica | 10036099 |
| Radiation vasculitis 10074671 Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Pseudovasculitis | 10065255 |
| Renal arteritis 10038373 Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Pulmonary vasculitis | 10037457 |
| Renal vasculitis 10038546 Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Radiation vasculitis | 10074671 |
| Retinal occlusive vasculitis 10085059 Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis 10047115 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Renal arteritis | 10038373 |
| Retinal vasculitis 10038905 Rheumatoid vasculitis 10048628 Segmented hyalinising vasculitis 10067527 Takayasu's arteritis 10043097 Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitis 10047111 Vasculitis 10047115 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Renal vasculitis | 10038546 |
| Rheumatoid vasculitis10048628Segmented hyalinising vasculitis10067527Takayasu's arteritis10043097Thromboangiitis obliterans10043540Type 2 lepra reaction10070517Urticarial vasculitis10048820Vaccination site vasculitis10076191Vascular purpura10047097Vasculitic rash10047111Vasculitis10047115Vasculitis gastrointestinal10048319Vasculitis necrotising10047124 | Retinal occlusive vasculitis | 10085059 |
| Segmented hyalinising vasculitis10067527Takayasu's arteritis10043097Thromboangiitis obliterans10043540Type 2 lepra reaction10070517Urticarial vasculitis10048820Vaccination site vasculitis10076191Vascular purpura10047097Vasculitic rash10047111Vasculitis10047115Vasculitis gastrointestinal10048319Vasculitis necrotising10047124 | Retinal vasculitis | 10038905 |
| Takayasu's arteritis10043097Thromboangiitis obliterans10043540Type 2 lepra reaction10070517Urticarial vasculitis10048820Vaccination site vasculitis10076191Vascular purpura10047097Vasculitic rash10047111Vasculitis10047115Vasculitis gastrointestinal10048319Vasculitis necrotising10047124 | Rheumatoid vasculitis | 10048628 |
| Thromboangiitis obliterans 10043540 Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis 10047115 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Segmented hyalinising vasculitis | 10067527 |
| Type 2 lepra reaction 10070517 Urticarial vasculitis 10048820 Vaccination site vasculitis 10076191 Vascular purpura 10047097 Vasculitic rash 10047111 Vasculitis 10047115 Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Takayasu's arteritis | 10043097 |
| Urticarial vasculitis Vaccination site vasculitis Vascular purpura Vasculitic rash Vasculitis Vasculitis 10047097 Vasculitis 10047111 Vasculitis Vasculitis gastrointestinal Vasculitis necrotising 10048319 | Thromboangiitis obliterans | 10043540 |
| Vaccination site vasculitis10076191Vascular purpura10047097Vasculitic rash10047111Vasculitis10047115Vasculitis gastrointestinal10048319Vasculitis necrotising10047124 | Type 2 lepra reaction | 10070517 |
| Vascular purpura10047097Vasculitic rash10047111Vasculitis10047115Vasculitis gastrointestinal10048319Vasculitis necrotising10047124 | Urticarial vasculitis | 10048820 |
| Vasculitic rash10047111Vasculitis10047115Vasculitis gastrointestinal10048319Vasculitis necrotising10047124 | Vaccination site vasculitis | 10076191 |
| Vasculitis10047115Vasculitis gastrointestinal10048319Vasculitis necrotising10047124 | Vascular purpura | 10047097 |
| Vasculitis gastrointestinal 10048319 Vasculitis necrotising 10047124 | Vasculitic rash | 10047111 |
| Vasculitis necrotising 10047124 | Vasculitis | 10047115 |
| | Vasculitis gastrointestinal | 10048319 |
| Viral vasculitis 10056281 | e | 10047124 |
| | Viral vasculitis | 10056281 |

#### Single items PTs:

Glomerulonephritis

Glomerulonephritis acute

Glomerulonephritis chronic

Glomerulonephritis membranoproliferative

Glomerulonephritis membranous

Glomerulonephritis proliferative

Glomerulonephritis rapidly progressive

Mesangioproliferative glomerulonephritis

Immunotactoid glomerulonephritis

Fibrillary glomerulonephritis

Membranous-like glomerulopathy with masked IgG-kappa deposits

Immune-mediated nephritis

Serum sickness

Immune complex level increased

Type III immune complex mediated reaction

# Appendix VII Definition of Concomitant Medication Category

### **Definition of Concomitant Medication Category**

| etanautine N04AB01 anti-parkinson medication orphenadrine (chloride) N04AB02 anti-parkinson medication tribexyphenidyl N04AA01 anti-parkinson medication biperiden N04AA02 anti-parkinson medication biperiden N04AA02 anti-parkinson medication metizene N04AA03 anti-parkinson medication medication metizene N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication procyclidine N04AA05 anti-parkinson medication procyclidine N04AA06 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication anti-parkinson medication dexetimide N04AA08 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication mazaticol N04AA10 anti-parkinson medication mazaticol N04AA10 anti-parkinson medication anti-parkinson medication bornaprine N04AA11 anti-parkinson medication anti-parkinson medication bornaprine N04AA11 anti-parkinson medication anti-parkinson medication tropatepine N04AC01 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication neostigmine N07AA01 Autonomic dysfunction medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication hordstigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication who pyridostigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA03 Autonomic dysfunction medication hordstigmine N07AA03 Autonomic dysfunction medication hordstigmine N07AA03 Autonomic dysfunction medication anti-parkinson medication hordstigmine N04BA01 anti-parkinson medication hordspone N04BX02 anti-parkinson medication anti-parkinson medication hordspone N04BX03 anti-parkinson medication hordspone N04BX04 anti-parkinson medication hordspone N04BX04 anti-parkinson medication hordspone N04BX04 anti-parkinson medication hordspone N04BX04 anti-parkinson medication hordspone N04BX04 anti-parkinson medication N04BA05 anti-parkinson medication N04BA06 anti-parkinson | Name | ATC code | Category |
|---|---|---|---|
| trihexyphenidyl biperiden N04AA01 anti-parkinson medication biperiden N04AA02 anti-parkinson medication biperiden N04AA03 anti-parkinson medication metixene N04AA03 anti-parkinson medication metixene N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication medication procyclidine N04AA04 anti-parkinson medication profenamine N04AA05 anti-parkinson medication anti-parkinson medication dexetimide N04AA08 anti-parkinson medication anti-parkinson medication anti-parkinson medication dexetimide N04AA08 anti-parkinson medication anti-parkin | etanautine | N04AB01 | anti-parkinson medication |
| biperiden N04AA02 anti-parkinson medication biperiden N04AA02 anti-parkinson medication metixene N04AA03 anti-parkinson medication metixene N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication anti-parkinson medication dexetimide N04AA08 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication dexetimide N04AA09 anti-parkinson medication medication anti-parkinson medication dexetimide N04AA09 anti-parkinson medication mazaticol N04AA10 anti-parkinson medication anti-parkinson medication bornaprine N04AA11 anti-parkinson medication anti-parkinson medication benzatropine N04AC01 anti-parkinson medication benzatropine N04AC01 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication neostigmine N07AA01 Autonomic dysfunction medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication N07AA03 Autonomic dysfunction medication when to toleapone N04BX01 anti-parkinson medication entacapone N04BX01 anti-parkinson medication levodopa medication N04BA01 anti-parkinson medication levodopa decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA03 anti-parkinson medication medication N04BA04 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA05 anti-parkinson me | orphenadrine (chloride) | N04AB02 | anti-parkinson medication |
| biperiden metixene N04AA02 anti-parkinson medication metixene N04AA03 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication procyclidine N04AA05 anti-parkinson medication anti-parkinson medication dexetimide N04AA08 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication mazaticol N04AA09 anti-parkinson medication mazaticol N04AA10 anti-parkinson medication bornaprine N04AA10 anti-parkinson medication anti-parkinson medication bornaprine N04AA11 anti-parkinson medication bornaprine N04AC11 anti-parkinson medication etybenzatropine N04AC01 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA03 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication enticapone N04BX02 anti-parkinson medication holdapone N04BX03 anti-parkinson medication levodopa M04BX04 anti-parkinson medication N04BA05 anti-parkinson medication H04BA06 anti-parkinson medication H04BA06 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson | trihexyphenidyl | N04AA01 | anti-parkinson medication |
| metixene N04AA03 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication procyclidine N04AA05 anti-parkinson medication profenamine N04AA05 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication maraticol N04AA10 anti-parkinson medication maraticol N04AA11 anti-parkinson medication morphisms N04AA11 anti-parkinson medication morphisms N04AA11 anti-parkinson medication tropatepine N04AC01 anti-parkinson medication etybenzatropine N04AC01 anti-parkinson medication medication medication medication medication etybenzatropine N04AC02 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication medication pyridostigmine N07AA01 Autonomic dysfunction medication neostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication medication medication medication neostigmine, combinations N07AA03 Autonomic dysfunction medication ambenonium N07AA03 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication anti-parkinson medication neoticapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA03 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medicatio | biperiden | N04AA02 | anti-parkinson medication |
| procyclidine N04AA04 anti-parkinson medication procyclidine N04AA04 anti-parkinson medication north M04AA05 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication mazaticol N04AA09 anti-parkinson medication mazaticol N04AA10 anti-parkinson medication mazaticol N04AA11 anti-parkinson medication mazatropine N04AA11 anti-parkinson medication medication more mazatropine N04AC01 anti-parkinson medication medicati | biperiden | N04AA02 | anti-parkinson medication |
| procyclidine N04AA04 anti-parkinson medication profenamine N04AA05 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication M04AA08 anti-parkinson medication M04AA09 anti-parkinson medication M04AA10 anti-parkinson medication M04AA11 anti-parkinson medication mazaticol N04AA11 anti-parkinson medication morpatepine N04AA12 anti-parkinson medication morpatepine N04AA12 anti-parkinson medication morpatepine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA01 Autonomic dysfunction medication morparidostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication medication medication morparidostigmine, combinations N07AA03 Autonomic dysfunction medication medication morparime, combinations N07AA30 Autonomic dysfunction medication norparkinson medication medication norparkinson medication medication norparkinson medication medication norparkinson medication medication norparkinson medication medication medication norparkinson medication medication norparkinson medication medication norparkinson med | metixene | N04AA03 | anti-parkinson medication |
| profenamine N04AA05 anti-parkinson medication dexetimide N04AA08 anti-parkinson medication M04AA08 anti-parkinson medication M04AA08 anti-parkinson medication M04AA09 anti-parkinson medication M04AA10 anti-parkinson medication M04AA10 anti-parkinson medication M04AA11 anti-parkinson medication M04AA11 anti-parkinson medication M04AA12 anti-parkinson medication modication M04AC01 anti-parkinson medication M04AC01 anti-parkinson medication M04AC02 Autonomic dysfunction medication M04AC02 Autonomic dysfunction medication M04AC02 Autonomic dysfunction medication M04AC02 Autonomic dysfunction medication M04AC03 Autonomic dysfunction medication M04AC03 Autonomic dysfunction medication M04AC03 Autonomic dysfunction medication M04AC03 Autonomic dysfunction medication M04AC03 Autonomic dysfunction medication M04AC04 Autonomic dysfunction medication M04AC04 Autonomic dysfunction medication M04AC04 Autonomic dysfunction medication M04AC04 Autonomic dysfunction medication M04AC04 Autonomic dysfunction medication M04BC04 Autonomic | procyclidine | N04AA04 | anti-parkinson medication |
| dexetimide N04AA08 anti-parkinson medication which anti-parkinson medication sub-parkinson medic | procyclidine | N04AA04 | anti-parkinson medication |
| dexetimide N04AA08 anti-parkinson medication phenglutarimide N04AA09 anti-parkinson medication mazaticol N04AA10 anti-parkinson medication bornaprine N04AA11 anti-parkinson medication tropatepine N04AA12 anti-parkinson medication benzatropine N04AC01 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication etybenzatropine N07AA01 Autonomic dysfunction medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication oneostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication budipine N04BX03 anti-parkinson medication opicapone N04BX04 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication COMT inhibitor melevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | profenamine | N04AA05 | anti-parkinson medication |
| phenglutarimide N04AA09 anti-parkinson medication mazaticol N04AA10 anti-parkinson medication sormaprine N04AA11 anti-parkinson medication hornaprine N04AA12 anti-parkinson medication henzatropine N04AA12 anti-parkinson medication etybenzatropine N04AC01 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication neostigmine N07AA01 Autonomic dysfunction medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication neostigmine, combinations N07AA31 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication hudipine N04BX03 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa, decarboxylase inhibitor N04BA03 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilefrine C01CA01 Autonomic dysfunction medication | dexetimide | N04AA08 | anti-parkinson medication |
| mazaticol N04AA10 anti-parkinson medication bornaprine N04AA11 anti-parkinson medication tropatepine N04AA12 anti-parkinson medication benzatropine N04AC01 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication budipine N04BX03 anti-parkinson medication opicapone N04BX04 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication COMT inhibitor melevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | dexetimide | N04AA08 | anti-parkinson medication |
| bornaprine N04AA11 anti-parkinson medication tropatepine N04AA12 anti-parkinson medication N04AA12 anti-parkinson medication substance of the property of the parkinson medication anti-parkinson medication neostigmine N07AA01 Autonomic dysfunction medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication distipmine N04BX03 anti-parkinson medication levodopa N04BX04 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA01 anti-parkinson medication levodopa, decarboxylase inhibitor N04BA02 anti-parkinson medication N04BA03 anti-parkinson medication nelevodopa decarboxylase inhibitor N04BA04 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 ant | phenglutarimide | N04AA09 | anti-parkinson medication |
| tropatepine N04AA12 anti-parkinson medication benzatropine N04AC01 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication neostigmine N07AA01 Autonomic dysfunction medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication ambenonium N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication budipine N04BX03 anti-parkinson medication levodopa N04BX04 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA01 anti-parkinson medication levodopa decarboxylase inhibitor N04BA03 anti-parkinson medication COMT inhibitor melevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | mazaticol | N04AA10 | anti-parkinson medication |
| benzatropine N04AC01 anti-parkinson medication etybenzatropine N04AC02 anti-parkinson medication neostigmine N07AA01 Autonomic dysfunction medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA03 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication picapone N04BX03 anti-parkinson medication elevodopa N04BX04 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication elevodopa, decarboxylase inhibitor N04BA03 anti-parkinson medication nelevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication nelevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilefrine C01CA01 Autonomic dysfunction medication | bornaprine | N04AA11 | anti-parkinson medication |
| etybenzatropine N04AC02 anti-parkinson medication neostigmine N07AA01 Autonomic dysfunction medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication picapone N04BX03 anti-parkinson medication elevodopa and decarboxylase inhibitor N04BA01 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilefrine C01CA01 Autonomic dysfunction medication | tropatepine | N04AA12 | anti-parkinson medication |
| neostigmine N07AA01 Autonomic dysfunction medication neostigmine N07AA01 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication budipine N04BX03 anti-parkinson medication opicapone N04BX04 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA01 anti-parkinson medication anti-parkinson medication levodopa, decarboxylase inhibitor N04BA02 anti-parkinson medication M04BA03 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA03 anti-parkinson medication medication M04BA03 anti-parkinson medication anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication etilefrine C01CA01 Autonomic dysfunction medication | benzatropine | N04AC01 | anti-parkinson medication |
| neostigmineN07AA01Autonomic dysfunction medicationpyridostigmineN07AA02Autonomic dysfunction medicationpyridostigmineN07AA02Autonomic dysfunction medicationdistigmineN07AA03Autonomic dysfunction medicationdistigmineN07AA03Autonomic dysfunction medicationambenoniumN07AA30Autonomic dysfunction medicationneostigmine, combinationsN07AA51Autonomic dysfunction medicationtolcaponeN04BX01anti-parkinson medicationentacaponeN04BX02anti-parkinson medicationbudipineN04BX03anti-parkinson medicationopicaponeN04BX04anti-parkinson medicationlevodopaN04BA01anti-parkinson medicationlevodopa and decarboxylase inhibitorN04BA02anti-parkinson medicationCOMT inhibitorN04BA03anti-parkinson medicationmelevodopaN04BA04anti-parkinson medicationmelevodopa and decarboxylase inhibitorN04BA05anti-parkinson medicationetilevodopa and decarboxylase inhibitorN04BA06anti-parkinson medicationfludrocortisoneH02AA02Autonomic dysfunction medicationetilefrineC01CA01Autonomic dysfunction medication | etybenzatropine | N04AC02 | anti-parkinson medication |
| pyridostigmine N07AA02 Autonomic dysfunction medication pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication Mo7AA03 Autonomic dysfunction medication ambenonium N07AA03 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication medication with tolcapone N04BX02 anti-parkinson medication hudipine N04BX03 anti-parkinson medication opicapone N04BX04 anti-parkinson medication levodopa N04BA01 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa, decarboxylase inhibitor N04BA03 anti-parkinson medication Mo4BA03 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | neostigmine | N07AA01 | Autonomic dysfunction medication |
| pyridostigmine N07AA02 Autonomic dysfunction medication distigmine N07AA03 Autonomic dysfunction medication M07AA03 Autonomic dysfunction medication M07AA03 Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication N07AA51 Autonomic dysfunction medication meostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication medication metacapone N04BX02 anti-parkinson medication medication will budipine N04BX03 anti-parkinson medication medication medicapone N04BX04 anti-parkinson medication levodopa N04BA01 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication melevodopa, decarboxylase inhibitor N04BA03 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | neostigmine | N07AA01 | Autonomic dysfunction medication |
| distigmine N07AA03 Autonomic dysfunction medication N07AA03 Autonomic dysfunction medication Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication N07AA51 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication anti-parkinson medication neotacapone N04BX02 anti-parkinson medication neotacapone N04BX03 anti-parkinson medication neotacapone N04BX04 anti-parkinson medication neotacapone N04BX04 anti-parkinson medication neotacapone N04BA01 anti-parkinson medication neotacapone neotacapone N04BA02 anti-parkinson medication neotacapone neotacapone N04BA03 anti-parkinson medication neotacapone | pyridostigmine | N07AA02 | Autonomic dysfunction medication |
| distigmine N07AA03 Autonomic dysfunction medication ambenonium N07AA30 Autonomic dysfunction medication neostigmine, combinations N07AA51 Autonomic dysfunction medication tolcapone N04BX01 anti-parkinson medication anti-parkinson medication hudipine N04BX02 anti-parkinson medication anti-parkinson medication picapone N04BX04 anti-parkinson medication levodopa N04BA01 anti-parkinson medication anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa, decarboxylase inhibitor N04BA03 anti-parkinson medication COMT inhibitor melevodopa and decarboxylase inhibitor N04BA04 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | pyridostigmine | N07AA02 | Autonomic dysfunction medication |
| ambenonium N07AA30 Autonomic dysfunction medication N07AA51 Autonomic dysfunction medication N04BX01 entacapone N04BX02 anti-parkinson medication N04BX03 anti-parkinson medication N04BX04 anti-parkinson medication N04BX05 anti-parkinson medication N04BX06 anti-parkinson medication N04BX07 anti-parkinson medication N04BX08 anti-parkinson medication N04BX09 anti-parkinson medication N04BA01 levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication N04BA03 anti-parkinson medication N04BA03 anti-parkinson medication N04BA03 anti-parkinson medication melevodopa and decarboxylase inhibitor melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | distigmine | N07AA03 | Autonomic dysfunction medication |
| neostigmine, combinations N07AA51 Autonomic dysfunction medication anti-parkinson medication entacapone N04BX02 anti-parkinson medication budipine N04BX03 anti-parkinson medication opicapone N04BX04 anti-parkinson medication levodopa N04BA01 levodopa and decarboxylase inhibitor N04BA02 levodopa, decarboxylase inhibitor and COMT inhibitor melevodopa M04BA04 molevodopa and decarboxylase inhibitor melevodopa N04BA05 melevodopa and decarboxylase inhibitor N04BA05 melevodopa and decarboxylase inhibitor N04BA06 melevodopa and decarboxylase inhibitor N04BA06 fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | distigmine | N07AA03 | Autonomic dysfunction medication |
| tolcapone N04BX01 anti-parkinson medication entacapone N04BX02 anti-parkinson medication budipine N04BX03 anti-parkinson medication opicapone N04BX04 anti-parkinson medication levodopa N04BA01 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa, decarboxylase inhibitor and COMT inhibitor melevodopa N04BA04 anti-parkinson medication melevodopa N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | ambenonium | N07AA30 | Autonomic dysfunction medication |
| entacapone N04BX02 anti-parkinson medication budipine N04BX03 anti-parkinson medication opicapone N04BX04 anti-parkinson medication levodopa N04BA01 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa, decarboxylase inhibitor and COMT inhibitor melevodopa N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | neostigmine, combinations | N07AA51 | Autonomic dysfunction medication |
| budipine N04BX03 anti-parkinson medication opicapone N04BX04 anti-parkinson medication levodopa N04BA01 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa, decarboxylase inhibitor and COMT inhibitor melevodopa N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | tolcapone | N04BX01 | anti-parkinson medication |
| opicapone N04BX04 anti-parkinson medication levodopa N04BA01 anti-parkinson medication levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa, decarboxylase inhibitor and COMT inhibitor melevodopa N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | entacapone | N04BX02 | anti-parkinson medication |
| levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa, decarboxylase inhibitor and COMT inhibitor melevodopa N04BA03 anti-parkinson medication melevodopa N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | budipine | N04BX03 | anti-parkinson medication |
| levodopa and decarboxylase inhibitor N04BA02 anti-parkinson medication levodopa, decarboxylase inhibitor and COMT inhibitor melevodopa N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | opicapone | N04BX04 | anti-parkinson medication |
| levodopa, decarboxylase inhibitor and COMT inhibitor melevodopa N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | levodopa | N04BA01 | anti-parkinson medication |
| melevodopa N04BA04 anti-parkinson medication melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | levodopa and decarboxylase inhibitor | N04BA02 | anti-parkinson medication |
| melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | | N04BA03 | anti-parkinson medication |
| melevodopa and decarboxylase inhibitor N04BA05 anti-parkinson medication etilevodopa and decarboxylase inhibitor N04BA06 anti-parkinson medication fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | melevodopa | N04BA04 | anti-parkinson medication |
| fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | _ | N04BA05 | |
| fludrocortisone H02AA02 Autonomic dysfunction medication etilefrine C01CA01 Autonomic dysfunction medication | | N04BA06 | _ |
| etilefrine C01CA01 Autonomic dysfunction medication | | H02AA02 | _ |
| | etilefrine | C01CA01 | |
| | etilefrine | C01CA01 | |

| Name | ATC code | Category |
|--------------------------|----------|----------------------------------|
| isoprenaline | C01CA02 | Autonomic dysfunction medication |
| isoprenaline | C01CA02 | Autonomic dysfunction medication |
| norepinephrine | C01CA03 | Autonomic dysfunction medication |
| dopamine | C01CA04 | Autonomic dysfunction medication |
| norfenefrine | C01CA05 | Autonomic dysfunction medication |
| phenylephrine | C01CA06 | Autonomic dysfunction medication |
| dobutamine | C01CA07 | Autonomic dysfunction medication |
| oxedrine | C01CA08 | Autonomic dysfunction medication |
| oxedrine | C01CA08 | Autonomic dysfunction medication |
| metaraminol | C01CA09 | Autonomic dysfunction medication |
| methoxamine | C01CA10 | Autonomic dysfunction medication |
| mephentermine | C01CA11 | Autonomic dysfunction medication |
| dimetofrine | C01CA12 | Autonomic dysfunction medication |
| prenalterol | C01CA13 | Autonomic dysfunction medication |
| dopexamine | C01CA14 | Autonomic dysfunction medication |
| gepefrine | C01CA15 | Autonomic dysfunction medication |
| ibopamine | C01CA16 | Autonomic dysfunction medication |
| midodrine | C01CA17 | Autonomic dysfunction medication |
| octopamine | C01CA18 | Autonomic dysfunction medication |
| fenoldopam | C01CA19 | Autonomic dysfunction medication |
| cafedrine | C01CA21 | Autonomic dysfunction medication |
| arbutamine | C01CA22 | Autonomic dysfunction medication |
| theodrenaline | C01CA23 | Autonomic dysfunction medication |
| epinephrine | C01CA24 | Autonomic dysfunction medication |
| amezinium metilsulfate | C01CA25 | Autonomic dysfunction medication |
| ephedrine | C01CA26 | Autonomic dysfunction medication |
| droxidopa | C01CA27 | Autonomic dysfunction medication |
| combinations | C01CA30 | Autonomic dysfunction medication |
| etilefrine, combinations | C01CA51 | Autonomic dysfunction medication |
| emepronium | G04BD01 | Autonomic dysfunction medication |
| emepronium | G04BD01 | Autonomic dysfunction medication |
| flavoxate | G04BD02 | Autonomic dysfunction medication |
| meladrazine | G04BD03 | Autonomic dysfunction medication |
| oxybutynin | G04BD04 | Autonomic dysfunction medication |
| oxybutynin | G04BD04 | Autonomic dysfunction medication |
| terodiline | G04BD05 | Autonomic dysfunction medication |
| propiverine | G04BD06 | Autonomic dysfunction medication |
| tolterodine | G04BD07 | Autonomic dysfunction medication |
| solifenacin | G04BD08 | Autonomic dysfunction medication |
| trospium | G04BD09 | Autonomic dysfunction medication |
| darifenacin | G04BD10 | Autonomic dysfunction medication |
| fesoterodine | G04BD11 | Autonomic dysfunction medication |
| mirabegron | G04BD12 | Autonomic dysfunction medication |

| Name | ATC code | Category |
|---------------------------|----------|----------------------------------|
| desfesoterodine | G04BD13 | Autonomic dysfunction medication |
| octreotide | H01CB02 | Autonomic dysfunction medication |
| vasopressin (argipressin) | H01BA01 | Autonomic dysfunction medication |
| desmopressin | H01BA02 | Autonomic dysfunction medication |
| lypressin | H01BA03 | Autonomic dysfunction medication |
| lypressin | H01BA03 | Autonomic dysfunction medication |
| terlipressin | H01BA04 | Autonomic dysfunction medication |
| ornipressin | H01BA05 | Autonomic dysfunction medication |